#### The GlaxoSmithKline group of companies

| Division | : | Worldwide Development |
|------------------|---|-----------------------------------|
| Information Type | : | Reporting and Analysis Plan (RAP) |

Title: Reporting and Analysis Plan for A Phase IIb, Multicenter, Open-label, Rollover Study Evaluating the Efficacy, Safety and Tolerability of Long-acting Cabotegravir Plus Long-acting Rilpivirine Administered Every Two Months in HIV-1 infected Adults who are Virologically Suppressed and Participated in Study LAI116482Compound Number: GSK1265744Effective Date: 31-JAN-2020

#### **Description:**

- The purpose of this RAP is to describe the planned analyses and output to be included in the Clinical Study Report for Protocol 209035.
- This RAP is intended to describe the efficacy, safety and tolerability analyses required for the study.
- This RAP will be provided to the study team members to convey the content of the Statistical Analysis Complete (SAC) deliverable.

#### **RAP Author(s):**

| Approver | Date | Approval Method |
|------------------------------------|------------|-----------------|
| PPD | 31-01-2020 | Email |
| Senior Statistician II, Quanticate | 31-01-2020 | Elliali |

Copyright 2020 the GlaxoSmithKline group of companies. All rights reserved. Unauthorised copying or use of this information is prohibited.

## The GlaxoSmithKline group of companies

# **RAP Team Approvals:**

| Approver | Date | Approval Method |
|---|---|---|
| Clinical Development Manager, ([HIV] [ViiV Sci Med Officer]) | 31-01-2020 | Email |
| Programming Manager (HIV, Clinical Programming) | 31-01-2020 | Email |

# **Clinical Statistics and Clinical Programming Line Approvals:**

| Approver | Date | Approval Method |
|---|---|---|
| Manager, Statistics (Infectious Diseases, Clinical Statistics) | 31-01-2020 | Email |
| Programming Manager (Infectious Diseases, Clinical Programming) | 31-01-2020 | Email |

# **TABLE OF CONTENTS**

| | | | PAGE |
|---|---|---|---|
| 1. | INTRO | DDUCTION | 6 |
| 2. | SUMN | MARY OF KEY PROTOCOL INFORMATION | 6 |
| | 2.1. | Changes to the Protocol Defined Statistical Analysis Plan | |
| | 2.2. | Study Objective(s) and Endpoint(s) | |
| | 2.3. | Study Design | |
| | 2.4. | Statistical Hypotheses / Statistical Analyses | |
| 3. | PLAN | NED ANALYSES | 10 |
| | 3.1. | Interim Analyses | 10 |
| | 3.2. | Final Analyses | 10 |
| 4. | | YSIS POPULATIONS | |
| | 4.1. | Protocol Deviations | 11 |
| 5. | | SIDERATIONS FOR DATA ANALYSES AND DATA HANDLING | |
| | | /ENTIONS | |
| | 5.1.<br>5.2. | Study Treatment & Sub-group Display Descriptors | |
| | 5.2.<br>5.3. | Baseline Definitions | |
| | 5.3.<br>5.4. | Examination of Covariates, Other Strata and Subgroups | |
| | 5.4. | 5.4.1. Covariates and Other Strata | |
| | | 5.4.2. Examination of Subgroups | |
| | 5.5. | Multiple Comparisons and Multiplicity | |
| | 0.0. | 5.5.1. Primary Comparison of Interest | |
| | 5.6. | Other Considerations for Data Analyses and Data Handling | |
| | | Conventions | 14 |
| 6. | | Y POPULATION ANALYSES | |
| | 6.1. | Overview of Planned Study Population Analyses | |
| | 6.2. | Prior and Concomitant Medications | 16 |
| 7. | | CACY ANALYSES | |
| | 7.1. | Primary Efficacy Analyses | |
| | | 7.1.1. Endpoint / Variables | |
| | | 7.1.2. Summary Measure | |
| | | 7.1.3. Population of Interest | |
| | | <ul><li>7.1.4. Strategy for Intercurrent (Post-treatment selection) Events</li><li>7.1.5. Statistical Analyses / Methods</li></ul> | |
| | 7.2. | Secondary Efficacy Analyses | |
| | 1.2. | 7.2.1. Endpoint / Variables | |
| | | 7.2.2. Summary Measure | |
| | | 7.2.3. Population of Interest | |
| | | 7.2.4. Strategy for Intercurrent (Post-treatment selection) Events | |
| | | 7.2.5. Statistical Analyses / Methods | |
| | 7.3. | Exploratory Efficacy Analyses | |
| 8. | SVEE | TY ANALYSES | 21 |
| Ο. | 8.1. | | |

#### CONFIDENTIAL

| | 8.2.<br>8.3.<br>8.4. | Adverse | Injection Site Reactionsaboratory Analyses<br>Events of Special Interest Analysesfety Analyses | 21<br>22 |
|---|---|---|---|---|
| 9. | ΗΕΔΙΊ | ГН ОПТСО | DMES ANALYSES | 23 |
| J. | 9.1. | | / Variables | |
| | 9.2. | • | / Measure | |
| | 9.3. | • | n of Interest | |
| | 9.4. | • | for Intercurrent (Post-treatment selection) Events | |
| | 9.5. | | I Analyses / Methods | |
| 10. | VIROL | .OGY | | .24 |
| 11 | DEEEL | DENCES | | 26 |
| 11. | KEFE | KENCES | | . 20 |
| 12. | APPE | NDICES | | .27 |
| | 12.1. | Appendix | 1: Protocol Deviation Management and Definitions for Per | |
| | | | Population | |
| | | | Exclusions from Per Protocol Population | |
| | 12.2. | | 2: Schedule of Activities | . 29 |
| | | 12.2.1. | Protocol Defined Schedule of Events for CAB LA + RPV | |
| | | 40.00 | LA Q2M Administration | .29 |
| | | 12.2.2. | Protocol Defined Schedule of Events for DTG + RPV | 00 |
| | | 40.00 | Administration | .33 |
| | | 12.2.3. | Protocol Defined Schedule of Events for Long Term Follow Up | 25 |
| | 12.3. | Annondiv | 3: Assessment Windows | |
| | 12.3. | 12.3.1. | Definitions of Assessment Windows for Analyses | |
| | | 12.3.1. | Definitions of Assessment Windows for Data Other than | . 31 |
| | | 12.0.2. | Health Outcomes | 37 |
| | | 12.3.3. | Assessment Window for Study Conclusion | |
| | | 12.3.4. | Assessment Window for Health Outcome Data | |
| | | | 12.3.4.1. HIVTSQs, HIVTSQc, HIVDQoL, Preference | |
| | | | 12.3.4.2. Reasons for Switch | |
| | | 12.3.5. | Multiple assessments within an Analysis Window | 42 |
| | 12.4. | Appendix | 4: Study Phases and Treatment State | .43 |
| | | 12.4.1. | Study Phases | |
| | | 12.4.2. | Treatment State | |
| | | | 12.4.2.1. Treatment States for AE Data | .45 |
| | 12.5. | Appendix | 5: Data Display Standards & Handling Conventions | |
| | | 12.5.1. | Reporting Process | |
| | | 12.5.2. | Reporting Standards | |
| | 12.6. | | 6: Derived and Transformed Data | |
| | | 12.6.1. | General | |
| | | 12.6.2. | Study Population | |
| | | 12.6.3. | Efficacy | |
| | | 12.6.4.<br>12.6.5. | Safety Health Outcomes | |
| | | 12.6.5.<br>12.6.6. | Virology | |
| | 12.7. | | 7: Reporting Standards for Missing Data | |
| | 14.1. | | Premature Withdrawals | |
| | | | T TOTALGEO TELLIGIOTATION | |

#### **CONFIDENTIAL**

| | 12.7.2. | Handling of Missing Data | |
|---|---|---|---|
| | | 12.7.2.1. Handling of Missing and Partial Dates | 75 |
| 12.8. | <b>Appendix</b> | 8: Values of Potential Clinical Importance | 76 |
| | 12.8.1. | Laboratory Values | 76 |
| | 12.8.2. | ECG | 76 |
| 12.9. | <b>Appendix</b> | 9: Snapshot Algorithm Details | 77 |
| | | 10: Identification of Adverse Events of Special Interest | |
| | | 11: Abbreviations & Trade Marks | |
| | | Abbreviations | |
| | | Trademarks | |
| 12.12. | | 12: List of Data Displays | |
| | | Data Display Numbering | |
| | | Mock Example Shell Referencing | |
| | | Deliverables | |
| | | Study Population Tables | |
| | | Efficacy Tables | |
| | | Efficacy Figures | |
| | | Safety Tables | |
| | | Safety Figures | |
| | | Health Outcomes Tables | |
| | | Virology Tables | |
| | | <b>0</b> , | |
| | | .ICH Listings | |
| 10.10 | | Non-ICH Listings | |
| 12.13. | Appendix | c 13: Example Mock Shells for Data Displays | .140 |

#### 1. INTRODUCTION

The purpose of this reporting and analysis plan (RAP) is to describe the analyses to be included in the Clinical Study Report for Protocol:

| Revision Chronology: | | |
|---|---|---|
| 2018N356280_00 | 16-MAY-2018 | Original |
| 2018N356280_01 | 22-JUN-2018 | This amendment was completed to clarify procedures, adjust exclusion criteria, add missing risk assessment language and to clean up minor grammatical errors. |

#### 2. SUMMARY OF KEY PROTOCOL INFORMATION

# 2.1. Changes to the Protocol Defined Statistical Analysis Plan

The following are changes or deviations to the originally planned statistical analysis specified in the 209035 protocol amendment 1 [(Dated: 22/JUN/2018)]:

- PK samples would not be analysed and no PK outputs would be produced. Due to the
  vast amount of PK data available from other studies examining CAB LA + RPV LA
  PK data, CPMS decided not to evaluate PK data from this study. Additionally, the
  time points of PK sample collection correspond to peak, rather than trough,
  concentrations.
- Data from the digital assistance program was not collected due to cost concerns of using Ensemble and will not be analysed.

# 2.2. Study Objective(s) and Endpoint(s)

| Objectives | Endpoints |
|---|---|
| Primary Objectives | Primary Endpoints |
| To demonstrate the antiviral activity of CAB LA + RPV LA every 2 months in suppressed HIV-1 infected antiretroviral therapy ART-experienced participants | <ul> <li>Proportion of participants with HIV-RNA ≥ 50 c/mL<br/>as per FDA Snapshot algorithm at Month 12</li> </ul> |
| Secondary Objectives | Secondary Endpoints |
| To demonstrate the antiviral and immunologic activity of CAB LA + RPV LA every 2 months and oral DTG +RPV once daily | <ul> <li>Proportion of participants with plasma HIV-1 RNA &lt;50 c/mL (c/mL) at Month 12 using the FDA Snapshot algorithm</li> <li>Proportion of participants with protocol-defined confirmed virologic failure (CVF) over time</li> <li>Proportion of participants with HIV-RNA greater than or equal to 50 c/mL as per FDA Snapshot algorithm over time</li> <li>Absolute values and changes from Baseline in viral load and CD4+ cell counts over time</li> </ul> |
| To demonstrate the safety and | Incidence and severity of AEs and laboratory |

| Objectives | Endpoints |
|---|---|
| tolerability of CAB LA + RPV LA every 2 months and oral DTG + RPV once daily To assess viral resistance in | <ul> <li>abnormalities over time</li> <li>Proportion of participants who discontinue treatment due to AEs over time</li> <li>Change from Baseline in laboratory parameters over time</li> <li>Incidence of treatment emergent genotypic and</li> </ul> |
| participants experiencing protocol-<br>defined confirmed virologic failure | phenotypic resistance to CAB, RPV, and DTG + RPV |
| To assess participant reported health-related quality of life, treatment satisfaction, injection tolerability, and treatment acceptance. | <ul> <li>Change from Baseline (Day 1) in HIVDQoL at Months 6 and 12 (or Withdrawal)</li> <li>Change from baseline (Day 1) in total "treatment satisfaction" score, and individual item scores of the HIV Treatment Satisfaction Status Questionnaire (HIVTSQs) at Months 6 and 12 (or Withdrawal)</li> <li>Change in treatment satisfaction over time using the HIV Treatment Satisfaction Change Questionnaire HIVTSQc at Month 12 (or Withdrawal).</li> </ul> |
| Exploratory Objectives | Exploratory Endpoints |
| <ul> <li>To assess reason for switching using a single question</li> <li>To assess preference using a single question</li> </ul> | <ul> <li>The 'Preference" question will be used to assess preference for CAB LA + RPV LA every 2 months compared to prior oral CAB + RPV regimen, at Month 12 using a single dichotomous preference question.</li> <li>The "Reason for Switch" question will be administered at Day 1 (Baseline) to assess the reasons for willingness to switch to LA injectable ART or to another oral regimen.</li> </ul> |

#### 2.3. Study Design



- § All participants in LATTE administered oral CAB 30 mg + RPV 25 mg
- † Access commercially once Q8W is approved
- # Access longer term via commercial route. Participants will continue to receive DTG + RPV if located in a region where not commercially available.

# Design Features

The study is a Phase IIb, open-label, 2 arms, multicenter rollover study designed to assess the antiviral activity and safety of CAB LA + RPV LA administered every 2 months in approximately 100 adult HIV-1 infected participants from the LATTE study.

Participants who fulfill eligibility requirements will be entered into the study to receive CAB LA + RPV LA Q2M or the oral DTG + RPV regimen for at least 12 months, until commercially available.

Any participant who receives at least one dose of CAB LA and/or RPV LA and discontinues the CAB LA + RPV LA regimen for any reason will enter a 52-week LTFU Phase. Those participants must remain on suppressive HAART for at least 52 weeks after the last dose of CAB LA and/or RPV LA.

#### Dosing

#### Group 1:

First Injections (Loading Doses) – Day 1 and Month 2

#### Day 1:

- Receive last dose of oral CAB + RPV regimen
- Receive CAB LA 600 mg given as 1 X 3 mL IM injection
- Receive RPV LA 900 mg given as 1 X 3 mL IM injection

#### Month 2:

- Receive CAB LA 600 mg given as 1 X 3 mL IM injection
- Receive RPV LA 900 mg given as 1 X 3 mL IM injection

Maintenance Injections – every 2 months (Q2M) following Month 2 Month 4 to End of Study (two 3 mL injections every 2 months):

- Receive CAB LA 600 mg given as 1 X 3 mL IM injection
- Receive RPV LA 900 mg given as 1 X 3 mL IM injection

| Overview of St | Overview of Study Design and Key Features |
|---|---|
| | Group 2: |
| | Day 1 to Month 12 (once daily FDC tablet taken with food): |
| | Take one tablet of DTG 50 mg + RPV 25 mg once daily |
| | See the protocol Table 2. |
| Time & | Refer to Appendix 2: Schedule of Activities |
| Events | |
| Treatment | Participants transitioning from the LATTE study on oral CAB + RPV treatment will |
| Assignment | transition to their elected treatment regimen, either Q2M administration of CAB LA |
| | + RPV LA or oral DTG + RPV single tablet regimen. |
| Interim | No Interim Analysis will be conducted. |
| Analysis | |

# 2.4. Statistical Hypotheses / Statistical Analyses

No statistical hypotheses of treatment comparisons will be conducted within this study.

#### 3. PLANNED ANALYSES

At least one analyses will be conducted to evaluate primary and secondary objectives of the protocol after all subjects have completed their visits at Month 12. Further data cuts and analyses may be conducted as necessary after Month 12 to support regulatory publications. The Month 12 analysis will be primary. Further analyses may be conducted when all subjects on CAB LA + RPV LA have completed their Month 26 visit or when all subjects have completed the study (final End-of-Study analysis).

## 3.1. Interim Analyses

No Interim Analysis will be conducted.

#### 3.2. Final Analyses

The primary analysis will be conducted to evaluate the primary objective of the study at Month 12. These analyses will be performed after the completion of the following sequential steps:

- 1. All participants have completed Month 12 as defined in the protocol.
- 2. All required database cleaning activities have been completed and final database release (DBR) and database freeze (DBF) has been declared by Data Management.

A final End-of-Study analysis will be conducted when all subjects have completed the study as defined in the protocol. Additional analysis may be conducted when all subjects on CAB LA + RPV LA have completed their Month 26 visit.

#### 4. ANALYSIS POPULATIONS

| Population | Definition / Criteria | | Analyses Evaluated |
|---|---|---|---|
| All Participants | | • | Study Population |
| Screened | For disposition displays, except for the listing of | | |
| | subjects who were rescreened, only the latest re- | | |
| | screening data will be included. All screening data | | |
| | will be summarized or listed for other displays. | | |
| All Participants | All participants transitioning from the LATTE study | • | Study Population |
| Enrolled | and signed the informed consent form (ICF). | | |
| Safety Population | All participants who receive at least one dose of IP | • | Safety |
| | on or after Day 1 visit. | | · |
| | Participants will be assessed according to actual | | |
| | treatment received. | | |
| Intent-to-Treat | All participants who receive at least one dose of IP | • | Study Population |
| Exposed | during on or after Day 1 visit. | • | Efficacy |
| Population (ITT- | Participants will be analyzed according to the | | , |
| E) | selected treatment regardless of what treatment was | | |
| | actually received. This population will be used for all | | |
| | summaries unless otherwise specified. | | |

| Population | Definition / Criteria | Analyses Evaluated |
|---|---|---|
| Per-Protocol<br>Exposed (PP-E) | All participants in the ITT-E Population who comply with the protocol except for major protocol violators. Protocol deviations that would exclude subjects from the PP-E population are defined in Section 4.1 (Protocol Deviations) and Appendix 1 (Protocol Deviation Management and Definition for Per-Protocol Population). | • PP |
| Confirmed Virologic Failure (CVF) | All participants in the ITT-E population who met Confirmed Virologic Failure (CVF) criteria. | <ul><li>Virology</li><li>Efficacy</li></ul> |
| Long-tem Follow-<br>up | All subjects receiving at least one dose of CAB LA and/or RPV LA who have discontinued the CAB LA + RPV LA regimen and have at least one Long-term Follow-up phase clinic visit (i.e. have at least one long-term follow-up visit shown in the study database, LTFU month 1, LTFU month 3, etc). | Safety |

Refer to Appendix 12: List of Data Displays which details the population used for each display.

#### 4.1. Protocol Deviations

Important protocol deviations (including deviations related to study inclusion/exclusion criteria, conduct of the trial, patient management or patient assessment) will be summarised and listed.

Important deviations which result in exclusion from the analysis population will also be summarised and listed. (Please refer to Appendix 1: Protocol Deviation Management and Definitions for Per Protocol Population).

Protocol deviations will be tracked by the study team throughout the conduct of the study in accordance with the Protocol Deviation Management Plan.

- Data will be reviewed prior to freezing the database to ensure all important deviations and deviations which may lead to exclusion from the analysis are captured and categorised on the protocol deviations dataset.
- This dataset will be the basis for the summaries and listings of protocol deviations.

A separate summary and listing of all inclusion/exclusion criteria deviations will also be provided. This summary will be based on data as recorded on the inclusion/exclusion page of the eCRF.

# 5. CONSIDERATIONS FOR DATA ANALYSES AND DATA HANDLING CONVENTIONS

## 5.1. Study Treatment & Sub-group Display Descriptors

| Treatment Group Descriptions | | | |
|---|---|---|---|
| | RandAll NG Data Displays for Reporting | | |
| Code | Description | Description | Order in TLF |
| Α | CAB LA (600 mg) + RPV LA (900 mg) Q2M | Q2M | 1 |
| В | Oral DTG (50mg) + RPV (25mg) daily | DTG + RPV | 2 |

#### 5.2. Baseline Definitions

Baseline information to be collected at Day 1 includes general medical history and current medical conditions. Laboratory and health outcomes assessments will also be assessed. Questionnaire/surveys are recommended to be administered at the beginning of the visit before any other assessments are conducted, in the order specified. For participants who agree to the optional assessment, a whole blood sample for genetic research should be collected at Day 1 (if not already collected during participation in the LATTE study). For all endpoints (except as noted in baseline definitions) the baseline value will be the latest pre-dose assessment with a non-missing value, including those from unscheduled visits. If time is not collected, Day 1 assessments are assumed to be taken prior to first dose and used as baseline. See the protocol Section 8.2 for more details.

Unless otherwise stated, if baseline data is missing no derivation will be performed and baseline will be set to missing.

#### 5.3. Multicentre Studies

Data will be summarized for all centres combined. The primary efficacy endpoint will be summarized by Country. Countries will be combined if the number of participants enrolled is low.

### 5.4. Examination of Covariates, Other Strata and Subgroups

#### 5.4.1. Covariates and Other Strata

The list of covariates may be used in descriptive summaries. Additional covariates of clinical interest may also be considered.

| Category | Details |
|------------|------------------------------|
| Strata | None |
| Covariates | See details in Section 5.4.2 |

## 5.4.2. Examination of Subgroups

The following is a list of subgroups that may be used in descriptive summaries. Additional subgroups of clinical interest may also be considered.

- If the percentage of subjects is small within a particular subgroup, then the subgroup categories may be combined.
- Additional covariates of clinical interest may also be considered.

| Category | Covariates and / or Subgroups |
|---|---|
| Demographic and Baseline<br>Characteristic Subgroups | <ul> <li>Age (years): <ul> <li>35, 35 - &lt;50,≥50</li> <li>≤18, 19 - 64, ≥65 (FDAAA requirement)</li> <li>18 - 64, 65 - 84, ≥85 (EMA requirement)</li> </ul> </li> <li>Race: <ul> <li>White, Non-White</li> <li>Black/African American, Non-Black/African American</li> </ul> </li> <li>Sex at birth: <ul> <li>Female</li> <li>Male</li> </ul> </li> <li>Country: <ul> <li>Canada</li> <li>United States</li> </ul> </li> <li>Derived Baseline Centers for Disease Control and Prevention (CDC) category: <ul> <li>Stage II</li> <li>Stage III</li> <li>Baseline BMI (kg/m²)</li> <li>&lt;30</li> <li>≥30</li> </ul> </li> </ul> |
| Additional subgroup for common drug-related study drug injection site reaction (ISR) with maximum toxicity grade | For each preferred term of the common drug-related study drug ISR with maximum toxicity grade (pain, induration, nodules and any other study drug ISR with ≥5% subjects in either treatment arm) during the maintenance phase: • Needle Length for Last CAB Injection prior to and including the onset date of the earliest corresponding drug-related CAB ISR with maximum toxicity grade during the maintenance phase: ≤1.5, >1.5 to <2, ≥2 inches • Needle Length for Last RPV Injection prior to and including the onset date of the earliest corresponding drug-related RPV ISR with maximum toxicity grade during the maintenance phase: ≤1.5, >1.5 to <2, ≥2 inches Note: If there is no ISR of interest reported during maintenance |

| Category | Covariates and / or Subgroups |
|---|---|
| | phase for a subject, the needle length of last injection during |
| | maintenance phase will be used in the summary. |

# 5.5. Multiple Comparisons and Multiplicity

## 5.5.1. Primary Comparison of Interest

No formal statistical analysis will be performed for this study. The primary endpoint will be summarized based on the ITT-E population.

# 5.6. Other Considerations for Data Analyses and Data Handling Conventions

Other considerations for data analyses and data handling conventions are outlined in the appendices:

| Section | Component |
|---------|-------------------------------------------------------------------|
| 12.3 | Appendix 3: Assessment Windows |
| 12.4 | Appendix 4: Study Phases and Treatment Emergent Adverse Events |
| 12.5 | Appendix 5: Data Display Standards & Handling Conventions |
| 12.6 | Appendix 6: Derived and Transformed Data |
| 12.7 | Appendix 7: Reporting Standards for Missing Data |
| 12.8 | Appendix 8: Values of Potential Clinical Importance |
| 12.9 | Appendix 9: Snapshot Algorithm Details |
| 12.10 | Appendix 10: Identification of Adverse Events of Special Interest |

### 6. STUDY POPULATION ANALYSES

#### 6.1. Overview of Planned Study Population Analyses

The study population will be based on the Intent-to-Treat Exposed population, unless otherwise specified.

Study population analyses including analyses of subject's disposition, protocol deviations, demographic and baseline characteristics, prior and concomitant medications, and exposure and treatment compliance will be based on GSK Core Data Standards.

Table 1 provides an overview of the planned study population analyses, with details of the planned displays presented in Appendix 12: List of Data Displays.

Table 1 Overview of Planned Study Population Analyses

| Display Type | Data Displays Generated | |
|---|---|---|
| | Table | Listing |
| Randomization | | |
| Randomization [1] | | <b>Y</b> [2] |
| Subject Disposition | | |
| Study Populations [3] | Υ | |
| Study Recruitment [3] | Υ | Υ |
| Reasons for Screening Failures [3] | Υ | Υ |
| Rescreened Subjects [3] | | Y |
| Age Ranges | Y | |
| Subject Disposition | <b>Y</b> [4][5] | |
| Reasons for Withdrawal by Visit | <b>Y</b> [4][5] | Y |
| IP Discontinuation | Y | Y |
| Important Protocol Deviations | Y | Υ |
| Deviations leading to exclusion from PP | Y | Y |
| Inclusion and Exclusion Criteria Deviations | Y | Y |
| Demography and Baseline | · | |
| Demographics Characteristics | Y | Υ |
| Race & Racial Combinations [6] | Y | Υ |
| Hepatitis Status | Y | |
| CDC Classification of HIV infection (2014) | Y | |
| Distribution of CD4+ Cell Counts at Baseline | Y | |
| HIV-1 Risk Factors | Y | |

| Display Type | Data Dis <sub>l</sub> | olays Generated |
|---|---|---|
| | Table | Listing |
| Medical Conditions, Concomitant Medications & Antiretrov | viral Therapy | |
| Medical Conditions (Current/Past) [7] | Υ | |
| Medical Conditions: Sub-conditions (Current/Past) [7,8] | Υ | |
| Concomitant Medications (non-ART) | <b>Y</b> [9] | |
| Concomitant Antiretroviral Medications During Maintenance Phase | | Y |
| ART Medications Received During LTFU Phase | | Y |
| Lipid Modifying Agents (Baseline and During Maintenance Phase) | Y | |
| Substance use | Υ | |
| Medical History of Seizure | | Y |
| Other | | |
| Extent of Exposure to IP <sup>[10]</sup> | Υ | |
| Adherence to Injection Dosing Schedule for CAB/RPV <sup>[10]</sup> | Υ | |

#### NOTES:

- T = Tables, L = Listings, Y = Display Generated,
- 1. All Participants Enrolled population
- 2. Listing of planned and actual treatment.
- 3. All Participants Screened population.
- 4. Subjects who have not been recorded as either completing or withdrawing from the study will be categorized as "Ongoing at time of the analysis" for summary purposes.
- 5. Analysis of subject disposition will be performed for each study phase separately, as well as for overall study conclusion.
- 6. The five high level FDA race categories and designated Asian subcategories will be summarised along with all combinations of high level categories which exist in the data. The nine race categories collected will be summarised along with categories for mixed race. A by-subject listing of race will also be produced.
- 7. Medical conditions will be coded using the Medical Dictionary for Regulatory Activities (MedDRA).
- 8. Sub conditions are Cardiovascular, Gastrointestinal, Metabolism and Nutrition, Psychiatric, Renal and Urinary, Nervous System Conditions and Hepatobiliary
- 9. Summarised by Ingredient ATC Level 1, Ingredient combinations and Combination term ATC Level 1 (EG Includes single-ingredient medications with multi-ingredient medications labeled according to the sum of their ingredients, e.g., "TYLENOL Cold and Flu" would appear as "CHLORPHENAMINE MALEATE + DEXTROMETHORPHAN HYDROBROMIDE + PARACETAMOL + PSEUDOEPHEDRINE HYDROCHLORIDE" under the ATC headings for "Nervous System" and "Respiratory System" (the combination's ATC classifications).)
- 10. Safety Population

#### 6.2. Prior and Concomitant Medications

Non-ART and/or ART Medications will be classified by categories shown in Table 2. The same medication may be classified by more than one category. For example, if the Non-ART medication was started prior to the Maintenance treatment start date and was stopped at Month 6 while subject was still receiving study treatment, this medication would be considered both 'prior' and 'concomitant during maintenance'.

Table 2 Derived Data for Non-ART Medications/ART Medications

| | Definition |
|---|---|
| Prior | ART Medication Taken ≤ Maintenance Treatment Start Date |
| | Non-ART Medication Taken < Maintenance Treatment Start Date |
| Concomitant during | Maintenance Treatment Start Date ≤ Non-ART Medication Taken < LTFU |
| Maintenance | ART Start Date |
| | Maintenance Treatment Start Date < ART Medication Taken < LTFU ART |
| | Start Date |
| Received during | For subjects Who received at least one CAB and/or RPV injection and |
| Long-term Follow-up | have started LTFU ART: |
| | Non-ART/ART Medication Taken ≥ LTFU ART Start Date |

#### NOTES:

- Please refer to Appendix 7: Reporting Standards for Missing Data for handling of missing and partial dates for medications. Use the rules in this table if medication date is completely missing.
- If subjects have missing LFTU ART start date, only the lower bound will be considered in the derivation.

#### 7. EFFICACY ANALYSES

# 7.1. Primary Efficacy Analyses

No formal statistical analysis will be performed for the primary endpoint of the study.

#### 7.1.1. Endpoint / Variables

Proportion of participants with plasma HIV-1 RNA  $\geq$  50 copies/mL as per Food and Drug Administration (FDA) Snapshot algorithm at Month 12.

#### 7.1.2. Summary Measure

Number of subjects and percentage of participants with HIV-1 RNA ≥50 c/mL at Month 12 (defined by the US FDA snapshot algorithm) will be provided by treatment group.

#### 7.1.3. Population of Interest

The primary efficacy results will be based on the Intent-To-Treat Exposed population, unless otherwise specified.

#### 7.1.4. Strategy for Intercurrent (Post-treatment selection) Events

As defined by the Snapshot algorithm, HIV-1 RNA  $\geq$  50 c/mL is determined by the last available HIV-1 RNA measurement while the participant is on treatment within the analysis visit window of interest.

Participants without on-treatment HIV-1 RNA data for the visit of interest and who discontinue treatment for reasons not related to adverse event while having HIV-1 RNA  $\geq$  50 c/mL at time of discontinuation or who change study treatment not permitted per protocol before the analysis window are classified as having HIV-1 RNA  $\geq$  50 c/mL.

Full details of the snapshot algorithm are defined in Appendix 9: Snapshot Algorithm Details.

#### 7.1.5. Statistical Analyses / Methods

Details of the planned displays are provided in Appendix 12: List of Data Displays and will be based on GSK data standards and statistical principles.

Unless otherwise specified, endpoints / variables defined in Section 7.1.1 will be summarised using descriptive statistics, graphically presented (where appropriate) and listed.

#### 7.2. Secondary Efficacy Analyses

#### 7.2.1. Endpoint / Variables

The secondary efficacy endpoints for the study are listed below:

- Proportion of participants with plasma HIV-1 RNA <50 c/mL (c/mL) at Month 12 using the FDA Snapshot algorithm
- Proportion of participants with protocol-defined confirmed virologic failure (CVF) over time
- Proportion of participants with HIV-1 RNA  $\geq$  50 c/mL as per FDA Snapshot algorithm over time
- Absolute values and changes from Baseline in viral load and cluster of differentiation 4 (CD4+) cell counts over time

#### 7.2.2. Summary Measure

Number of subjects and percentage of participants with HIV-1 RNA < 50 c/mL at Month 12 (defined by the US FDA snapshot algorithm) will be presented by treatment group.

Number of subjects and percentage of participants with protocol-defined confirmed virologic failure (CVF) will be presented by treatment group and by visit.

Number of subjects and percentage of participants with HIV-1 RNA  $\geq$  50 c/mL (defined by the US FDA snapshot algorithm) will be presented by treatment group and by visit.

Descriptive statistics of the absolute values and changes from Baseline in viral load and cluster of differentiation 4 (CD4+) cell counts will be presented by treatment group and by visit.

#### 7.2.3. Population of Interest

The secondary efficacy analyses will be based on the Intent-to-Treat Exposed population, unless otherwise specified.

## 7.2.4. Strategy for Intercurrent (Post-treatment selection) Events

As defined by the snapshot algorithm, participants with last available HIV-1 RNA measurement < 50 c/mL while the participant is on treatment within the analysis visit window of interest are classified as HIV-1 RNA < 50 c/mL.

Participants without on-treatment HIV-1 RNA data for the visit of interest and who discontinue treatment for reasons not related to adverse event while having HIV-1 RNA  $\geq$  50 c/mL at time of discontinuation or who change study treatment not permitted per protocol before the analysis window are classified as having HIV-1 RNA  $\geq$  50 c/mL.

#### 7.2.5. Statistical Analyses / Methods

Details of the planned displays are provided in Appendix 12: List of Data Displays and will be based on GSK data standards and statistical principles.

Unless otherwise specified, endpoints / variables defined in Section 7.2.1 will be summarised using descriptive statistics, graphically presented (where appropriate) and listed.

# 7.3. Exploratory Efficacy Analyses

Table 3 provides an overview of the planned exploratory efficacy analyses. Details of the planned displays are provided in Appendix 12: List of Data Displays and will be based on GSK data standards and statistical principles. The exploratory efficacy analyses will be based on the Intent-to-Treat Exposed population, unless otherwise specified.

Table 3 Overview of Exploratory Efficacy Analyses

| | Absolute | | | Change from Baseline | | | | |
|---|---|---|---|---|---|---|---|---|
| Endpoints | Summary | | Individual | | Summary | | Individual | |
| | Т | F | F | L | Т | F | F | Г |
| Plasma HIV-1 RNA over ti | me | | | | | | | |
| By visit | <b>Y</b> [1] | | <b>Y</b> [2] | <b>Y</b> [3] | Y[1] | | | <b>Y</b> [3] |
| Target Detected vs | | | | | | | | |
| Target Not Detected by | Υ | | | <b>Y</b> [5] | | | | |
| visit [4] | | | | | | | | |
| Confirmed Virologic Failu | re (CVF) | ) | | | | | | |
| CVF overall | Υ | | | | | | | |
| Plasma HIV-1 RNA at | | | | | | | | |
| time of suspected and | Υ | | | | | | | |
| confirmed virologic failure | | | | | | | | |
| CD4+ cell counts over time | ne | | | | | | | |
| Observed <sup>[6]</sup> | Υ | | | | Υ | | | |
| HIV-1 conditions and dise | ase pro | gression | 1 | | | | | |
| HIV Conditions | | | | | | | | |
| including/excluding | Υ | | | Υ | | | | |
| Recurrences as recorded | Ī | | | I | | | | |
| in eCRF | | | | | | | | |
| HIV Disease | Υ | | | | | | | |
| Progressions <sup>[7]</sup> | 1 | | | | | | | |

#### NOTES:

- T = Table, F = Figure, L = Listing, Y = Yes display generated.
- Summary = Represents TF related to any summaries (i.e. descriptive statistics) of data.
- Individual = Represents FL related to any displays of individual participant's data.
- 1. Using log10 transformed values.
- 2. Individual plasma HIV-1 RNA only for participants who are in the category of 'viral load ≥50 c/mL' at Month 12 per Snapshot algorithm or who are CVF participants. The figures will display all HIV-1 RNA values collected.
- 3. For CVF participant and, participants with viral load ≥ 50 c/mL during the Maintenance Phase.
- 4. See Section 12.6.3 for definition of "Target Detected" and "Target Not Detected", and for the specification of corresponding summary table.
- 5. Target Detected" and "Target Not Detected" are included in the listing for plasma HIV-1 RNA by visit.
- 6. Using available data without imputation for missing values.
- 7. See Section 12.6.3 for HIV disease progressions.

#### 8. SAFETY ANALYSES

The safety analyses will be based on the Safety population, unless otherwise specified.

#### 8.1. Adverse Events Analyses

Adverse events analyses including the analysis of adverse events (AEs), Serious (SAEs) and other significant AEs will be based on GSK Core Data Standards. The details of the planned displays are provided in Appendix 12: List of Data Displays.

#### 8.1.1. Injection Site Reactions

For the summary of Injection Site Reaction Adverse Events by Visit and Maximum Severity (Overall and by Common ISRs): ISRs will be assigned based on onset date to the most recent planned IM injection visit prior or equal to the AE onset date.

Maximum grade at each visit will be derived as the maximum grade among ISRs assigned to the particular visit, with consideration for whether the summary applies to a particular preferred term (vs. across preferred terms), or drug-related associated to CAB and/or RPV, or stratification by needle length (refer to Section 5.4.2).

Drug-related ISRs (based on investigator discretion) will be attributed to the causal agent (CAB vs. RPV) when this can be determined specifically based the side of injection administration and the side of the reported ISR (as collected in the eCRF). If we are unable to determine the causal agent in those cases where both drugs are given on one side and the ISR is reported non-specifically, then the attribution to a specific causal agent will remain unknown.

Common study drug ISR adverse events are defined by MedDRA preferred terms including injection site pain, injection site induration, injection site nodules and preferred terms of any other ISR with  $\geq$ 5% participants in the CAB LA + RPV LA arm, coming from study drug injections. The same set of common terms will be applied to 'overall' (CAB and/or RPV), CAB alone, RPV alone.

ISRs will be attributed to the needle length ( $\leq 1.5$ , > 1.5 to < 2,  $\geq 2$  inches) when this can be determined specifically based on the side of injection administration and the side of the reported ISR (as collected in the eCRF). If we are unable to determine the needle length in those events where both drugs are given on one side and their needle lengths are different, then the attribution to a needle length will remain unknown.

# 8.2. Clinical Laboratory Analyses

Laboratory evaluations including the analyses of chemistry laboratory tests, hematology laboratory tests, urinalysis, and liver function tests will be based on GSK Core Data Standards. The details of the planned displays are in Appendix 12: List of Data Displays.

#### 8.3. Adverse Events of Special Interest Analyses

Adverse events of special interest (AESI) are determined for CAB and/or RPV based on pre-clinical and clinical experience, along with information for the Integrase Inhibitor class of HIV medications and RPV safety profile. Table 4 shows the currently identified AESI, drug(s) of Interest and the reasons for inclusion. Changes to the MedDRA dictionary may occur between the start of the study and the time of reporting, and/or emerging data from on-going studies may highlight additional adverse events of special interest, therefore the list of AESIs may change at the time of reporting.

A summary by system organ class and preferred term will be provided for each of AESI. For Depression, anxiety and suicidal ideation/behaviour AESI, a summary by system organ class, maximum DAIDS toxicity grade and prior history will be provided. The details of the planned grouping and planned displays are provided in Section 12.10 and Appendix 12: List of Data Displays.

Table 4 Adverse Events of Special Interest

| Adverse Events of Special Interest | Drug(s) of Interest | Reason for Inclusion |
|---|---|---|
| Hepatic Safety Profile: Assessment of Risk of hepatoxicity | CAB+RPV | Clinical, Class, Regulatory<br>Interest, More prevalent in<br>HIV population |
| Hypersensitivity Reactions (HSR) | САВ | Class, Regulatory Interest,<br>Occurs in HIV population |
| Rash | RPV | Class, Regulatory Interest,<br>Occurs in HIV population |
| Prolongation of the Corrected QT Interval of the ECG in Supratherapeutic Doses | RPV | Non-clinical, Clinical,<br>Regulatory Interest |
| Suicidal Ideation/Behaviour | CAB+RPV | Clinical, Class, Regulatory<br>Interest, More prevalent in<br>HIV population |
| Depression | CAB+RPV | Clinical, Class, Regulatory<br>Interest, More prevalent in<br>HIV population |
| Bipolar Disorder | CAB+RPV | Clinical, Class, Regulatory<br>Interest, More prevalent in<br>HIV population |
| Psychosis | CAB+RPV | Clinical, Class, Regulatory<br>Interest, More prevalent in<br>HIV population |

| Adverse Events of Special Interest | Drug(s) of Interest | Reason for Inclusion |
|---|---|---|
| Mood Disorders | CAB+RPV | Clinical, Class, Regulatory<br>Interest |
| Anxiety | CAB+RPV | Clinical, Class, Regulatory<br>Interest |
| Sleep Disorders | CAB+RPV | Clinical, Class, Regulatory<br>Interest, More prevalent in<br>HIV population |
| Injection Site Reactions (ISR) from Study Drug Injections [1] | CAB+RPV | Clinical |
| Seizures and Seizure-like Events | CAB | Clinical, Regulatory Interest |
| Weight Gain | CAB | Clinical, Class |
| Rhabdomyolysis | CAB | Clinical, Class |
| Pancreatitis | CAB | More prevalent in HIV population |
| Impact on Creatinine | CAB+RPV | Regulatory Interest,<br>Therapeutic Area, More<br>prevalent in HIV population |
| Safety in Pregnancy | CAB | Regulatory Interest, Class |

#### NOTE:

# 8.4. Other Safety Analyses

The analyses of non-laboratory safety test results including ECGs and vital signs will be based on GSK Core Data Standards, unless otherwise specified. The details of the planned displays are presented in Appendix 12: List of Data Displays.

ECG values of potential clinical importance are defined as a QTc of > 500 msec or increase from baseline in QTc  $\ge 60$  msec.

## 9. HEALTH OUTCOMES ANALYSES

# 9.1. Endpoint / Variables

- Change from Baseline (Day 1) in HIVDQoL at Months 6 and 12 (or Withdrawal)
- Change from baseline (Day 1) in total "treatment satisfaction" score, and individual item scores of the HIV Treatment Satisfaction Status Questionnaire (HIVTSQs) at Months 6 and 12 (or Withdrawal)

<sup>1.</sup> A separate analysis will be performed for ISRs from study drug injections as described in Section 8.1.1.

- Change in treatment satisfaction over time using the HIV Treatment Satisfaction Change Questionnaire HIVTSQc at Month 12 (or Withdrawal).
- Preference between injections of LA HIV treatment and daily oral HIV treatment at Month 12. This is an exploratory endpoint.
- Reasons for switching to injectable HIV treatment at Baseline (Day 1). This is an exploratory endpoint.

# 9.2. Summary Measure

Summary statistics of the above endpoints will be presented by treatment group.

#### 9.3. Population of Interest

The health outcomes outputs will be based on the Intent-to-Treat Exposed population, unless otherwise specified.

# 9.4. Strategy for Intercurrent (Post-treatment selection) Events

No imputations would be performed for any missing data.

#### 9.5. Statistical Analyses / Methods

Details of the planned displays are provided in Appendix 12: List of Data Displays and will be based on GSK Data Standards and statistical principles.

Unless otherwise specified, endpoints / variables defined in Section 9.1 will be

summarised using descriptive statistics, graphically presented (where appropriate) and listed.

#### 10. VIROLOGY

The virology analyses will mainly use genotype and phenotype data based on plasma sample for CVF population, unless otherwise specified. Additional analyses for HIV-1 resistance may be carried out on peripheral blood mononuclear (PBMC) samples collected at Day 1 or Withdrawal.

If pre-treatment genotypic/phenotypic results are available from both the central laboratory and Monogram Biosciences, then Baseline genotype/phenotype will be determined based only upon the data provided by Monogram assays.

Table 5 Overview of Planned Virology Analyses

| | | Absolute | | |
|---|---|---|---|---|
| Endpoints | Sun | nmary | Individual | |
| | Т | F | F | L |
| Genotypic resistance at time of CVF <sup>[1]</sup> | · | | | |
| Prevalence of Resistance Mutations | Y[2] | | | Υ |
| Prevalence of Genotypic Susceptibility | Y | | | |
| Phenotypic resistance at time of CVF <sup>[1]</sup> | <u>.</u> | • | • | • |
| Prevalence of Phenotype | Y[3] | | | Υ |

| | Absolute | | | |
|---|---|---|---|---|
| Endpoints | Sum | mary | Individual | |
| | T | F | F | L |
| Fold Change to CAB and RPV | Υ | | | <b>Y</b> [4] |
| IN, PR/RT Replication Capacity | | | | Υ |
| Other | | | | |
| Viral load, Genotypic and Phenotypic data for | | | | |
| Participants with genotype and/or phenotype data | | | | <b>Y</b> [4] |
| for CVF participants | | | | |
| Net Assessment | Υ | | | |

#### NOTES:

- T = Table, F = Figure, L = Listing, Y = Yes display generated.
- Summary = Represents TF related to any summaries (i.e. descriptive statistics) of the observed raw data.
- Individual = Represents FL related to any displays of individual participant observed raw data.
- 1. For the CVF as indicated by two consecutive plasma HIV-1 RNA levels ≥200 c/mL after prior suppression to <200 c/mL, the first visit of these two consecutive visits is defined as 'the suspected visit', and the 2nd one is the confirmed visit. Sample used for resistance testing is taken at the suspected visit, and only tested once a participant confirms virological failure at a subsequent visit. If the test fails with the sample at the suspected visit, we will just report it as 'no data'. The sample from the confirmed visit may be used for exploratory analyses.</p>
- No. and percentage of participants with IN resistance mutations or major mutations in the classes of NNRTI, NRTI, PI, respectively, as defined in Section 12.6.6.
- 3. Separate outputs by phenotypic susceptibility and by number of drugs to which participants are phenotypic resistant or partial sensitive or sensitive.
- 4. Fold change to CAB and RPV will be included in the listing for viral load, genotypic and phenotypic data for participants with genotype and/or phenotype data for CVF and non-CVF participants.

#### 11. REFERENCES

- Grundy S.M., et al. Executive summary of the third report of the National Cholesterol Education Program (NCEP) Expert Panel on Detection, Evaluation and Treatment of High Blood Cholesterol in Adults (Adult Treatment Panel III). JAMA. 2001; 285 (19):2486-2497.
- HIVDQoL user guidelines, Health Psychology Research Unit, Royal Holloway, University of London, 2018
- HIVTSQ user guidelines, Health Psychology Research Unit, Royal Holloway, University of London, 2016
- Levey AI, Christopher HS, Hocine T, John HE, Harold IF, Tom G, et al. Estimating Glomerular Filtration Rate from Serum Creatinine and Cystatin C. N Engl J Med 2012, 367: 20-29.
- Wee HL, Tan CE, Goh SY, Li SC. Usefulness of the Audit of Diabetes-Dependent Quality-of-Life (ADDQoL) questionnaire in participants with diabetes in a multi-ethnic Asian country. *Pharmacoeconomics*. 2006;24(7):673-82.
- Wensing AM et al. 2019 Update of the Drug Resistance Mutations in HIV-1 Volume 27 Issue 3 July/August 2019

#### 12. APPENDICES

# 12.1. Appendix 1: Protocol Deviation Management and Definitions for Per Protocol Population

#### 12.1.1. Exclusions from Per Protocol Population

Important protocol deviations leading to exclusion from the Per Protocol population are those deviations which may

- i. directly impact the efficacy endpoint of HIV-1 RNA; or
- ii. lead to permanent discontinuation of IP/withdrawal and hence indirectly impact the efficacy endpoint by causing data to be missing.

The following criteria define the protocol deviations which, if they occur prior to an analysis timepoint of interest (e.g. Month 12), will lead to exclusion of a subject from the Per-Protocol population for that analysis. Potential protocol deviations leading to exclusion from PP population will be reviewed by the study team to confirm that they meet these criteria. A final review will occur before the clinical database has been frozen for analysis.

A subject meeting any of the following criteria will be excluded from the Per Protocol population based on case-by-case clinical determination:

| Number | Exclusion Description |
|---|---|
| 01 | Participant deviates from any inclusion or exclusion criteria that may significantly affect exposure, response to therapy or participant safety or that are fundamentally inconsistent with the intended study population, as recorded in the Protocol Deviation form in the eCRF based on study team review (where indicated in the PDMP as case-by-case determination). |
| 02 | Participant has maintenance phase non-compliance (including IM dosing errors) with investigational product up to an analysis timepoint of interest, meeting one of the following conditions: 1. Month 12 analysis only: • Q2M arm: two or more injection intervals affected by over dosage deviations (e.g. extra injection or excessive volume administered, length of time between injections less than 7 weeks, excluding split doses). 2. ≥10% of total time on-treatment with under dosing deviations. The percentage of total time on-treatment with under dosing deviations will be calculated by (the total number of non-compliant dosing days / the total number of intended exposure days) * 100%. Number of Intended Exposure Days = Date of Last Viral Load – Start Date of Study Treatment + 1, where the last viral load refers to the last on-treatment viral load up to Study Day 360 for Q2M arm and study day of last nominal Month 12 visit for DTG + RPV arm during maintenance phase for Month 12 analysis. |

| Number | Exclusion Description |
|---|---|
| | The total number of non-compliant dosing days up to the analysis timepoint visit (or date of IP discontinuation/withdrawal, whichever is earlier), is derived as follows (summing across all instances): • Q2M arm: |
| | <ul> <li>Length of time (in days) until next injection from date of dosage deviation (e.g. 2 mL administered instead of 3 mL).</li> <li>Length of time (in days) in excess beyond 67 days between injections.</li> <li>Length of time (in days) in excess beyond 67 days from last injection until start of oral bridging post Month 4.</li> <li>Interrupted days in oral bridging if the oral dose has been interrupted for 3 or more consecutive days and the primary interruption reason is not adverse event or laboratory abnormality (based on the eCRF Exposure forms). 3 days will be assumed if such interrupted days are not available in the database.</li> <li>DTG + RPV arm: Durations of interruptions for reasons other than</li> </ul> |
| | treatment-related adverse events or laboratory abnormalities (based on Exposure eCRF forms). |
| 03 | Prohibited medications: receiving ART medication other than that prescribed/allowed by the study (excluding permanent changes in ART regimen; such cases will be retained as 'HIV1-RNA ≥50 c/mL' in the per protocol snapshot analysis) or receiving prohibited concomitant medication that would impact exposure or response to therapy with duration and route of administration taken into consideration, as recorded in the Protocol Deviation form in the eCRF based on study team review (where indicated in the PDMP as case-by-case determination). |
| 04 | Permanent discontinuation of IP/withdrawal due to a reason of "Protocol Deviation" (as recorded in the eCRF). |
| 05 | Other important protocol deviations that exclude Participant from Per protocol population as recorded in the Protocol Deviation form in the eCRF based on study team review (where indicated in the PDMP as case-by-case determination). |

# 12.2. Appendix 2: Schedule of Activities

## 12.2.1. Protocol Defined Schedule of Events for CAB LA + RPV LA Q2M Administration

| Procedures Q2M | a | | | | | | ı | Vionth | | | | | | | E |
|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|
| | Day 1 a | 2 º | 4 | 6 | 8 | 10 | 12 | 14 | 16 | 18 | 20b | <b>22</b> <sup>b</sup> | 24 | 26 | WD t. m |
| Written Informed Consent | Х | | | | | | | | | | | | | | |
| Demography | Х | | | | | | | | | | | | | | |
| Eligibility Verification | Х | | | | | | | | | | | | | | |
| Physical Exam | Х | | | | | | | | | | | | | | |
| Medical History | Х | | | | | | | | | | | | | | |
| Center for Disease Control and Prevention (CDC) Classification | Х | | | | | | | | | | | | | | |
| Rapid Plasma Reagin (RPR) | Х | | | | | | | | | | | | | | |
| Symptom Directed Physical<br>Exam, injection site reaction<br>(ISR) and Medical<br>Assessment <sup>c</sup> | Х | Х | Х | Х | Х | Х | Х | Х | Х | Х | Х | Х | Х | Х | Х |
| Vital Signs<br>(blood pressure [BP], heart<br>rate [HR]) <sup>d</sup> | Х | Х | X | | Х | | Х | | Х | | Х | | Х | | Х |

| Procedures Q2M | æ | | | | | | l | Vonth | | | | | | | F |
|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|
| | Day 1 ª | 2 º | 4 | 6 | 8 | 10 | 12 | 14 | 16 | 18 | 20b | 22 <sup>b</sup> | 24 | 26 | WD 'r m |
| Weight, Height & body mass index (BMI)e | Х | Х | Х | | Х | | Х | | Х | | Х | | Х | | Х |
| HIV Associated Conditions,<br>AE and serious adverse<br>event (SAE) Assessments,<br>Con Meds | Х | Х | Х | Х | Х | Х | Х | Х | X | Х | Х | Х | Х | Х | Х |
| 12-Lead electrocardiogram (ECG) <sup>f</sup> | Х | | | | | | Х | | | | | | | | Х |
| Clinical Chemistry and<br>Hematology | Х | Х | Х | | Х | | Х | | Х | | Х | | Х | | Х |
| Pregnancy Testing (U)rine or (S)erum <sup>g</sup> | U | U | U | U | U | U | U | U | U | U | U | U | U | U | U |
| HIV-1 RNA and sample for storage <sup>h</sup> | Х | Х | Х | Х | Х | Х | Х | Х | Х | Х | Х | Х | Х | Х | Х |
| CD4+ | Х | Х | Х | | Х | | Х | | Х | | Х | | Х | | Х |
| Urinalysis | Х | | | | | | | | | | | | | | Х |

| Procedures Q2M | В | | | | | | ı | Month | | | | | | | _ |
|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|
| | Day 1 ª | 2 ° | 4 | 6 | 8 | 10 | 12 | 14 | 16 | 18 | 20b | <b>22</b> b | 24 | 26 | WD i, m |
| Fasting Glucose,<br>Cholesterol (Total, high<br>density lipoprotein [HDL]<br>and low density lipoprotein<br>[LDL]) and Triglycerides i | X | | | | | | X | | | | | | Х | | Х |
| Prothrombin time (PT)/<br>partial thromboplastin time<br>(PTT)/international<br>normalized ratio (INR) | X | | | | | | | | | | | | | | Х |
| PK Diary<br>(D)ispensation and (R)eview | R | | | | | | | | | | | | | | |
| PK Sample (S)torage <sup>j</sup> | S | | | | | | S | | | | | | | | S |
| LA Study Intervention<br>Administration <sup>k</sup> | Х | Х | Х | Х | Х | Х | Х | Х | Х | Х | Х | Х | Х | Х | |
| HIVTSQc | | | | | | | Χ | | | | | | | | Х |
| HIVTSQs | Х | | | Х | | | Χ | | | | | | | | Х |
| HIVDQoL | Х | | | Х | | | Х | | | | | | | | Х |
| Preference | | | | | | | Х | | | | | | | | |
| Reason for Switch | Х | | | | | | | | | | | | | | |

| Procedures Q2M | R | | Month | | | | | | | | | E | | | |
|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|
| | Day 1 | 2 º | 4 | 6 | 8 | 10 | 12 | 14 | 16 | 18 | 20b | 22 <sup>b</sup> | 24 | 26 | WD to |
| Participant Visit Reminder<br>Contact | Х | Х | Х | Х | Х | Х | Х | Х | Х | Х | Х | Х | Х | Х | |
| Participant Contact Detail<br>Confirmation | Х | Х | Х | Х | Х | Х | Х | Х | Х | Х | Х | Х | Х | Х | |

See footnote "b" for continuation of visit schedule after Month 26. Continue until either locally approved and commercially available, the participant no longer derives clinical benefit or meets a protocol-defined reason for discontinuation or until development is terminated.

- a. The Day 1 visit will take place during Week 312 (or Week 324 in the event of unavoidable delays) of the LATTE study, the participant's last week on study. LATTE participants eligible for POLAR study dosing will take final dose of CAB 30 mg + RPV 25 mg in the clinic within 2 hours of the Q2M IM regimen. For IM dosing administration loading doses are required. (Day 1=1st loading dose; Month 2=2nd loading dose)
- b. Continue this pattern for visits for the remainder of the study. For example, Month 28 will be conducted just like Month 20, Month 30 will be conducted just like Month 22 and so on.
- c. Physical exams should be conducted as part of normal routine clinical care but data will not be collected in the electronic case report form (eCRF). Medical assessments include any decisions the study staff must make for participant management.
- d. Measure vital signs after about 5 minutes of rest in a semi-supine position.
- e. Height collected at Day 1 only.
- f. On Day 1, ECGs should be performed in triplicate at least 5 minutes apart and following 5 minutes of rest in a semi-supine position within 1 hour prior to first dose. Also on Day 1, a 2-hour post dose ECG will be performed for all participants. The 2-hour post dose ECG on Day 1 can also be used for the LATTE Week 312 (or Week 324, if needed) visit. ECG evaluations at other visits should be obtained after dosing, preferably 2-4 hours post dosing.
- g. A (-) urine pregnancy test is required prior to any injection and as required by medical monitor after a treatment interruption. A (+) urine test should be confirmed with a stat serum test. If (+), participant will need to be withdrawn.
- h. Plasma for storage samples are collected for possible future analyses, back-up in cases of loss/damage in transit and geno/pheno analyses for virologic failures.
- i. Fast overnight; however, a minimum of a 6 hour fast is acceptable.
- Take PK samples pre-dose.
- k. Q2M Injections are 1 x CAB LA 600 mg IM + 1 x RPV LA 900 mg IM. If possible, injections should be spaced approximately 2 cm from one another and from the site of any previous injection and or any injection site reaction. Bring RPV LA to approximately room temperature prior to injecting. Time and location of injection (right or left) as well as needle length used will be collected in the eCRF. IM dosing is expected to occur during the month in which the participant's projected visit falls (as according to the Day 1 visit). An additional (+ or -) 7day window from date of projected visit is stipulated for IM dosing. All decisions regarding dose interruption/ resumption must be discussed with the medical monitor in advance.

#### 12.2.2. Protocol Defined Schedule of Events for DTG + RPV Administration

| Procedures for DTG+RPV | Day 1 a | Month 3 | Month 6 | Month 9 | Month 12 | WD j | Notes |
|---|---|---|---|---|---|---|---|
| Written Informed Consent | Х | | | | | | a. The Day 1 visit will take place during Week 312 (or Week 324 in the event of unavoidable delays) of the LATTE study, the |
| Demography | Х | | | | | | participant's last week on study. LATTE participants eligible for POLAR study dosing will take final dose of CAB 30 mg + RPV 25 |
| Eligibility Verification | Х | | | | | | mg in the clinic. See Section 6.2 of the protocol for dosing administration. b. Physical exams should be conducted as part of normal routine |
| Physical Exam | Х | | | | | | clinical care but data will not be collected in the eCRF. Medical assessments include any decisions the study staff must make for |
| Medical History | Х | | | | | | participant management. c. Measure vital signs after about 5 minutes of rest in a semi-supine |
| CDC Classification | Х | | | | | | position. d. Height collected at Day 1 only. |
| RPR | Х | | | | | | e. On Day 1, ECGs should be performed in triplicate at least 5 minutes apart and following 5 minutes of rest in a semi-supine position within 1 hour prior to first dose. Also on Day 1, a 2-hour |
| Symptom Directed Physical Exam and Medical Assessment <sup>b</sup> | | Х | Х | Х | Х | Х | post dose ECG will be performed for all participants. The 2-hour post dose ECG on Day 1 can also be used for the LATTE Week 312 (or Week 324, if needed) visit. ECG evaluations at other |
| Vital Signs(BP, HR) ° | Х | Х | Х | Х | Х | Х | visits should be obtained after dosing, preferably 2-4 hours post dosing. |
| Weight, Height & BMI d | Х | Х | Х | Х | Х | Х | f. Plasma for storage samples are collected for possible future analyses, back-up in cases of loss/damage in transit and geno/pheno analyses for virologic failures. |
| HIV Associated Conditions, AE and SAE Assessments, Con Meds | Х | Х | Х | Х | Х | Х | g. A (-) urine pregnancy test is required prior to any administration of drug and as required by medical monitor after a treatment interruption. A (+) urine test should be confirmed with a stat |

I. Or Long-Term Follow Up

m. Follow Up Visit - Conduct ~4 weeks after the last dose of investigational product (IP) if not entering Long-Term Follow Up and only if the participant has ongoing AEs or lab abnormalities at the last on-study visit. May be conducted by telephone.

| Procedures for DTG+RPV | Day 1 a | Month 3 | Month 6 | Month 9 | Month 12 | WD j | Notes |
|---|---|---|---|---|---|---|---|
| 12-Lead ECG ° | Х | | | | Х | Х | serum test. If (+), participant will need to be WD. h. Fast overnight; however, a minimum of a 6 hour fast is |
| HIV-1 RNA | Х | Х | Х | Х | Х | Χ | acceptable. i. DTG 50 mg + RPV 25 mg. Administer daily with food |
| CD4+ | Х | Х | Х | Х | Х | Х | j. Follow Up Visit - Conduct ~4 weeks after the last dose of IP and only if the participant has ongoing AEs or lab abnormalities at the last on-study visit. May be conducted by telephone. |
| Plasma for Storage <sup>f</sup> | Х | Х | Х | Х | Х | Х | |
| PK Sample for Storage | | | | | | S | |
| Clinical Chemistry and Hematology | Х | Х | X | Х | X | Х | |
| Pregnancy Testing <sup>g</sup> | U | U | U | U | U | U | |
| Urinalysis | Х | | | | | Χ | |
| Fasting: Glucose, Cholesterol (Total, HDL and LDL) and Triglycerides h | Х | | | | | Х | |
| PT/PTT/INR | Х | | | | | Х | |
| HIVTSQc | | | | | Х | Х | |
| HIVTSQs | Х | | Х | | Х | Х | |
| HIVDQoL | Х | | Х | | Х | Х | |
| Participant Visit Reminder Contact | Х | Х | Х | Х | Х | | |
| Participant Contact Detail Confirmation | Х | Х | Х | Х | Х | | |

| Procedures for DTG+RPV | Day 1 a | Month 3 | Month 6 | Month 9 | Month 12 | <b>WD</b> i | Notes |
|---|---|---|---|---|---|---|---|
| Study Treatment Dispensation i | Х | Х | Х | Х | Х | | |

# 12.2.3. Protocol Defined Schedule of Events for Long Term Follow Up

| Procedures for Long-Term Follow Up | Month 1 a | Month<br>3 | Month<br>6 | Month<br>9 | Month 12 | WD | Notes |
|---|---|---|---|---|---|---|---|
| HIV Associated Conditions, AE and SAE<br>Assessments, Con Meds | Х | Х | Х | Х | Х | Х | Every effort should be made to enter participants into the Long-<br>Term Follow Up if they withdraw from or discontinue the study after |
| HIV-1 RNA | Х | Х | Х | Х | Х | Х | <ul><li>receiving at least one dose of CAB LA and / or RPV LA.</li><li>a. The start of the 52-week follow up period begins the day of the</li></ul> |
| CD4+ | Х | Х | Х | Х | Х | Х | last CAB LA and/or RPV LA dose. b. Women of childbearing potential only. S = Serum |
| Plasma for Storage | X | Х | Х | Х | Х | Χ | c. Fast overnight; however, a minimum of a 6 hour fast is acceptable. |
| PK Sample for Storage | S | S | S | S | S | S | d. Women of childbearing potential should continue to receive counselling on the need to use adequate contraception for the |
| Clinical Chemistry and Hematology | X | Х | Х | Х | X | X | entirety of the Long-Term Follow-Up Period. e. Investigators must discuss choice of HAART regimen and |
| Pregnancy Testing b | S | S | S | S | S | S | timing of initiation with the medical monitor before initiating. This regimen may be supplied regionally by GlaxoSmithKline |
| Urinalysis | Х | | | | Х | Х | (GSK) or reimbursement will be provided. |
| Fasting: Glucose, Cholesterol (Total, HDL and LDL) and Triglycerides ° | | | | | X | Х | |
| PT/PTT/INR | | | | | Х | Х | |

| Procedures for Long-Term Follow Up | Month 1 a | Month<br>3 | Month<br>6 | Month<br>9 | Month 12 | WD | Notes |
|---|---|---|---|---|---|---|---|
| Contraception Counselling d | Х | Х | Х | Х | Х | Х | |
| HAART Dispensation e | Х | Х | Х | Х | Х | Х | |
## 12.3. Appendix 3: Assessment Windows

## 12.3.1. Definitions of Assessment Windows for Analyses

Laboratory data, vital signs, ECGs, health outcomes assessments, and genotypic/phenotypic data will be assigned to assessment windows according to actual dates rather than the nominal visit labels as recorded on the eCRF or in the laboratory database.

In most cases the window around an assessment will include all dates from the midpoints between the target day and that of the previous and the proceeding visits. In general, the nominal target study day for Month m is ((m-1)\*30)+1 for Q2M and (m\*30)+1 for DTG + RPV.

For parameters which are not scheduled to be assessed at particular visits, the all-inclusive assessment windows will still be used; however, data summaries will only report scheduled visits. Assessments at unscheduled visits will be included for 'any time On-treatment' time points and in data listings, as well any algorithms that make use of additional data (e.g., Snapshot).

Prior to visit slotting, assessments are first assigned to a study phase (maintenance, and Long Term Follow Up) based on the Tables in Section 12.4.1 and treatment state based on Section 12.4.2.

Maintenance phase assessments other than health outcomes are assigned based on Maintenance Phase Study Day, as shown in Table 6, Table 7, Table 8 and Table 9. The analysis visits from Month 2 to Month 12 and so on should be only applied to the assessments that are already assigned to Maintenance phase (on-treatment).

Long-term Follow-up phase assessments are assigned based on the LTFU study day as shown in Table 10. The analysis visits in LTFU should be only applied to the assessments that are already assigned to LTFU phase regardless of treatment state. See Section 12.6.1 for derivation of Maintenance and LTFU Study Day.

## 12.3.2. Definitions of Assessment Windows for Data Other than Health Outcomes

Table 6 Assessment Windows for Screening and Maintenance Phase Data for CAB LA + RPV LA arm

| All Parameters<br>(except for<br>where noted) | Target Study<br>Day | Analysis Window | Analysis<br>Timepoint |
|---|---|---|---|
| | 1 | Baseline information to be collected at nominal visit Day 1 which is the last available recorded value up to and including the Maintenance treatment start | Baseline |

| All Parameters<br>(except for<br>where noted) | Target Study<br>Day | Analysis Window | Analysis<br>Timepoint |
|---|---|---|---|
| | | date, excluding 2-hour post-dose<br>ECG taken on the Maintenance<br>treatment start date | |
| | 1 | Date of first maintenance dose of IP+ | Day 1 |
| | 31 | 2 ≤ Study Day ≤ 60 | Month 2* |
| | 91 | 61 ≤ Study Day ≤ 120 | Month 4 |
| | 151 | 121 ≤ Study Day ≤ 180 | Month 6 |
| | 211 | 181 ≤ Study Day ≤ 240 | Month 8 |
| | 271 | 241 ≤ Study Day ≤ 300 | Month 10 |
| | 331 | 301 ≤ Study Day ≤ 360 | Month 12 |
| | 391 | 361 ≤ Study Day ≤ 420 | Month 14 |
| | 451 | 421 ≤ Study Day ≤ 480 | Month 16 |
| | 511 | 481 ≤ Study Day ≤ 540 | Month 18 |
| | 571 | 541 ≤ Study Day ≤ 600 | Month 20 |
| | 631 | 601 ≤ Study Day ≤ 660 | Month 22 |
| | 691 | 661 ≤ Study Day ≤ 720 | Month 24 |
| | 751 | 721 ≤ Study Day ≤ 780 | Month 26 |
| | (( <i>m</i> -1)*30)+1 | $(((m-1)*30)-29) \le \text{Study Day} \le (((m-1)*30)+30)$ | Month <i>m</i> , <i>m</i> =28, 30, |
| If a | participant perm | nanently discontinued study treatme | |
| NOTES | | Date > max (Date of Last Oral<br>Dose of CAB+RPV + 1, Date of<br>Last Injection + 67) | Follow-up# |

Table 7 Assessment Windows for Screening and Maintenance Phase Data for DTG + RPV arm

| All Parameters<br>(except for<br>where noted) | Target Study<br>Day | Analysis Window | Analysis<br>Timepoint |
|---|---|---|---|
| | 1 | Baseline information to be collected at nominal visit Day 1 which is the last available recorded value upto and including the Maintenance treatment start date, excluding 2-hour post-dose | Baseline |

<sup>+</sup> Only non-baseline records from the mentioned assessment window will be assigned to Day 1.

<sup>\*</sup> The second loading injections will be administered 1 month (Month 2 visit, start of the second month of the study) after initial loading dose (CAB LA 600 mg + RPV LA 900 mg), with subsequent injections (CAB LA 600 mg + RPV LA 900 mg) occurring every 2 months thereafter.

<sup>#</sup> Follow-up will be derived only for participants who permanently discontinued study treatment.

| All Parameters<br>(except for<br>where noted) | Target Study<br>Day | Analysis Window | Analysis<br>Timepoint |
|---|---|---|---|
| | | ECG taken on the Maintenance treatment start date | |
| | 1 | Date of first maintenance dose of IP+ | Day 1 |
| | 91 | 2 ≤ Study Day ≤ 135 | Month 3 |
| | 181 | 136 ≤ Study Day ≤ 225 | Month 6 |
| | 271 | 226 ≤ Study Day ≤ 315 | Month 9 |
| | 361 | 316 ≤ Study Day ≤ (Study Day of Nominal Month 12 visit) | Month 12 |
| If a | If a participant permanently discontinued study treatment: | | |
| | | Date > Date of Last Oral Dose of DTG + 1 | Follow-up# |

Table 8 Assessment Windows for Summary of Snapshot Data for CAB LA + RPV LA arm— Data assigned to Maintenance Phase Only

| Snapshot Ana | Analysis Timepoint | |
|---|---|---|
| (If no on-treatment viral load data | | |
| winc | , | |
| Default | Expanded +45 Day Upper<br>Window <sup>a</sup> | |
| Last available recorded value up to | Last available recorded value up to | Baseline |
| and including the date of first | and including the date of first | Daseille |
| Maintenance Phase dose of IP | Maintenance Phase dose of IP | |
| 2 ≤ Study Day ≤ 60 | 2 ≤ Study Day ≤ 75 | Month 2 |
| 61 ≤ Study Day ≤ 120 | 61 ≤ Study Day ≤ 135 | Month 4 |
| 121 ≤ Study Day ≤ 180 | 121 ≤ Study Day ≤ 195 | Month 6 |
| 181 ≤ Study Day ≤ 240 | 181 ≤ Study Day ≤ 255 | Month 8 |
| 241 ≤ Study Day ≤ 300 | 241 ≤ Study Day ≤ 315 | Month 10 |
| 285 ≤ Study Day ≤ 375 | 285 ≤ Study Day ≤ 375 | Month 12 |
| 361 ≤ Study Day ≤ 420 | 301 ≤ Study Day ≤ 435 | Month 14 |
| 421 ≤ Study Day ≤ 480 | 421 ≤ Study Day ≤ 495 | Month 16 |
| 421 ≤ Study Day ≤ 540 | 421 ≤ Study Day ≤ 555 | Month 18 |
| 541 ≤ Study Day ≤ 600 | 421 ≤ Study Day ≤ 615 | Month 20 |
| 601 ≤ Study Day ≤ 660 | 601 ≤ Study Day ≤ 675 | Month 22 |
| 661 ≤ Study Day ≤ 720 | 601 ≤ Study Day ≤ 735 | Month 24 |
| 721 ≤ Study Day ≤ 780 | 601 ≤ Study Day ≤ 795 | Month 26 |
| $(((m-1)*30)-29) \le \text{Study Day} \le$ | ((( <i>m</i> -1)*30)-29) ≤ Study Day ≤ | Month <i>m</i> , <i>m</i> =28, 30, |
| (((m-1)*30)+30) | ((( <i>m</i> -1)*30)+45) | |

NOTES:

<sup>+</sup> Only non-baseline records from the mentioned assessment window will be assigned to Day 1.

<sup>#</sup> Follow-up will be derived only for participants who permanently discontinued study treatment.

- For post-baseline visits (i.e. Month 2 and afterwards), apply Snapshot analysis windows only to viral load data that is on-treatment (per Table 15) within the Maintenance Phase (per Table 13).
- An on-treatment viral load assessment may be assigned to more than one snapshot analysis window, e.g. on-treatment assessment taken on Study Day 300 will be in both Month 10 and Month 12.
- a.± 45 Day window is always used at key analysis timepoint of Month 12.

Table 9 Assessment Windows for Summary of Snapshot Data for DTG + RPV arm— Data assigned to Maintenance Phase Only

| Snapshot Ana (If no on-treatment viral load data wind | Analysis Timepoint | |
|---|---|---|
| Default Expanded +67 Day Upper Window <sup>a</sup> | | |
| Last available recorded value up to<br>and including the date of first<br>Maintenance Phase dose of IP | Last available recorded value up to<br>and including the date of first<br>Maintenance Phase dose of IP | Baseline |
| 2 ≤ Study Day ≤ 135 | 2 ≤ Study Day ≤ 157 | Month 3 |
| 136 ≤ Study Day ≤ 225 | 136 ≤ Study Day ≤ 247 | Month 6 |
| 226 ≤ Study Day ≤ 315 | 226 ≤ Study Day ≤ 337 | Month 9 |
| 293 ≤ Study Day ≤ (Study Day of Nominal Month 12 Visit) | 293 ≤ Study Day ≤ (Study Day of Nominal Month 12 Visit) | Month 12 |

- For post-baseline visits (i.e. Month 3 and afterwards), apply Snapshot analysis windows only to viral load data that is on-treatment (per Table 15) within the Maintenance Phase (per Table 13).
- An on-treatment viral load assessment may be assigned to more than one snapshot analysis window, e.g. ontreatment assessment taken on Study Day 300 will be in both Month 9 and Month 12.
- a.- 67 Day window is always used at key analysis timepoint of Month 12.

Table 10 Assessment Windows for Summaries of Long-Term Follow Up
Phase Data for Subjects Who Received At least One Injection of
CAB+RPV and Permanently Discontinued from Study Treatment

| Analysis Window | Analysis<br>Timepoint | Target Study<br>Day of Window |
|---|---|---|
| 1 ≤ LTFU Study Day ≤ 67 | LTFU Month 1 | 30 |
| 68 ≤ LTFU Study Day ≤ 135 | LTFU Month 3 | 90 |
| 136 ≤ LTFU Study Day ≤ 225 | LTFU Month 6 | 180 |
| 226 ≤ LTFU Study Day ≤ 315 | LTFU Month 9 | 270 |
| 316 ≤ LTFU Study Day ≤ 405 | LTFU Month 12 | 360 |
| (30*m - 44) ≤ LTFU Study Day≤ (30*m + 45) | LTFU Month <i>m</i> ,<br><i>m</i> = 15, 18, | 7*m |

#### NOTES:

An assessment may be slotted to both LTFU and Maintenance Phase

## 12.3.3. Assessment Window for Study Conclusion

The study conclusion and phase conclusion records in disposition data will be slotted based on Table 6 and Table 7 However, if the discontinuation date is post-treatment (based on Table 15), the record will be slotted to the last on-treatment visit within the same phase rather than follow up.

#### 12.3.4. Assessment Window for Health Outcome Data

## 12.3.4.1. HIVTSQs, HIVTSQc, HIVDQoL, Preference

HIVTSQs, HIVTSQc, HIVDQoL, and Preference questionnaire assessments will be assigned to analysis visits as follows:

- 1. Baseline: Like other data, Baseline will be defined as last available recorded value up to and including the date of first Maintenance phase dose of study treatment. Baseline is not applicable for HIVTSQc and Preference assessments
- 2. Post-Baseline:
  - a. if the nominal visit identifier as captured in the source dataset corresponds to a scheduled collection per the Time and Events Schedule (see Section 12.2 and Table 11) and the assessment is collected in the Maintenance Phase (per Table 13), then the nominal visit identifier will be kept as the analysis visit.
  - b. if the nominal visit identifier is unscheduled or withdrawal, then the following procedure will be used:
    - i. Assign the assessment to a study phase according to Table 13. Proceed to step ii if the assessment is assigned to the Maintenance Phase.
    - ii. Identify the 'last nominal visit' with the HO assessment performed prior to the unscheduled/withdrawal visit to be slotted.
    - iii. The unscheduled/withdrawal visit will be slotted to the planned nominal visit subsequent to the 'last nominal visit'. If the 'last nominal visits' does not exist (e.g. no records originate from a planned nominal visit), then the unscheduled/withdrawal visit will be slot to the first planned nominal visit after Day 1.

Example 1, for HIVDQoL, the planned nominal visits are Day 1, Month 6 and Month 12. If a participant has the 'last nominal visit' (with HIVDQoL assessment) at Month 6 prior to withdrawal at Month 8, the withdrawal assessment will be slotted to the subsequent planned nominal visit of Month 12.

Example 2, for HIVDQoL, if there is unscheduled visit between Month 6 and Month 12. This unscheduled visit will be slotted to Month 12 per the rule. In this case, there are two assessments with analysis visit equal to Month 12 (i.e. the slotted value and the value at original nominal Month 12 visit). The original nominal value will be selected for summary per the rule below for multiple records—see Section 12.3.5.

Table 11 **Planned Nominal Visit of Health Outcome Data** 

| Endpoints | Day 1 | Month 6 | Month 12 |
|--------------|-------|---------|----------|
| HIVTSQc | | | Χ |
| HIVTSQs | Χ | Х | Χ |
| HIVDQoL | Χ | Х | Χ |
| Preference * | | | Х |

#### 12.3.4.2. **Reasons for Switch**

Reasons for Switch assessments are planned to be taken at nominal Day 1 visit only. The assessments taken within ± 2 weeks window from Maintenance phase treatment start date will be regarded as evaluable. The assessments taken outside this window will be excluded from the summary.

#### 12.3.5. Multiple assessments within an Analysis Window

If after window assignment there are multiple valid assessments of a parameter within the same window, then the following hierarchy will be used to determine the value to be used for summary statistics of observed values:

#### For data other than health outcome

- 1. The assessment closest to the window target Study Day;
- 2. If there are multiple assessments equidistant from the target Study Day, then the mean of these values will be used. For HIV-1 RNA, the geometric mean of the number of copies will be used as opposed to the arithmetic mean.

### For Health outcome data,

- 1. If there are multiple on-treatment assessments assigned to the same analysis visit, the assessment from the planned nominal visit will be used for summary statistics.
- 2. If there are multiple on-treatment assessments assigned to the same analysis visit and none originates from a planned nominal visit (e.g. two unscheduled/withdrawal nominal visits), then a. the assessment closest to the window target Study Day will be used:

  - b. if there are multiple assessments equidistant from the target Study Day, then the earliest assessment will be used.

Assessments not chosen for use in summary statistics by this algorithm will still appear in the associated listings. Also, all applicable valid assessments, irrespective of proximity to study day. will be used when categorizing values across visits, such as 'maximum grade' or 'at any time', and for any algorithm that has specific rules for which observation to use (e.g. snapshot algorithm or CVF identification).

<sup>\*</sup> not collected for DTG+RPV.

## 12.4. Appendix 4: Study Phases and Treatment State

## 12.4.1. Study Phases

Assessments and events will be classified according to the time of occurrence relative to the Treatment Start Date defined in Section 12.6.1.

AEs will be assigned to study phases as defined in Table 12. For example, adverse events on/after start of Maintenance phase IP and prior to start of LTFU ART will be assigned to the Maintenance Phase.

Laboratory data (efficacy, safety and virology), HIV associated Conditions, health outcomes assessments, vital signs, and ECGs will be assigned to study phases as defined as in Table 13. For example, assessments/events occurring after start of Maintenance Phase IP and up to and including start of LTFU ART will be assigned to the Maintenance Phase.

Assessments/events are assigned to study phases sequentially, starting from the top of each table. No study phases will be assigned to medications.

Table 12 Assignment of Study Phases for AEs

| Study Phase | Date range |
|---|---|
| Screening | Date < Maintenance Treatment Start Date |
| Maintenance | CAB LA + RPV LA:Maintenance Treatment Start Date ≤ Date < LTFU ART Start Date |
| | For AEs leading to withdrawal and started on the same date as LTFU ART Start Date, Maintenance Phase, instead of Long-term Follow-up phase, will be assigned. |
| | DTG + RPV: Maintenance Treatment Start Date ≤ Date < Date of nominal Month 12 visit |

#### NOTES:

- Date = AE Start date
- If participants have the missing LTFU ART start date, only the lower bound will be considered.
- Maintenance Treatment Start Date: refer to Treatment Start Date in Section 12.6.1

Table 13 Assignment of Study Phases for Lab Assessments (including Virology), ECG, Vital Sign, Health Outcomes, and HIV associated conditions

| Study Phase | Date range |
|---|---|
| Screening | Date ≤ Maintenance Treatment Start Date Note: 2-hour post-dose ECG taken on the Maintenance Treatment Start Date |
| | will be excluded. |
| Maintenance | CAB LA + RPV LA: |
| | Maintenance Treatment Start Date < Date ≤ LTFU ART Start Date |
| | DTG + RPV: |
| | Maintenance Treatment Start Date < Date ≤ Date of nominal Month 12 visit |
| | Note: 2-hour post-dose ECG taken on the Maintenance Treatment Start Date will be included. |

- Date = start or assessment date
- If participants have the missing LTFU ART start date, only the lower bound will be considered.
- Maintenance Treatment Start Date: refer to Treatment Start Date in Section 12.6.1

Table 14 Assignment to Long-Term Follow-Up Phase

| Study Phase | Date range |
|-------------|-------------------------------------------------------------|
| Long-Term | Date > max(Last IM Injection Date, Last Oral Dose End Date) |
| Follow-Up | |

#### NOTES:

- Date = start or assessment date
- For AEs leading to withdrawal and started on the same date as LTFU HAART Start Date, maintenance phase instead of long-term follow-up phase, will be assigned. Refer to Table 12 for details.

Only participants who received at least one CAB and/or RPV injection will enter the long-term follow-up.

Note that the long-term follow-up phase and maintenance phase are not necessarily mutually exclusive and are to be defined with separate phase variables in the datasets. For example, CAB LA + RPV LA subject who has Month 10 injection and withdrawal at Month 12 without receiving Month 12 injection, the "Month 12 withdrawal visit" belongs to both the maintenance phase and long-term follow-up phase.

#### 12.4.2. Treatment State

Within each treatment study phase (i.e. Maintenance and LTFU—based on assignment of study phase described in Section 12.4.1), only those assessments which occur within the ranges shown in Table 15 will be considered 'on-treatment' for the given phase. No treatment states will be assigned to medications.

Table 15 Treatment State within Study Phases

| Study Phase <sup>a</sup> | Treatment State | Date Range |
|---|---|---|
| Screening | Pre-treatment | All assessments/events within the phase |
| Maintenance | On-treatment | CAB LA + RPV LA: |
| | | Date ≤ max (Date of Last Oral Dose of |
| | | CAB+RPV + 1, Date of Last Injection + 67) |
| | | DTG + RPV: |
| | | Date ≤ Last Oral Dose Date + 1 |
| | Post-treatment | CAB LA + RPV LA: |
| | | Date > max (Date of Last Oral Dose of |
| | | CAB+RPV + 1, Date of Last Injection + 67) |
| | | DTG + RPV: |
| | | Date > Last Oral Dose Date + 1 |
| Long-Term | On-treatment | Date ≤ min(LTFU ART start date, max(Last |
| Follow-up | | Injection Date + 67, Last Oral dose Date + 1)) |
| | Post-treatment | Date > min(LTFU ART start date, max(Last |
| | | Injection Date + 67, Last Oral dose Date + 1)) |

- Treatment State is determined after data has been assigned to the study phases as defined in Section 12.4.1
- b. Last injection and/or last oral dose of CAB+RPV are only applied to subjects who permanently discontinue from study treatment. The assessments for participants who did not permanently discontinue the study treatment will be considered 'On-treatment'
- c. Date = Assessment/Start Date.

#### 12.4.2.1. Treatment States for AE Data

For adverse events, partial AE start date will use imputation as described in Section 12.7.2.1. In the case of a completely missing start date, the event will be considered to have started On-treatment at Maintenance phase unless an end date for the AE is provided which is before start of study treatment at Maintenance phase; in such a case the AE is assigned as Pre-treatment.

Within each treatment study phase, only those AE with onset date within the ranges shown in Table 15 will be considered 'on-treatment' for the given phase. The onset date will be derived based on Table 16.

# Table 16 Days since First Dose of Each Study Phase, Days since Phase Start, AE Duration and Relation to Study Treatment

| | Definition |
|---|---|
| Days since<br>First Dose<br>(Days) <sup>a</sup> | AE Start Date – Maintenance Treatment Start Date + 1 |
| Days since | AE Start Date – Date of Last Dose of Study Treatment prior to/on |
| Last Dose | the Start Date of AE + 1 |
| (Days) <sup>a</sup> | |
| Days since | For AEs in Maintenance Phase: |
| Phase Start | AE Start Date - Maintenance Treatment Start Date + 1 |
| | For AEs in Long-term Follow-up Phase: |
| | AE Start Date – Date of Last Dose of Study Treatment <sup>b</sup> |
| Duration | AE Resolution Date – AE Start Date + 1 |
| (Days) | |
| Drug-related | If relationship is marked 'YES' on Inform/CRF OR value is |
| | missing. |

#### NOTES:

- a. Days since First/Last Dose will only be derived for AEs assigned to maintenance phase and long-term follow-up phase.
- b. Date of Last Dose of Study Treatment = max (Last IM Injection Date, Last Oral Bridging End Date), only applicable to participants who permanently discontinued study treatment.

# 12.5. Appendix 5: Data Display Standards & Handling Conventions

## 12.5.1. Reporting Process

| Software | |
|---|---|
| The currently supported versions of SAS software will be used. | |
| Reporting Area | |
| HARP Server | : us1salx00259 |
| HARP Compound : \ARPROD\GSK1265744\mid209035 | |
| A 1 : D ( ) | |

#### **Analysis Datasets**

- Analysis datasets will be created according to CDISC standards (SDTM IG Version 3.2 & ADaM IG Version 1.1).
- For creation of ADaM datasets (ADCM/ADAE), the same version of dictionary datasets will be implemented for conversion from SI to SDTM.

#### **Generation of RTF Files**

RTF files will be generated for every reporting effort described in the RAP.

## 12.5.2. Reporting Standards

#### General

 The current GSK Integrated Data Standards Library (IDSL) will be applied for reporting, unless otherwise stated (IDSL Standards Location:

https://spope.gsk.com/sites/IDSLLibrary/SitePages/Home.aspx):

- 4.03 to 4.23: General Principles
- 5.01 to 5.08: Principles Related to Data Listings
- 6.01 to 6.11: Principles Related to Summary Tables
- 7.01 to 7.13: Principles Related to Graphics

#### **Formats**

- GSK IDSL Statistical Principles (5.03 & 6.06.3) for decimal places (DP's) will be adopted for reporting of data based on the raw data collected, unless otherwise stated.
- Numeric data will be reported at the precision collected on the eCRF.
- The reported precision from non eCRF sources will follow the IDSL statistical principles but may be adjusted to a clinically interpretable number of DP's.

### **Planned and Actual Time**

- Reporting for tables, figures and formal statistical analyses:
  - Planned time relative to dosing will be used in figures, summaries, statistical analyses and calculation of any derived parameters, unless otherwise stated.
  - The impact of any major deviation from the planned assessment times and/or scheduled visit days on the analyses and interpretation of the results will be assessed as appropriate.
- Reporting for Data Listings:
  - Planned and actual time relative to study drug dosing will be shown in listings (Refer to IDSL Statistical Principle 5.05.1).
  - Unscheduled or unplanned readings will be presented within the subject's listings.

### **Unscheduled Visits**

Unscheduled visits will be assigned to a study visit using the all-inclusive windows defined in Section 12.3.

However, data summaries will only report visits that are planned assessment time points for each parameter (according to the Time and Events table).

Assessments at unscheduled visits will be included for 'any time On-treatment' planned assessment time points and in data listings, as well any algorithms that make use of additional data (e.g., Snapshot).

| Descriptive Summary Statistics | |
|---|---|
| Continuous Data | Refer to IDSL Statistical Principle 6.06.1 |
| Categorical Data | N, n, frequency, % |
| Graphical Displays | |
| Refer to IDSL Statistical Principals 7.01 to 7.13. | |

## 12.6. Appendix 6: Derived and Transformed Data

#### 12.6.1. General

### **Multiple Measurements at One Time Point**

• If after window assignment there are multiple valid assessments of a parameter within the same window, refer to Section 12.3.5 for determination of the value to be used for summary statistics of observed values. Assessments not chosen for use in summary statistics will still appear in the associated listings. Also, all applicable valid assessments irrespective of proximity to the target study day, will be used when categorizing values across visits, such as 'maximum grade' or 'at any time', and for any algorithm that has specific rules for which observation to use (e.g. snapshot algorithm or CVF identification).

#### **Treatment Start Date**

Treatment start date is defined for the Maintenance Phase as follows:

- For subjects who were on CAB LA + RPV LA, this is the date of the first injection dose entered onto the IP exposure eCRF form.
- For subjects who were on oral DTG + RPV, this is the date of the first oral dose entered onto the IP exposure eCRF form.

For the long-term follow-up phase (only for CAB LA + RPV LA arm):

- If a participant is still on study treatment, or permanently discontinued the study treatment and did not have any previous injections, treatment start date is missing.
- If a participant permanently discontinued the study treatment and had at least one injection, treatment start date is the date of first HAART treatment after the last dose of study treatment (oral or injection).

#### Study Day

The Study Day of an event (e.g., lab assessment, vital sign, ECG, start date of AE or HIV associated condition) will be derived as the number of days between the date of the event and the start date of study treatment on Maintenance phase as follows:

if date of event ≥ start date of study treatment, then

Study Day = Date of Event – Start Date of Maintenance Phase IP + 1

if date of event < start date of study treatment, then

Study Day = Date of Event – Start Date of Maintenance Phase IP

Note that the start date of study treatment on Maintenance phase is considered to be on Study Day 1 and the day before this is Study Day -1; i.e., there is no Study Day 0.

## Long-Term Follow Up Study Day

The Long-Term Follow Up (LTFU) Study Day of an event (e.g., lab assessment, start date of AE or HIV associated condition) will be derived as the number of days between the date of the event and the end of IP treatment [i.e max (Last IM Injection Date, Last Oral Bridging End Date)]as follows:

If the onset of event falls in Long-term Follow up phase, then

LTFU Study Day = date of event – end date of IP

## **Change from Baseline**

Post-Dose Visit Value – Baseline

• Unless otherwise specified, the baseline definitions specified in Section 5.2 will be used for derivations for endpoints / parameters.

## 12.6.2. Study Population

## **Demographics and Baseline Characteristics**

#### Age

- Age, in whole years, will be calculated with respect to the subject's Baseline visit.
- GSK standard IDSL algorithms will be used for calculating age where birth date will be imputed as follows:
  - Any subject with a missing date and month will have this imputed as '30th June'.
- Birth date will be presented in listings as 'YYYY'.
- Completely missing dates of birth will remain as missing, with no imputation applied.
   Consequently, the age of the subject will not be calculated and will remain missing.

#### **Body Mass Index (BMI)**

• Calculated as Weight (kg) / Height (m)<sup>2</sup>

#### **Hepatitis Status**

- Hepatitis C status will be determined using antibody and/or hepatitis C virus (HCV) RNA assessments performed during screening or during the conduct of the study.
- If both antibody and virus RNA assessments are available, then the latter will take precedence and positive/negative status will be based on whether HCV RNA is detectable (i.e., ≥ limit of quantification) or not.
- A participant will be considered positive for hepatitis B virus (HBV) if they have a positive surface antigen or detectable HBV DNA result. "HBV DNA DETECTED" in the lab comment takes precedence over HBV DNA test result for positive hepatitis B status, for example, if a participant has HBV test result below level of detection, however, the lab comment shows that HBV DNA detected, this participant will be considered positive for hepatitis B. If HBV DNA result is available, it will be used to qualify hepatitis B status as positive or negative (positive if ≥ limit of quantification); otherwise Hepatitis B status will be determined using the surface antigen result.
- Hepatitis status at entry will be based on the assessments prior to/on the start of the study treatment.

#### **Demographics and Baseline Characteristics**

## **Lipid-modifying Agents**

- The following ATC codes correspond to lipid-modifying agents:
  - ATC Level 2: C10
  - ATC Level 3: C10A, C10B (if Level 2 is not available)
  - ATC Level 4: C10AA, C10AB, C10AC, C10AD, C10AX, C10BA, C10BX (if level 2, 3 are not available)
- Participants are considered to have used a lipid-modifying agent at baseline if they are taking the medication at the time of their baseline fasting lipid testing date.
- Participants are also considered to have used a lipid-modifying agent at baseline if they stopped their lipid modifying medication within 12 weeks prior to their baseline fasting lipid testing date.

## **Extent of Exposure**

Exposure to CAB LA +RPV LA injection and to DTG + RPV oral will be calculated from the IP eCRF pages.

#### CAB LA + RPV LA:

- Exposure = Number of IP injections received during Maintenance Phase.
- Overall exposure to IP = min(Date of Latest Maintenance Phase visit, max(Date of Last Injection + 67, Date of Last Dose of Oral CAB+RPV)) – Date of First Study Injection + 1 Note: Last Injection and/or Last Dose of Oral CAB+RPV are only applicable to those who permanently discontinued study treatment.

#### DTG + RPV:

- Exposure = IP Stop Date IP Start Date + 1
- Overall exposure to IP = min(Date of Latest Maintenance Phase visit, Date of Last Dose of DTG + RPV) – Date of First Dose + 1
- There will be no adjustments to the exposure duration for any missed doses.

Duration of dosing in subject years will be calculated as the sum of subject duration of dosing in days (across all subjects)/365.25.

Subjects who were enrolled but did not report an IP start date will be categorised as having zero days of exposure.

For DTG + RPV arm, missing IP discontinuation date will be imputed, for purposes of calculating exposure, as the date of last visit or the recorded date of withdrawal/completion, whichever is earlier.

## Adherence to CAB LA + RPV LA Injection Schedule

Timeliness of Injections relative to Date of Projected Dosing Visits is assessed by using "actual injection visit date - projected visit date from first injection". The injections of interest in adherence analysis are those after first injection. Each injection visit is counted only once. Individual CAB and RPV injections administered at the same visit are not counted twice. "Extra" unscheduled injections are excluded from all derivations. For example, if during a scheduled visit a participant receives 1 ml

of injection instead of 3 ml due to a dosing error, but this participant returns one week later for the remaining 2 ml injection, then the additional visit is excluded. If a participant receives an extra injection at an unscheduled visit by mistake, this visit will also be excluded.

The planned interval is 60 days for the CAB LA + RPV LA arm. Relative days between two planned consecutive visits for injections relative to the planned interval will be calculated as below:

Relative Days=Actual number of days between adjacent injections – 60.

For example, if the time interval between two scheduled consecutive visits for injections is 55 days then relative days = 55 - 60 = -5; if the interval is 60 days then relative days = 65 - 60 = 5 The relative days will be grouped as below:

```
<-14 days
-14 to -8 days
-7 to -4 days
-3 to -2 days
-1 day
0 days
1 day
2 to 3 days
4 to 7 days
8 to 14 days
>14 days
Missed Injection without Oral Bridging
```

Missed Injection with Oral Bridging

In the case that a scheduled injection visit is missed, the time interval between the preceding and the subsequent scheduled injection will be calculated. For example, if Month 8 injection is missed, then the number of days between the actual Month 6 and Month 10 injections will be calculated. To calculate the proportion of injection intervals for each of the above category of relative days, the denominator is the total count of time intervals between adjacent injection visits for CAB LA + RPV LA arm.

## 12.6.3. **Efficacy**

#### **Snapshot**

- The Snapshot algorithm is intended to be primarily a virologic assessment of the endpoint, and as such follows a "virology first" hierarchy.
- 'HIV-1 RNA <50 c/mL' or 'HIV-1 RNA ≥50 c/mL' within an analysis window (see Table 8 and Table 9) is typically determined by the last available HIV-1 RNA measurement in that window while the subject is On-treatment in the Maintenance Phase (as assigned based on Section 12.4.1).</li>
- When no HIV-1 RNA data is available within a window, a subject cannot be assigned to the

category of 'HIV-1 RNA < 50 c/mL'. Depending on the reason for lack of data, the subject will be classified as a 'HIV-1 RNA≥50' or reported as 'No Virologic Data at Month X'; in the latter case, the algorithm further classifies the nature of the missing data. Typically, a subject withdrawn (i) due to AE or, (ii) for another reason yet was suppressed at the time, will be counted as 'No Virologic Data at Month X'. Should a subject withdraw for reasons other than AE and was not suppressed at the time, they will be categorized as 'HIV-1 RNA≥50'.

- Full details of the algorithm, including the handling of special cases, are included in Section 12.9
- For each scheduled assessment time, the Snapshot response rate for a given threshold (e.g., <50 c/mL) is defined as:

Snapshot Response Rate= Number of responders in that analysis window Number of subjects in the analysis population

• For each scheduled assessment time, the Snapshot 'HIV-1 RNA≥50'rate for a given threshold (e.g., ≥50 c/mL) is defined as:

SnapshotVF Rate= Number of VFs in that analysis window Number of subjects in the analysis population

#### Plasma HIV-1 RNA

- For summaries and analyses which use HIV-1 RNA level as a continuous measure, the logarithm to base 10 of the value will be used.
- HIV-1 RNA results may be provided as censored values, such as <40 or >9,999,999 c/mL. For
  the purposes of summary statistics, such values will be replaced by the next value beyond the
  limit of detection, e.g., 39 or 10,000,000 c/mL, respectively, for the given examples. Data
  listings will show the censored values as provided.

## Target Detected / Target Non Detected/Super low viral load testing

- When a measurement of plasma HIV-1 RNA is below the limit of quantification (i.e. 40 c/mL) and is qualitatively observable that will be denoted as a "Target Detected" measure, while HIV-1 RNA below the limit of quantification that is not qualitatively observable that will be denoted as "Target Not Detected". Any measurements <40 c/mL characterised as "Target Non Detected" or "Target Detected" will be captured in the database.</li>
- Super low viral load will also be tested by BioMNTR lab for Viral loads below the limit of quantification at some visits (e.g. Month 12)

### **Confirmed Virologic Failure (CVF)**

- The definition of CVF is provided in the Protocol, Section 7.1.4 Definition of Protocol-Defined Confirmed Virologic Failure
- In case there are multiple plasma HIV-1 RNA results on the same day, the worst result (i.e. the largest value) will be used in determination of CVF.

### Summary for Participants per Viral Load Category by Visit

- Summary will be based on observed available data, with no imputation for missing values. The
  proportion of participants in each viral load category will be calculated using the denominator
  and numerator specified below:
  - Denominator: Number of participants with on-treatment viral load within the snapshot visit window.
  - Numerator: Number of participants with plasma HIV-1 RNA in the specified category based on the last on-treatment viral load assessment collected within the snapshot visit window.

## **HIV-1 Disease progression Stage**

- Categories:
  - CDC Stage I at Maintenance Baseline to CDC Stage III;
  - CDC Stage II at Maintenance Baseline to CDC Stage III;
  - CDC Stage III at Maintenance Baseline to new CDC Stage III event and
  - CDC Stage I, II, III at Maintenance Baseline to death.

Please refer to Protocol (Appendix 8: CDC Classification for HIV-1 Infection (2014)) for defining Stage.

- For the purpose of analysis, the CDC at Baseline and at post-baseline during Maintenance phase will be derived as below:
  - At Baseline, the 'Baseline CDC stage' for each subject was assessed by the investigator and recorded in the eCRF. However, for the analysis, Maintenance Baseline CDC stage will be re-derived based on Maintenance Baseline CD4+ values as well as whether any HIV-associated conditions present at Baseline per the Criteria's thresholds (Appendix 8 in Protocol).
  - To analyse disease progression, the most advanced post-baseline CDC stage within the period of interest (e.g. Maintenance Phase) will be derived based on the occurrences of new AIDS-defining conditions (please refer to Appendix 8 in Protocol for the list of AIDs-defining Conditions) as well as the nadir value of Maintenance CD4+. For example,
    - If a subject with CDC 'Stage I' at Maintenance Baseline had the lowest Maintenance Phase CD4+ =120 cell/mm³ without new AIDs-defining conditions, then HIV disease progression for this subject during the Maintenance phase would be considered as 'CDC stage I at Baseline to CDC stage III'.
    - If a subject with CDC 'Stage II' at Baseline had the lowest Maintenance Phase CD4+ =220 cell/mm³ AND had at least one new AIDs-defining condition, then HIV disease progression for this subject during the Maintenance Phase would be considered as 'CDC stage II at Baseline to CDC stage III'.

## 12.6.4. Safety

#### **Adverse Events**

#### **DAIDS Grading**

 Clinical adverse events will be graded based on the Division of AIDS Table for Grading the Severity of Adult and Pediatric Adverse Events Version 2.1, March 2017, as specified in the protocol Appendix 2.

## Potential QTc Interval Prolonging Events of Interest

Potential QTc Interval Prolonging Events of Interest cases will be identified based on Standardised MedDRA Query (SMQ) for Torsade de pointes/QT prolongation, broad (MedDRA). The terms per this reference are listed below.

#### AE preferred term

| Adverse Events |
|----------------------------------------------|
| Electrocardiogram QT interval abnormal |
| Electrocardiogram QT prolonged |
| Long QT syndrome |
| Long QT syndrome congenital |
| Torsade de pointes |
| Ventricular tachycardia |
| Cardiac arrest |
| Cardiac death |
| Cardiac fibrillation |
| Cardio-respiratory arrest |
| Electrocardiogram repolarisation abnormality |
| Electrocardiogram U wave inversion |
| Electrocardiogram U wave present |
| Electrocardiogram U-wave abnormality |
| Loss of consciousness |
| Sudden cardiac death |
| Sudden death |
| Syncope |
| Ventricular arrhythmia |
| Ventricular fibrillation |
| Ventricular flutter |
| Ventricular tachyarrhythmia |

### **Laboratory Parameters**

- If a laboratory value which is expected to have a numeric value for summary purposes, has a non-detectable level reported in the database, where the numeric value is missing, but typically a character value starting with '<x' or '>x' (or indicated as less than x or greater than x in the comment field) is present, the number of significant digits in the observed values will be used to determine how much to add or subtract in order to impute the corresponding numeric value. If a character value starting with "<=x", then the numeric value will be x.
  - $\circ$  Example 1: 2 Significant Digits = '< x ' becomes x 0.01
  - Example 2: 1 Significant Digit = '> x' or '>=x' becomes x + 0.1
  - Example 3: 0 Significant Digits = '< x' becomes x 1

## Estimate of Glomerular Filtration Rate (GFR) (Levey, 2012)

• Chronic Kidney Disease Epidemiology Collaboration (CKD-EPI) equation [Levey, 2012].will be used by the central laboratory to provide an estimate of GFR, in mL/min per 1.73 m², as follows:

#### **Laboratory Parameters**

GFR = 
$$141 \times \min \left(\frac{\text{CRT}_{\text{mg/dL}}}{\kappa}, 1\right)^{\alpha} \times \max \left(\frac{\text{CRT}_{\text{mg/dL}}}{\kappa}, 1\right)^{-1.209} \times 0.993^{\text{Age}} \times [1.018 \text{ if Female}] \times [1.159 \text{ if Black}]$$

where age (in years) is at time of assessment,  $\kappa$  = 0.7 if female or 0.9 if male,  $\alpha$  = -0.329 if female and -0.411 if male, min() indicates the minimum of CRT/ $\kappa$  or 1, max() indicates the maximum of CRT/ $\kappa$  or 1, and CRTmg/dL is serum creatinine concentration in mg/dL. The serum creatinine concentration in mg/dL is obtained from GSK standard units of  $\mu$ mol/L as CRTmg/dL =0.0113x CRT $\mu$ mol/L.

• The CKD-EPI GFR will also be calculated using Cystatin C, as follows

133 X min(Scys/0.8, 1) -0.499 X max (Scys/0.8, 1)-1.328 X 0.996 Age X[0.932 if female]

Where Scys is serum cystatin C mg/Liter, min indicates the minimum of Scr/0.8 or 1, and max indicates the maximum of Scys/0.8 or 1

# Lab Toxicities – DAIDS Grading based on Version 2.1, March 2017, as specified in the protocol of Appendix 2

- Toxicities will be based on the Division of AIDS (DAIDS) grading system, Version 2.1, March 2017, as specified in the protocol of Appendix 2.
- Toxicity grades provided by the central laboratory do not distinguish between abnormally high or low criteria, when both are relevant for a particular parameter.
- When summarising toxicity grades for such parameters, they will be categorised as to whether they are above or below the midpoint of normal range.

| Parameter | Below Midpoint for those ≥Grade 1 | Above Midpoint for those ≥Grade 1 |
|---|---|---|
| Fasted glucose | Hypoglycemia | Hyperglycemia |
| Sodium | Hyponatremia | Hypernatremia |
| Potassium | Hypokalemia | Hyperkalemia |

## National Cholesterol Education Program (NCEP) Lipid Categories

 In addition to DAIDS toxicity grades (see protocol), lipid values will be categorized according to the 2001 NCEP Adult Lipid Guidelines [Grundy, 2001]

| Parameter | Value Range (mmol/L) | Value Range (mg/dL) | Category |
|---|---|---|---|
| Triglycerides | <1.70 | <150 | Normal |
| | 1.70 to <2.26 | 150 to <200 | Borderline High |
| | 2.26 to <5.65 | 200 to <500 | High |
| | ≥5.65 | ≥500 | Very High |
| Total Cholesterol | <5.18 | <200 | Desirable |
| | 5.18 to <6.21 | 200 to <240 | Borderline High |
| | ≥6.21 | ≥240 | High |
| HDL Cholesterol | <1.04 | <40 | Low |

| Laboratory Parameters | | | |
|-----------------------|---------------|-------------|--------------------|
| | 1.04 to <1.56 | 40 to <60 | Normal |
| | ≥1.56 | ≥60 | High |
| LDL Cholesterol | <2.59 | <100 | Optimal |
| | 2.59 to <3.37 | 100 to <130 | Near/Above Optimal |
| | 3.37 to <4.14 | 130 to <160 | Borderline High |
| | 4.14 to <4.92 | 160 to <190 | High |
| | ≥4.92 | ≥190 | Very High |

## **Other Safety Endpoints**

### **Corrected QTC**

When not entered directly in the eCRF, corrected QT intervals by Bazett's (QTcB) and Fridericia's (QTcF) formulas will be calculated, in msec, depending on the availability of other measurements.

If RR interval (in msec) is provided then missing QTcB and/or QTcF will be derived as

$$QTcB = \frac{QT}{\sqrt{RR/1000}} \qquad \qquad QTcF = \frac{QT}{\sqrt[3]{RR/1000}}$$

where uncorrected QT interval is also measured in msec.

If RR interval is not provided directly and one of QTcB or QTcF has been entered, then RR interval can be obtained from the above formulas and used to calculate the other correction method value; i.e.,

$$QTcB = \sqrt{\frac{QTcF^3}{QT}}$$

$$QTcF = \sqrt[3]{QT \cdot QTcB^2}$$

### 12.6.5. Health Outcomes

### **HIVTSQs**

## Questionnaire (Questions 1-12 are scored 0-6)

CCI - This section contained Clinical Outcome Assessment data collection questionnaires or indices, which are protected by third party copyright laws and therefore have been excluded.

#### **Treatment Satisfaction Score**

- Item 12 will not be included in Total Treatment Satisfaction Score. Instead, it will be treated as a stand-alone item only.
- Higher scores represent greater treatment satisfaction as compared to the past few weeks.
- A maximum of 5 items can be missing, which can be imputed to reflect the mean of the completed item scores. If 6 or more items are missing, then the treatment satisfaction scale score should not be computed and would remain missing.

### **Individual Item Scores**

- Items are rated as (CCI), etc.).
- Higher scores represent greater satisfaction with each aspect of treatment
- For individual item scores outputs, missing scores will not be computed (according to Page 7 of the [HIVDQoL User Guidelines, 2018]) and would remain missing.

#### **HIVTSQc**

## Questionnaire (Questions 1-12 are scored -3 to 3)

CCI - This section contained Clinical Outcome Assessment data collection questionnaires or indices, which are protected by third party copyright laws and therefore have been excluded.

## **Treatment Satisfaction Score (change)**

- Total Treatment Satisfaction Score is computed with items
   CCI
- Item 12 will be computed as an individual item only.
- The higher the score, the greater the improvement in satisfaction with treatment; the lower the score, the greater the deterioration in satisfaction with treatment. A score of 0 represents no change.
- A maximum of 5 items can be missing, the missing scores will be imputed with the mean of the
  completed item scores. If 6 or more items are missing, then the overall treatment satisfaction
  scale score should not be computed and will remain missing.

## **Individual Treatment Change Item Scores**

- Items are rated as ccl etc.) to ccl , etc.).
- The higher the score, the greater the improvement in satisfaction with each aspect of treatment and the lower the score, the greater the deterioration in satisfaction with each aspect of treatment.

#### **HIVDQoL**

## Questionnaire (Questions I and II are overview items and 1-26 are domain-specific items)

This questionnaire has been provided in three different languages: English (US and Canadian), French (Canadian), Spanish (US). Below is an example of the questionnaire.

third party copyright laws and therefore have been excluded.

| CCI - This section contained Clinical Outcome Assessment data collection questionnaires or indices, which are protected by third party copyright laws and therefore have been excluded. |
|---|
| third party copyright laws and therefore have been excluded. |

| CCI - This section contained Clinical Outcome Assessment data collection questionnaires or indices, which are protected by third party copyright laws and therefore have been excluded. |
|---|
| umu party copyright laws and merelore have been excluded. |

| CCI - This section contained Clinical Outcome Assessment data collection questionnaires or indices, which are protected by third party copyright laws and therefore have been excluded. |
|---|
| unite party copyright laws and therefore have been excluded. |

| CCI - This section contained Clinical Outcome Assessment dathird party copyright laws and therefore have been excluded. | ata collection questionnaires or indices, which are protected by |
|---|---|
| unitu party copyright laws and therefore have been excluded. | |

| CCI - This section contained Clinical Outcome Assessment da | ata collection questionnaires or indices, which are protected by |
|---|---|
| third party copyright laws and therefore have been excluded. | |

| CCI - This section contained Clinical Outcome Assessment data third party copyright laws and therefore have been excluded. | collection questionnaires or indices, which are protected by |
|---|---|
| unitu party copyright laws and therefore have been excluded. | |

| CCI - This section contained Clinical Outcome Assessment data collection questionnaires or indices, which party copyright laws and therefore have been excluded. | n are protected by third |
|---|---|
| party copyright laws and therefore have been excluded. | |

| CCI - This section contained Clinical Outcome Assessment dathird party copyright laws and therefore have been excluded. | nta collection questionr | naires or indices, whic | ch are protected by |
|---|---|---|---|
| third party copyright laws and therefore have been excluded. | | | |

| CCI - This section contained Clinical Outcome Assessment data collection questionnaires or indices, which are protected by third party copyright laws and therefore have been excluded. |
|---|
| and party obpyright have and allerelere have been excluded. |
| Individual Domain Items [HIVDQoL User Guidelines, 2018] |
| There are two overview items which are rated as: |
| O : CG |
| CCI - This section contained Clinical Outcome Assessment data collection questionnaires or indices, which are protected by third party copyright laws and therefore have been excluded. |
| are protected by third party copyright laws and therefore have been excluded. |
| The 26 domain-specific items include two rating scales, one measuring impact, part a, and the |
| other measuring the importance of the domain for QoL, part b. |
| The impact scores are rated as CCI The impact scores are rat |
| and the importance scores are rated as CCI to CCI |
| Weighted Impact Scores [HIVDQoL User Guidelines, 2018] |
| The impact ratings are multiplied by the corresponding importance rating to provide a |
| weighted-impact score for each applicable domain from CCI to CCI |

CCI

- If one part of a domain response (i.e. either part a or part b) is missing, a weighted impact score cannot be imputed for that question.
- If more than one option has been selected for a question, then if the options are consecutive (e.g. 2 and 3), then take the mid-point (i.e. 2.5) to be the final score for that question. However, if the two answers are not immediately next to each other (e.g., 0 and 3), treat the score as missing.

## Average Weighted Impact (AWI) Score [HIVDQoL User Guidelines, 2018]

- Weighted impact scores are summed and divided by the number of applicable domains (excluding domains with missing data), to give an overall AWI score. The non-applicable domains are hence ignored.
- If there are more than three items with missing scores out of the 14 core domain-specific items which do not have the N/A option, then the AWI score will not be computed.
- Item 23 and item 25 are not included when calculating AWI scores along with the two overview items I and II.

#### **Reason for Switch**

#### Questionnaire

You have chosen to continue participating in a clinical study where your daily oral HIV medication will be switched to a Long-Acting injectable HIV medication.

CCI

[select all that apply]:

CCI - This section contained Clinical Outcome Assessment data collection questionnaires or indices, which are protected by third party copyright laws and therefore have been excluded.

### **Data handling**

- If the questionnaire is taken beyond ± 2 weeks window from maintenance phase treatment start date (i.e. Study Day < -14 or Study Day > 14) it will be considered not evaluable and will not be included in the summary.
- Any missing values will remain missing (i.e. no imputation).

#### Preference question

#### Questionnaire

CCI - This section contained Clinical Outcome Assessment data collection questionnaires or indices, which are protected by third party copyright laws and therefore have been excluded.



## **12.6.6.** Virology

## Genotype

## **Amino Acid Changes**

- A mutation is considered present whenever the encoded amino acid residue differs from the amino acid that would have been encoded by the wild-type (e.g., HXB2, NL43) comparator gene; e.g., Q148K.
- If the encoded amino acid is seen as a mixture of wild-type and mutant amino acid, e.g., Q148Q/K, the mutated amino acid is considered present at the codon of interest.
- If the encoded amino acid is seen as a mixture of two or more amino acids, which may or may
  not include wild type, e.g., Q184K/H or Q184K/H/Q, etc., for the purposes of calculating the
  number of mutated amino acids, only one mutation is considered to be present at the codon of
  interest.

## **Representation of Amino Acid Changes**

| Mutations | Amino acid change |
|---|---|
| T69S | Single mutation from amino acid 'T' (vendor reference) to 'S' (sample) at codon '69' |
| Q148H/K/R | Mixture of amino acid mutations 'H', 'K' and 'R' (sample) from amino acid 'Q' |
| | (vendor reference) at codon '148' |
| _69_1T | First insertion of amino acid 'T' (sample) at codon '69' |
| _69_2S | Second insertion of amino acid 'S' (sample) at codon '69' |
| _69_3S/A | Third insertion of a mixture of amino acids 'S' and 'A' (sample) at codon '69' |
| L74L/- | Mixture of amino acid 'L' (sample) and a deletion at codon '74' |
| V75- | Single deletion of amino acid (sample) at codon '75' |

#### **Resistance Associated Mutations**

Known INI mutations associated with the development of resistance to BIC, RAL, EVG or DTG:

| Amino Acids in | H51Y, <b>T66A/I/K</b> , <b>E92Q/V</b> /G, Q95K, T97A, G118R, <b>F121Y</b> , E138A/K/T, |
|---|---|
| HIV Integrase for | G140A/C/R/S**, Y143C/H/R/K/S/G/A, P145S, Q146P, S147G, |
| Analysis | Q148H/K/R/N, V151A/I/L, S153F/Y, N155H/S/T, E157Q, G163R/K, |
| | S230R, D232N, R263K, L68V/I*, L74I/M*, E138D*, V151I*, G193E* |

#### NOTES:

Draft listing; may be modified in case of additional substantive data availability.

INI mutations listed taken from Stanford HIV Resistance Database (http://hivdb.stanford.edu/DR/cgi-bin/rules\_scores\_hivdb.cgi?class=INI cited 25Oct2019) and accessed on 28Jan2020.

INI substitutions listed above in bold had a score of =60.

 Major resistance mutations to other classes (i.e., NRTI, NNRTI, PI) as defined by the International Antiviral Society-USA (IAS-USA). The most up to date IAS-USA guidelines available at the time of DBF will be used in the analysis [Wensing, 2019].

| Class | Mutations |
|---|---|
| NRTIs | M41L, A62V, K65R/E/N, D67N, 69 insert, K70E/R, L74V, V75I, F77L, Y115F, F116Y, Q151M, M184V/I, L210W, T215Y/F, K219Q/E |
| NNRTIs | L100I, K101E/P, K103N/S, V106A/M, V108I, E138/A/G/K/Q/R, V179L,Y181C/I/V, Y188C/L/H, G190S/A, H221Y, P225H, F227C, M230I/L, |
| Pls | D30N, V32I , M46I/L, I47A/V, G48V, I50V/L, I54M/L/V, Q58E, T74P, L76V, V82A/T/F/L/S, N83D, I84V, N88S, L90M |

Note: List generated from IAS\_USA Guideline, [Wensing, 2019]

#### **Phenotype**

#### Phenotypic Susceptibility

Phenotypic susceptibility to all licensed antiretroviral drugs and CAB will be determined using PhenoSense HIV assays from Monogram Inc. and will be reported as fold change (FC) in IC50 relative to wild-type control virus NL4-3, i.e., FC of sample virus = IC50 of sample virus/IC50 of control virus.

Phenotypic susceptibilities will be categorised according to FC as shown in the tables below (based on Monogram PhenoSense assay). Clinical cutoffs (where available) or biological cutoffs by PhenoSense will be used to define the phenotypic susceptibility of background treatment by Monogram.

Replication capacity is generated as part of standard phenotypic assays

<sup>\*</sup> Denotes additional INI mutations added as they were identified during in vitro passage of DTG or seen in a previous DTG study in INI-experienced subjects (ING112574).

<sup>\*\*</sup>G140R is potentially associated with CAB based on in-stream data monitoring of CVF participants

| PhenoSense Algorithm | | | |
|----------------------|--------------|-------|-----------------------|
| Drug | Abbreviation | Class | PhenoSense cutoff |
| Abacavir | ABC | NRTI | $(4.5 - 6.5)^a$ |
| Lamivudine | 3TC | NRTI | 3.5 a |
| Didanosine | ddl | NRTI | (1.3 – 2.2) a |
| Stavudine | d4T | NRTI | 1.7 a |
| Zidovudine | AZT (ZDV) | NRTI | 1.9 |
| Emtricitabine | FTC | NRTI | 3.5 |
| Tenofovir | TDF (TAF) | NRTI | (1.4 – 4) a |
| Delavirdine | DLV | NNRTI | 6.2 |
| Efavirenz | EFV | NNRTI | 3 |
| Nevirapine | NVP | NNRTI | 4.5 |
| Etravirine | ETR | NNRTI | (2.9-10) a |
| Rilpivirine | RPV | NNRTI | 2.0 |
| Fosamprenavir/r | FPV/r | PI | (4-11) a |
| Atazanavir | ATV | PI | 2.2a |
| Atazanavir/r | ATV/r | PI | 5.2 a |
| Indinavir/r | IDV/r | PI | 10 a |
| Lopinavir/r | LPV/r | PI | (9 – 55) <sup>a</sup> |
| Nelfinavir | NFV | PI | 3.6 |
| Saquinavir/r | SQV/r | PI | (2.3 – 12) a |
| Tipranavir/r | TPV/r | PI | (2 – 8) a |
| Darunavir/r | DRV/r | PI | (10 – 90) a |
| Ritonavir | RTV | PI | 2.5 |
| Enfuvirtide | T20 | FI | 6.48 |
| Cabotegravir | CAB | INI | 2.5 |
| Raltegravir | RAL | INI | 1.5 |
| Elvitegravir | EVG | INI | 2.5 |
| Dolutegravir | DTG | INI | (4-13) a |
| Bictegravir | BIC | INI | (2.5 - 10) |

clinical cutoff (lower cutoff - higher cutoff).

Phenotypic susceptibility to each drug in a subject's background regimen is determined by applying drug-associated cutoffs as defined by the PhenoSense algorithm to the phenotypic fold resistance as below:

## **Full Sensitivity**

| Fold Change | Interpretation |
|--------------------------------------------|----------------|
| > clinical lower cutoff or biologic cutoff | resistance |
| ≤ clinical lower cutoff or biologic cutoff | sensitive |

## **Partial Sensitivity**

| Fold Change | Interpretation |
|------------------------------------------------------|---------------------|
| > clinical higher cutoff | resistance |
| ≤ clinical higher cutoff and > clinical lower cutoff | partially sensitive |
| ≤ clinical lower cutoff | sensitive |

PHENOTYP dataset from Monogram contains the phenotypic susceptibility for each drug derived from the cutoff listed above. Thus, phenotypic susceptibility (i.e. full sensitivity and partial sensitivity) will not be re-derived for our analysis.
## **Genotypic and Net Assessment Susceptibility**

Genotypic and Net assessment susceptibility to all licensed antiretroviral drugs and CAB will be determined from Monogram Inc. Net assessment susceptibility will be reported with the categories of 'resistance', 'partially sensitive', and 'sensitive' as what will be performed for phenotypic susceptibility. Genotypic and Net assessment susceptibility will be assessed at time of CVF using plasma sample, Genotypic susceptibility may be assessed at baseline using PBMC.

# 12.7. Appendix 7: Reporting Standards for Missing Data

# 12.7.1. Premature Withdrawals

| Element | Reporting Detail |
|---|---|
| General | Subject study completion (i.e. as specified in the protocol) was defined as: Participants are considered to have completed the study if they remain on therapy (i.e., have not permanently discontinued study intervention) and satisfy one of the following: |
| | Assigned to either treatment group, completed the Maintenance Phase (Month 12 for DTG +RPV participants only), remaining on study until commercial supplies of CAB LA + RPV LA Q2M or DTG + RPV regimens become locally available or development of CAB LA + RPV LA is terminated; |
| | Additionally, participants will continue this study until: |
| | the participant no longer derives clinical benefit, |
| | the participant meets a protocol-defined reason for discontinuation |
| | Participants who withdraw from CAB LA + RPV LA and go into the LTFU Phase will be considered to have prematurely withdrawn from the study intervention. |
| | • In addition to the 52-week Follow-Up phase required for participants who receive one or more injections with CAB LA or RPV LA, an in-clinic Follow-Up visit will be conducted approximately 4 weeks after the last dose of study medication for participants who withdraw from the DTG + RPV regimen with ongoing AEs, and serious adverse events (SAEs) and also any laboratory abnormalities that are considered to be AEs or potentially harmful to the participant, at the last on-study visit. Assessments at the Follow-up visit should reflect any ongoing complaints (e.g., blood draws to follow a laboratory abnormality). Follow-Up visits are not required for successful completion of the study. |
| | Withdrawn participants will not be replaced |
| | All available data from participants who were withdrawn from the study will be listed and all available planned data will be included in summary tables and figures, unless otherwise specified. |
| | Withdrawal visits will be slotted as per Appendix 3: Assessment Windows or will be summarised as withdrawal visits. |

# 12.7.2. Handling of Missing Data

| Element | Reporting Detail |
|---|---|
| General | <ul> <li>Missing data occurs when any requested data is not provided, leading to blank fields on the collection instrument:</li> <li>These data will be indicated by the use of a "blank" in subject listing displays. Unless all data for a specific visit are missing in which case the data is excluded from the table.</li> </ul> |

| Element | Reporting Detail |
|---|---|
| | <ul> <li>Answers such as "Not applicable" and "Not evaluable" are not considered to<br/>be missing data and should be displayed as such.</li> </ul> |
| Outliers | Any participants excluded from the summaries and/or statistical analyses will be documented along with the reason for exclusion in the clinical study report. |

# 12.7.2.1. Handling of Missing and Partial Dates

| Element | Reporting Detail |
|---|---|
| General | Partial dates will be displayed as captured in subject listing displays. |
| Adverse<br>Events | <ul> <li>The eCRF allows for the possibility of partial dates (i.e., only month and year) to be recorded for AE start and end dates; that is, the day of the month may be missing. In such a case, the following conventions will be applied for calculating the time to onset and the duration of the event: <ul> <li>Missing Start Day: First of the month will be used unless this is before the start date of study treatment; in this case the study treatment start date will be used and hence the event is considered On-treatment as per Appendix 4: Study Phases and Treatment Emergent Adverse Events.</li> <li>Missing Stop Day: Last day of the month will be used, unless this is after the stop date of study treatment; in this case the study treatment stop date will be used.</li> </ul> </li> <li>Completely missing start or end dates will remain missing, with no imputation applied. Consequently, time to onset and duration of such events will be missing.</li> </ul> |
| ART/Non-<br>ART<br>Medications<br>/Medical<br>History | <ul> <li>Partial dates recorded in the CRF will be imputed using the following convention: <ul> <li>If the partial date is a start date, a '01' will be used for the day and 'Jan' will be used for the month</li> <li>If the partial date is a stop date, a '28/29/30/31' will be used for the day (dependent on the month and year) and 'Dec' will be used for the month. If medications recorded in the eCRF as prior (e.g. recorded in prior ART or prior ATLAS ART forms, taken prior to study), the earlier date of the imputed and the day prior to the maintenance phase treatment start date will be used, i.e. min (imputed stop date, maintenance phase treatment start date - 1).</li> </ul> </li> <li>For medications with completely missing start date, they will be considered started prior to the maintenance phase treatment start date.</li> <li>For medications with completely missing stop date, they will be considered ongoing unless recorded in eCRF as prior (e.g. recorded in prior ART form, taken prior to study).</li> <li>For ART booster medications, the start and stop dates are not recorded in the database (i.e. missing), the dates will be imputed to be the same as the dates of their parent medications.</li> <li>The recorded partial date will be displayed in listings.</li> </ul> |
| Health | For the summary of individual item scores outputs, missing scores will not be |
| outcomes | computed. |

# 12.8. Appendix 8: Values of Potential Clinical Importance

# 12.8.1. Laboratory Values

| Element | Reporting Detail |
|---|---|
| Laboratory<br>Values and<br>Adverse | The central laboratory will flag lab parameter toxicities directly in the provided datasets based on Division of AIDS Table for Grading the Severity of Adult and Paediatric Adverse Events Version 2.1, March 2017 |
| Events | |

## 12.8.2. ECG

ECG values of potential clinical importance are defined as QTc > 500 msec or increase from baseline in QTc  $\geq$  60 msec.

## 12.9. Appendix 9: Snapshot Algorithm Details

## **Detailed Algorithm Steps**

- Consider an analysis visit window for Month X as defined in Table 8 and Table 9.
- The HIV1-RNA threshold of 50, copies/mL will be analysed, in this study
- The analysis window 'Month 12' and HIV1-RNA threshold of '50 copies/mL' are used for the purpose of illustration. A subject's Snapshot response and reason at Month 12 are categorized as below.
  - HIV1-RNA < **50** copies/mL
  - o HIV1-RNA ≥ **50** copies/mL

Data in window not below 50
Discontinued for lack of efficacy
Discontinued for other reason while not below 50
Change in background therapy\*

Discontinued study for other reasons
On study but missing data in window

 The steps in determining response and reasons are indicated in Table below, in the order stated.

#### **Detailed steps**

Please note that the following scenarios will NOT be penalized Per Snapshot algorithm (i.e. please exclude these scenarios from **Condition** 1-4).

 Dose reduction, dropping a component, or change in formulation (e.g. 'Tivicay + Kivexa' to 'Triumeq' with the identical ingredients)

| Condition ('Month 12' indicates Month 12 window) | Response | Reasons |
|---|---|---|
| If <i>non-permitted</i> change in background therapy <i>prior</i> to Month 12 | HIV1-RNA ≥ 50 | Change in background therapy |
| 2. If <b>permitted</b> change <sup>[a]</sup> in background therapy <b>prior to</b> Month 12 AND the latest on-treatment VL prior to/on the date of change is ≥ 50 c/m (NA to this study) | HIV1-RNA ≥ 50 | Change in background therapy |
| 3: If <i>non-permitted</i> change in background therapy | | |

<sup>\*</sup> Note: since changes in ART are not permitted in this protocol, all such subjects who change ART during the maintenance phase and prior to an analysis timepoint will be considered 'HIV1-RNA ≥ **50** copies/mL'. Participants with protocol permitted oral bridging treatment will not be considered 'HIV-1 RNA ≥ 50 c/mL' due to 'change in ART'.

| during | Month 12 | | |
|---|---|---|---|
| | Last on-treatment VL during Month 12 prior to/on the date of change ≥ 50 c/mL | HIV1-RNA ≥<br>50 | Data in window<br>not below 50 |
| | Last on-treatment VL during Month 12 prior to/on the date of change <50 c/mL | HIV1-RNA <<br>50 | |
| | No VL during Month 12 prior to/on the date of change | HIV1-RNA ≥<br>50 | Change in background therapy |
| Month 1 | mitted change <sup>[a]</sup> in background therapy during 2 AND the last on-treatment VL prior to/on the change is ≥ 50 c/mL (NA to this study) | | |
| 4.1 | this last on-treatment VL occurs prior to Month 12 | HIV1-RNA ≥<br>50 | Change in background therapy |
| | this last on-treatment VL occurs during Month 12 but prior to/on the date of change | HIV1-RNA ≥<br>50 | Data in window<br>not below 50 |
| 5: If non | e of the above conditions met | | |
| 5.1 | VL available during Month 12 | | |
| | Last on-treatment VL during Month 12 ≥ 50 c/mL | HIV1-RNA ≥<br>50 | Data in window<br>not below 50 |
| | <ul> <li>Last on-treatment VL during Month 12 &lt;50<br/>c/mL</li> </ul> | HIV1-RNA <<br>50 | |
| 5.2 | No VL during Month 12 | | |
| permane<br>participa<br>and the<br>to the fo<br>CAB LA<br>Min (ma | subjects still on study i.e. a participant has not ently discontinued the study treatment yet, or if a ant permanently discontinued the study treatment upper bound of analysis snapshot window is prior llowing date: + RPV LA arm: x(Date of last CAB LA + RPV LA injection + 67, last Dose of Oral CAB + RPV + 1), withdrawal date) | No virologic<br>data at Month<br>12 Window | On study but missing data in window |
| | RPV arm:<br>te of Last oral dose of DTG + RPV + 1, withdrawal | | |
| where 'V | Vithdrawal Date' refers to the date the participant | | |

| failed to complete per corresponding conclusion form. | | |
|---|---|---|
| 5.2.2 If subjects withdraw before/during Month 12 due to | | |
| 5.2.2.1 Safety reasons (e.g. AE/death, liver chemistry stopping criteria, renal toxicity withdrawal criteria, QTc withdrawal criteria etc, as recorded in eCRF Conclusion form) | No virologic<br>data at Month<br>12 Window | Disc due to<br>AE/death |
| 5.2.2.2 Non-safety related reasons (e.g. Lack of efficacy, protocol deviation, withdrew consent, loss to follow-up, study closed/terminated, investigator discretion et al, as recorded in eCRF Conclusion Form) | | |
| Last on-treatment VL <50 c/mL OR no on-<br>treatment VL available during study | No virologic<br>Data at Month<br>12 Window | Disc for other reasons |
| Last on-treatment VL ≥ 50 c/mL AND withdrawal due to Lack of efficacy | HIV1-RNA ≥<br>50 | Disc. for lack of efficacy |
| Last on-treatment VL ≥ 50 c/mL AND withdrawal due to all other non-safety related reasons | HIV1-RNA ≥<br>50 | Disc. for other<br>reason while<br>not below 50 |

a: Excluding permitted change in background therapy where change or decision to change is made prior to/on the first on-treatment viral result

#### **Examples from FDA guidance**

#### Data in Window

Virologic outcome should be determined by the last available measurement while the patient is on treatment and continued on trial within the time window:

• HIV-RNA = 580 copies/mL at Day 336, HIV-RNA below 50 copies/mL on Day 350. This should be categorized as HIV-RNA below 50 copies/mL.

#### No Data in Window

Discontinued study due to Adverse Event or Death:

- Any patient who discontinues because of an AE or death before the window should be classified as *Discontinued due to AE or Death* (as appropriate), regardless of the HIV-RNA result, even if the HIV-RNA is below 50 copies/mL at the time of discontinuation.
- However, if a patient has an HIV-RNA value in the time window and also discontinues in the time window, the viral load data should be used to classify the patient's response.
   This is the Virology First hierarchy:
  - a. HIV-RNA below 50 copies/mL at Day 336 and discontinues because of AE or even dies on Day 360 — this person is categorized as having HIV-RNA below 50 copies/mL.
  - b. HIV-RNA is 552 copies/mL on Day 336 and the patient discontinues on Day 360, the patient is categorized as having HIV-RNA greater than or equal to 50

copies/mL.

#### Discontinued for Other Reasons:

- Only patients who have achieved virologic suppression can be counted as *Discontinued* for Other Reasons.
- If a patient discontinues the study before the time window because of *lack of efficacy* then the patient should be included in the HIV-RNA greater than or equal to 50 row and not in the Discontinued for Other Reasons row.
- If a patient discontinues because of subject withdrew consent and his or her HIV-1 RNA
  result at the time of discontinuation was equal to or above 50 copies/mL, then he or she
  should be categorized as HIV-RNA greater than or equal to 50 and NOT as
  Discontinued for Other Reasons.
- If a patient discontinued because of *Lost to Follow-Up* and the last HIV-RNA result was 49 copies/mL, then the patient can be categorized as Discontinued for Other Reasons.
- If patients changed background treatment *not permitted by protocol* they should be captured in the HIV-RNA greater than or equal to 50 copies/mL row.

#### On study but missing data in window:

- If there are no data during Days 294 to 377, but there is an HIV-RNA below 50 copies/mL on Day 380, this patient should be considered *On Study but Missing Data in Window*.
- If there are no data during Days 294 to 377, but there is an HIV-RNA equal to or above 50 copies/mL on Day 280, this patient also should be classified as *On Study but Missing Data in Window.*

# 12.10. Appendix 10: Identification of Adverse Events of Special Interest

The adverse events of special interest are identified based on MedDRA coded values and/or AE data available in the study database. The system organ classes (SOCs), preferred terms (PTs) or codes, Standardised MedDRA Queries (SMQs), High Level Group Terms (HLGTs), and High Level Terms (HLTs) below are from MedDRA 22.0. In case there is a change to the version of MedDRA at time of reporting, the coded values based on the MedDRA version at the time of reporting will be used. The additional events may also be added based on the blinded review of AE data collected on study prior to the database freeze.

#### 1. Hepatic Safety Profile

CMO, 'Hanatia Digardara', CMO Cada, 20000005

Medical concept of hepatic failure and hepatitis. Sub- SMQs (1) 'Hepatic failure, fibrosis and cirrhosis and other liver damage-related conditions' and (2) 'Hepatitis, non-infectious', both of parent SMQ 'Hepatic Disorders'; only narrow terms selected from sub-SMQs. Some preferred terms e.g. PT 'hepatitis fulminant' are duplicated.

| SMQ: 'Hepatic Disorders'; SMQ Code: 20000005<br>Sub-SMQ: 'Hepatic failure, fibrosis and cirrhosis and other liver damage-related conditions'<br>Category: A<br>Scope: Narrow | |
|---|---|
| Preferred Term | PT Code |
| Acquired hepatocerebral degeneration | 10080860 |
| Acute hepatic failure | 10000804 |
| Acute on chronic liver failure | 10077305 |
| Acute yellow liver atrophy | 10070815 |
| Ascites | 10003445 |
| Asterixis | 10003547 |
| Bacterascites | 10068547 |
| Biliary cirrhosis | 10004659 |
| Biliary fibrosis | 10004664 |
| Cardiohepatic syndrome | 10082480 |
| Cholestatic liver injury | 10067969 |
| Chronic hepatic failure | 10057573 |
| Coma hepatic | 10010075 |
| Cryptogenic cirrhosis | 10063075 |

| Diabetic hepatopathy | 10071265 |
|------------------------------------|----------|
| Drug-induced liver injury | 10072268 |
| Duodenal varices | 10051010 |
| Gallbladder varices | 10072319 |
| Gastric variceal injection | 10076237 |
| Gastric variceal ligation | 10076238 |
| Gastric varices | 10051012 |
| Gastric varices haemorrhage | 10057572 |
| Hepatectomy | 10061997 |
| Hepatic atrophy | 10019637 |
| Hepatic calcification | 10065274 |
| Hepatic cirrhosis | 10019641 |
| Hepatic encephalopathy | 10019660 |
| Hepatic encephalopathy prophylaxis | 10066599 |
| Hepatic failure | 10019663 |
| Hepatic fibrosis | 10019668 |
| Hepatic hydrothorax | 10067365 |
| Hepatic infiltration eosinophilic | 10064668 |
| Hepatic lesion | 10061998 |
| Hepatic necrosis | 10019692 |
| Hepatic steato-fibrosis | 10077215 |
| Hepatic steatosis | 10019708 |
| Hepatitis fulminant | 10019772 |
| Hepatobiliary disease | 10062000 |
| Hepatocellular foamy cell syndrome | 10053244 |
| Hepatocellular injury | 10019837 |
| Hepatopulmonary syndrome | 10052274 |
| Hepatorenal failure | 10019845 |
| Hepatorenal syndrome | 10019846 |

| Intestinal varices haemorrhage | Hepatotoxicity | 10019851 |
|---|---|---|
| Liver dialysis 10076640 Liver disorder 10024670 Liver injury 10067125 Liver operation 100224714 Lupoid hepatic cirrhosis 10025125 Minimal hepatic encephalopathy 10066758 Minimal hepatic encephalopathy 10066758 Nodular regenerative hyperplasia 10051081 Nonalcoholic fatty liver disease 10082245 Non-alcoholic steatohepatitis 10053215 Non-cirrhotic portal hypertension 10077255 Oedema due to hepatic disease 10049631 Oesophageal varices haemorrhage 10030210 Peripancreatic varices 1007426 Portal hypertension 1007426 Portal hypertensive colopathy 10068923 Portal hypertensive enteropathy 10068923 Portal vein cavernous transformation 10073205 Portal vein cavernous transformation 10073205 Portopulmonary hypertension 10080267 Portopulmonary hypertension 10073205 Portopulmonary hypertension 10073205 Portopulmonary hypertension 10073205 Portopulmonary hypertension 10073205 Portopulmonary hypertension 10076281 Primary biliary cholangitis 10080425 Regenerative siderotic hepatic nodule 10080675 | Intestinal varices | 10071502 |
| Liver disorder 10024670 Liver injury 10067125 Liver operation 10062040 Liver transplant 10024714 Lupoid hepatic cirrhosis 10025125 Minimal hepatic encephalopathy 10076204 Mixed liver injury 10066758 Nodular regenerative hyperplasia 10051081 Nonalcoholic fatty liver disease 10082245 Non-alcoholic steatohepatitis 10053215 Non-cirrhotic portal hypertension 10077255 Oedema due to hepatic disease 10049631 Oesophageal varices haemorrhage 10030210 Peripancreatic varices 10073215 Portal hypertension 1007426 Portal hypertensive colopathy 1007426 Portal hypertensive enteropathy 10068923 Portal vein cavernous transformation 10073975 Portal vein dilatation 10073205 Portopulmonary hypertension 10067281 Primary biliary cholangitis 10080678 Regenerative siderotic hepatic nodule 10080678 | Intestinal varices haemorrhage | 10078058 |
| Liver injury 10067128 Liver operation 10062040 Liver transplant 10024714 Lupoid hepatic cirrhosis 10025128 Minimal hepatic encephalopathy 10076204 Mixed liver injury 10066758 Nodular regenerative hyperplasia 10051081 Nonalcoholic fatty liver disease 10082249 Non-alcoholic steatohepatitis 10073218 Non-cirrhotic portal hypertension 10077259 Oedema due to hepatic disease 10049631 Oesophageal varices haemorrhage 10030210 Peripancreatic varices 10073218 Portal hypertension 10074726 Portal hypertensive colopathy 10074926 Portal hypertensive enteropathy 10068923 Portal vein cavernous transformation 10073978 Portal vein dilatation 10073208 Portopulmonary hypertension 10067281 Primary biliary cholangitis 10080428 Regenerative siderotic hepatic nodule 10080678 | Liver dialysis | 10076640 |
| Liver operation 10062040 Liver transplant 10024714 Lupoid hepatic cirrhosis 10025129 Minimal hepatic encephalopathy 10076204 Mixed liver injury 10066756 Nodular regenerative hyperplasia 10051081 Nonalcoholic fatty liver disease 10082249 Non-alcoholic steatohepatitis 10053219 Non-cirrhotic portal hypertension 10077259 Oedema due to hepatic disease 10049631 Oesophageal varices haemorrhage 10030210 Peripancreatic varices 10073215 Portal fibrosis 10074726 Portal hypertension 10036200 Portal hypertensive colopathy 1007890 Portal hypertensive enteropathy 10068923 Portal vein cavernous transformation 10073973 Portal vein dilatation 10073208 Portopulmonary hypertension 10067281 Primary biliary cholangitis 10080678 Regenerative siderotic hepatic nodule 10080678 | Liver disorder | 10024670 |
| Liver transplant 10024714 Lupoid hepatic cirrhosis 10025128 Minimal hepatic encephalopathy 10076204 Mixed liver injury 10066758 Nodular regenerative hyperplasia 10051081 Nonalcoholic fatty liver disease 10082248 Non-alcoholic steatohepatitis 10053218 Non-cirrhotic portal hypertension 10077258 Oedema due to hepatic disease 10049631 Oesophageal varices haemorrhage 10030210 Peripancreatic varices 10073215 Portal fibrosis 10074726 Portal hypertension 10036200 Portal hypertensive colopathy 10079446 Portal hypertensive enteropathy 10050897 Portal vein cavernous transformation 10073205 Portal vein dilatation 10073205 Portopulmonary hypertension 10067281 Primary biliary cholangitis 10080425 Regenerative siderotic hepatic nodule 10080679 | Liver injury | 10067125 |
| Lupoid hepatic cirrhosis 10025129 Minimal hepatic encephalopathy 10076204 Mixed liver injury 10066758 Nodular regenerative hyperplasia 10051081 Nonalcoholic fatty liver disease 10082249 Non-alcoholic steatohepatitis 10053219 Non-cirrhotic portal hypertension 10077259 Oedema due to hepatic disease 10049631 Oesophageal varices haemorrhage 10030210 Peripancreatic varices 10073218 Portal fibrosis 10074726 Portal hypertension 10036200 Portal hypertensive colopathy 10079446 Portal hypertensive enteropathy 10058923 Portal vein cavernous transformation 10073208 Portal vein dilatation 10073208 Portal vein dilatation 10067281 Primary biliary cholangitis 10080428 Regenerative siderotic hepatic nodule 10080678 | Liver operation | 10062040 |
| Minimal hepatic encephalopathy 10076204 Mixed liver injury 10066758 Nodular regenerative hyperplasia 10051081 Nonalcoholic fatty liver disease 10082249 Non-alcoholic steatohepatitis 10053219 Non-cirrhotic portal hypertension 10077259 Oedema due to hepatic disease 10049631 Oesophageal varices haemorrhage 10030210 Peripancreatic varices 10073215 Portal fibrosis 10074726 Portal hypertension 10036200 Portal hypertensive colopathy 10079446 Portal hypertensive enteropathy 10068923 Portal vein cavernous transformation 10073205 Portal vein dilatation 10073205 Portal vein dilatation 10073205 Portopulmonary hypertension 10067281 Primary biliary cholangitis 10080425 Regenerative siderotic hepatic nodule 10080675 | Liver transplant | 10024714 |
| Mixed liver injury 10066758 Nodular regenerative hyperplasia 10051081 Nonalcoholic fatty liver disease 10082249 Non-alcoholic steatohepatitis 10053219 Non-cirrhotic portal hypertension 10077259 Oedema due to hepatic disease 10049631 Oesophageal varices haemorrhage 10030210 Peripancreatic varices 10073218 Portal fibrosis 10074726 Portal hypertension 10036200 Portal hypertensive colopathy 10079446 Portal hypertensive enteropathy 10068923 Portal vein cavernous transformation 10073979 Portal vein dilatation 10073209 Portal vein dilatation 10073209 Portopulmonary hypertension 10067281 Primary biliary cholangitis 10080429 Regenerative siderotic hepatic nodule 10080679 | Lupoid hepatic cirrhosis | 10025129 |
| Nodular regenerative hyperplasia 10051081 Nonalcoholic fatty liver disease 10082249 Non-alcoholic steatohepatitis 10053219 Non-cirrhotic portal hypertension 10077259 Oedema due to hepatic disease 10049631 Oesophageal varices haemorrhage 10030210 Peripancreatic varices 10073215 Portal fibrosis 10074726 Portal hypertension 10036200 Portal hypertensive colopathy 10079446 Portal hypertensive enteropathy 10050897 Portal vein cavernous transformation 10073979 Portal vein dilatation 10073209 Portopulmonary hypertension 10067281 Primary biliary cholangitis 10080679 Regenerative siderotic hepatic nodule 10080679 | Minimal hepatic encephalopathy | 10076204 |
| Nonalcoholic fatty liver disease Non-alcoholic steatohepatitis Non-cirrhotic portal hypertension Oedema due to hepatic disease 10049631 Oesophageal varices haemorrhage Peripancreatic varices 10073215 Portal fibrosis Portal hypertension 10079446 Portal hypertensive colopathy Portal hypertensive enteropathy Portal hypertensive gastropathy Portal vein cavernous transformation Portopulmonary hypertension 10073205 Portopulmonary hypertension 10080675 Regenerative siderotic hepatic nodule | Mixed liver injury | 10066758 |
| Non-alcoholic steatohepatitis Non-cirrhotic portal hypertension Oedema due to hepatic disease Oesophageal varices haemorrhage Peripancreatic varices 10073215 Portal fibrosis Portal hypertension Portal hypertensive colopathy Portal hypertensive enteropathy Portal hypertensive gastropathy Portal vein cavernous transformation Portal vein dilatation Portopulmonary hypertension Primary biliary cholangitis Regenerative siderotic hepatic nodule 1007325 1007925 10073215 | Nodular regenerative hyperplasia | 10051081 |
| Non-cirrhotic portal hypertension 10077258 Oedema due to hepatic disease 10049631 Oesophageal varices haemorrhage 10030210 Peripancreatic varices 10073215 Portal fibrosis 10074726 Portal hypertension 10036200 Portal hypertensive colopathy 10068923 Portal hypertensive enteropathy 10050897 Portal vein cavernous transformation 10073208 Portal vein dilatation 10073208 Portopulmonary hypertension 10067281 Primary biliary cholangitis 10080678 | Nonalcoholic fatty liver disease | 10082249 |
| Oedema due to hepatic disease 10049631 Oesophageal varices haemorrhage 10030210 Peripancreatic varices 10073215 Portal fibrosis 10074726 Portal hypertension 10036200 Portal hypertensive colopathy 10079446 Portal hypertensive enteropathy 10068923 Portal hypertensive gastropathy 10050897 Portal vein cavernous transformation 10073203 Portopulmonary hypertension 10067281 Primary biliary cholangitis 10080675 | Non-alcoholic steatohepatitis | 10053219 |
| Oesophageal varices haemorrhage10030210Peripancreatic varices10073215Portal fibrosis10074726Portal hypertension10036200Portal hypertensive colopathy10079446Portal hypertensive enteropathy10068923Portal hypertensive gastropathy10050897Portal vein cavernous transformation10073209Portal vein dilatation10073209Portopulmonary hypertension10067281Primary biliary cholangitis10080429Regenerative siderotic hepatic nodule10080679 | Non-cirrhotic portal hypertension | 10077259 |
| Peripancreatic varices Portal fibrosis Portal hypertension Portal hypertensive colopathy Portal hypertensive enteropathy Portal hypertensive gastropathy Portal vein cavernous transformation Portal vein dilatation Portopulmonary hypertension Primary biliary cholangitis Regenerative siderotic hepatic nodule 10073215 10073215 10074726 10079446 10079446 10068923 10068923 10073205 10073205 10067281 | Oedema due to hepatic disease | 10049631 |
| Portal fibrosis 10074726 Portal hypertension 10036200 Portal hypertensive colopathy 10079446 Portal hypertensive enteropathy 10068923 Portal hypertensive gastropathy 10050897 Portal vein cavernous transformation 10073209 Portopulmonary hypertension 10067281 Primary biliary cholangitis 10080679 Regenerative siderotic hepatic nodule 10080679 | Oesophageal varices haemorrhage | 10030210 |
| Portal hypertension 10036200 Portal hypertensive colopathy 10079446 Portal hypertensive enteropathy 10068923 Portal hypertensive gastropathy 10050897 Portal vein cavernous transformation 10073979 Portal vein dilatation 10073209 Portopulmonary hypertension 10067281 Primary biliary cholangitis 10080429 Regenerative siderotic hepatic nodule 10080679 | Peripancreatic varices | 10073215 |
| Portal hypertensive colopathy Portal hypertensive enteropathy Portal hypertensive gastropathy Portal vein cavernous transformation Portal vein dilatation Portopulmonary hypertension Primary biliary cholangitis Regenerative siderotic hepatic nodule 10079446 10068923 10050897 10073299 10073299 10067281 | Portal fibrosis | 10074726 |
| Portal hypertensive enteropathy Portal hypertensive gastropathy Portal vein cavernous transformation Portal vein dilatation Portopulmonary hypertension Primary biliary cholangitis Regenerative siderotic hepatic nodule 10068923 10050897 10073979 10073209 10067281 | Portal hypertension | 10036200 |
| Portal hypertensive gastropathy Portal vein cavernous transformation Portal vein dilatation Portopulmonary hypertension Primary biliary cholangitis Regenerative siderotic hepatic nodule 10050897 10073209 10073209 10067281 | Portal hypertensive colopathy | 10079446 |
| Portal vein cavernous transformation 10073979 Portal vein dilatation 10073209 Portopulmonary hypertension 10067281 Primary biliary cholangitis 10080429 Regenerative siderotic hepatic nodule 10080679 | Portal hypertensive enteropathy | 10068923 |
| Portal vein dilatation 10073209 Portopulmonary hypertension 10067281 Primary biliary cholangitis 10080429 Regenerative siderotic hepatic nodule 10080679 | Portal hypertensive gastropathy | 10050897 |
| Portopulmonary hypertension 10067281 Primary biliary cholangitis 10080429 Regenerative siderotic hepatic nodule 10080679 | Portal vein cavernous transformation | 10073979 |
| Primary biliary cholangitis 10080429 Regenerative siderotic hepatic nodule 10080679 | Portal vein dilatation | 10073209 |
| Regenerative siderotic hepatic nodule 10080679 | Portopulmonary hypertension | 10067281 |
| | Primary biliary cholangitis | 10080429 |
| Renal and liver transplant 10052279 | Regenerative siderotic hepatic nodule | 10080679 |
| • | Renal and liver transplant | 10052279 |

| Reye's syndrome | 10039012 |
|----------------------------------|----------|
| Povnold's syndromo | |
| Reynold's syndrome | 10070953 |
| Splenic varices | 10067823 |
| Splenic varices haemorrhage | 10068662 |
| Steatohepatitis | 10076331 |
| Subacute hepatic failure | 10056956 |
| Varices oesophageal | 10056091 |
| Varicose veins of abdominal wall | 10072284 |
| White nipple sign | 10078438 |

Category: A Scope: Narrow

| Preferred Term | PT Code |
|--------------------------------------------|----------|
| Acute graft versus host disease in liver | 10066263 |
| Allergic hepatitis | 10071198 |
| Alloimmune hepatitis | 10080576 |
| Autoimmune hepatitis | 10003827 |
| Chronic graft versus host disease in liver | 10072160 |
| Chronic hepatitis | 10008909 |
| Graft versus host disease in liver | 10064676 |
| Hepatitis | 10019717 |
| Hepatitis acute | 10019727 |
| Hepatitis cholestatic | 10019754 |
| Hepatitis chronic active | 10019755 |
| Hepatitis chronic persistent | 10019759 |
| Hepatitis fulminant | 10019772 |
| Hepatitis toxic | 10019795 |
| Immune-mediated hepatitis | 10078962 |

| Ischaemic hepatitis | 10023025 |
|-------------------------------|----------|
| Lupus hepatitis | 10067737 |
| Non-alcoholic steatohepatitis | 10053219 |
| Radiation hepatitis | 10051015 |
| Steatohepatitis | 10076331 |

## 2. Hypersensitivity Reactions (HSR)

Medical concept of hypersensitivity reactions/DRESS. Only narrow terms selected from Category A of SMQ 'Drug reaction with eosinophilia and systemic symptoms syndrome'. Algorithmic approach for this SMQ not used due to complexity in applying and poor specificity of remaining categories. Category A selected as PTs because more specific for concept (only narrow terms) and a pre-requisite for any combination in algorithmic search. Overlap of some preferred terms with SMQ 'Severe Cutaneous Adverse Reactions'. Plus, additional preferred terms selected from HGLT 'Allergic conditions' under SOC 'Immune system disorders.

| SMQ: Drug reaction with eosinophilia and systemic symptoms syndrome SMQ Code: 20000225 Category: A Scope: Narrow | |
|---|---|
| Preferred Term | PT Code |
| Drug reaction with eosinophilia and systemic symptoms | 10073508 |
| Pseudolymphoma | 10037127 |
| Additional preferred terms selected from HLGT 'Allergic conditions' under SOC 'Immune system disorders' | |
| Preferred Term | PT Code |
| Drug hypersensitivity | 10013700 |
| Hypersensitivity | 10020751 |
| Type IV Hypersensitivity reaction | 10053613 |
| Eosinophillia | 10014950 |
| Eye swelling | 10015967 |
| Eyelid oedema | 10015993 |
| Lip swelling | 10024570 |
| Angioedema | 10002424 |

| Circumoral oedema | 10052250 |
|-----------------------|----------|
| Face oedema | 10016029 |
| Idiopathic angioedema | 10073257 |
| Lip oedema | 10024558 |
| Mouth swelling | 10075203 |
| Oedema mouth | 10030110 |
| Periorbital oedema | 10034545 |
| Swelling face | 10042682 |
| Periorbital swelling | 10056647 |
| Swelling of eyelid | 10042690 |

# 3. Rash including severe cutaneous adverse reactions

Medical concept of rash including severe cutaneous adverse reactions. Only narrow terms from SMQ 'Severe cutaneous adverse reactions' selected. Plus several additional preferred terms selected from HLTs 'Rashes, eruptions and exanthems NEC', 'Pruritus NEC', 'Pustular conditions', 'Dermatitis ascribed to specific agent' all under SOC 'Skin and subcutaneous tissue disorders'.

| SMQ: Severe Cutaneous Adverse Reactions SMQ Code: 20000020 Category: A Scope: Narrow | |
|---|---|
| SMQ | PT Code |
| Acute generalised exanthematous pustulosis | 10048799 |
| Cutaneous vasculitis | 10011686 |
| Dermatitis bullous | 10012441 |
| Dermatitis exfoliative | 10012455 |
| Dermatitis exfoliative generalised | 10012456 |
| Drug reaction with eosinophilia and systemic symptoms | 10073508 |
| Epidermal necrosis | 10059284 |
| Erythema multiforme | 10015218 |
| Exfoliative rash | 10064579 |

| Oculomucocutaneous syndrome | 10030081 |
|---|---|
| Skin necrosis | 10040893 |
| Stevens-Johnson syndrome | 10042033 |
| Target skin lesion | 10081998 |
| Toxic epidermal necrolysis | 10044223 |
| Toxic skin eruption | 10057970 |
| Additional preferred terms selected from HLTs 'Rashes, eruptions and exanthems NEC', 'Pruritus NEC', 'Pustular conditions', 'Dermatitis ascribed to specific agent' all under SOC 'Skin and subcutaneous tissue disorders'. | |
| Preferred Term | PT Code |
| Eyelid rash | 10074620 |
| Genital rash | 10018175 |
| Mucocutaneous rash | 10056671 |
| Nodular rash | 10075807 |
| Perineal rash | 10075364 |
| Rash | 10037844 |
| Rash erythematous | 10037855 |
| Rash generalised | 10037858 |
| Rash macular | 10037867 |
| Rash maculo-papular | 10037868 |
| Rash maculovesicular | 10050004 |
| Rash morbilliform | 10037870 |
| Rash papular | 10037876 |
| Rash rubelliform | 10057984 |
| Rash scarlatiniform | 10037890 |
| Rash vesicular | 10037898 |
| Rash pruritic | 10037884 |
| Rash follicular | 10037857 |
| Rash pustular | 10037888 |

## 4. Prolongation of the Corrected QT Interval of the ECG in Supratherapeutic Doses

Notes: Medical concept of QT prolongation and complications. Only narrow terms from SMQ 'Torsade de pointes/QT prolongation' selected plus one additional PT under HLT 'ECG investigations'.

| SMQ: Torsade de pointes/QT prolongation<br>SMQ Code: 20000001<br>Category: A<br>Scope: Narrow | |
|---|---|
| Preferred Term | PT Code |
| Electrocardiogram QT interval abnormal | 10063748 |
| Electrocardiogram QT prolonged | 10014387 |
| Long QT syndrome | 10024803 |
| Long QT syndrome congenital | 10057926 |
| Torsade de pointes | 10044066 |
| Ventricular tachycardia | 10047302 |
| Additional preferred terms selected from HGLT ' ECG investigations' under SOC 'Investigations'. | |
| Preferred Term | PT Code |
| Electrocardiogram repolarisation abnormality | 10052464 |

## 5. Suicidal Ideation/Behaviour

Medical concept of suicidal ideation and behaviour. Sub-SMQ 'Suicide/self-injury' (SMQ) from parent SMQ of 'Depression and Suicide/Self Injury'. Only narrow terms from the sub-SMQ selected.

| SMQ: 'Depression and Suicide/Self Injury' SMQ Code: 20000035 Sub-SMQ: 'Suicide/self-injury' Category: A Scope: Narrow | |
|---|---|
| Preferred Term | PT Code |
| Assisted suicide | 10079105 |
| Columbia suicide severity rating scale abnormal | 10075616 |

| 10010144 |
|----------|
| 10012397 |
| 10022523 |
| 10022524 |
| 10036000 |
| 10051154 |
| 10065604 |
| 10042458 |
| 10042464 |
| 10077417 |
| 10082458 |
| 10081704 |

## 6. Depression

Medical concept of Depression. Sub-SMQ 'Depression (excl suicide and self injury)' (SMQ) from parent SMQ of 'Depression and Suicide/Self Injury'. Only narrow terms from the sub-SMQ selected.

| SMQ: "Depression and Suicide/Self Injury" SMQ Code: 20000035 Sub-SMQ: 'Depression (excl suicide and self injury)' Category: A Scope: Narrow | |
|---|---|
| Preferred Term | PT Code |
| Activation syndrome | 10066817 |
| Adjustment disorder with depressed mood | 10001297 |
| Adjustment disorder with mixed anxiety and depressed mood | 10001299 |
| Agitated depression | 10001496 |
| Anhedonia | 10002511 |
| Antidepressant therapy | 10054976 |
| Childhood depression | 10068631 |
| Decreased interest | 10011971 |

| Depressed mood | 10012374 |
|---------------------------------------|----------|
| Depression | 10012378 |
| Depression postoperative | 10012390 |
| Depressive symptom | 10054089 |
| Dysphoria | 10013954 |
| Electroconvulsive therapy | 10014404 |
| Feeling guilty | 10049708 |
| Feeling of despair | 10016344 |
| Feelings of worthlessness | 10016374 |
| Helplessness | 10077169 |
| Major depression | 10057840 |
| Menopausal depression | 10067371 |
| Mixed anxiety and depressive disorder | 10080836 |
| Perinatal depression | 10078366 |
| Persistent depressive disorder | 10077804 |
| Post stroke depression | 10070606 |
| Postictal depression | 10071324 |

## 7. Bipolar Disorder

Medical concept of bipolar disorder. All preferred terms from HLGT 'Manic and Bipolar mood disorders and disturbances' under SOC 'Psychiatric disorders'.

| Preferred Term | PT Code |
|----------------------|----------|
| Bipolar I disorder | 10004939 |
| Bipolar II disorder | 10004940 |
| Bipolar disorder | 10057667 |
| Cyclothymic disorder | 10011724 |
| Hypomania | 10021030 |
| Mania | 10026749 |

# 8. Psychosis

Medical concept of psychosis. Only narrow terms from SMQ 'Psychosis and psychotic disorders' selected.

| SMQ: 'Psychosis and psychotic disorders' SMQ Code: 20000117 Category: A Scope: Narrow | |
|---|---|
| Preferred Term | PT Code |
| Acute psychosis | 10001022 |
| Alcoholic psychosis | 10001632 |
| Alice in wonderland syndrome | 10001666 |
| Brief psychotic disorder with marked stressors | 10048549 |
| Brief psychotic disorder without marked stressors | 10056395 |
| Brief psychotic disorder, with postpartum onset | 10006362 |
| Charles Bonnet syndrome | 10063354 |
| Childhood psychosis | 10061040 |
| Clang associations | 10009232 |
| Cotard's syndrome | 10059591 |
| Delusion | 10012239 |
| Delusion of grandeur | 10012241 |
| Delusion of reference | 10012244 |
| Delusion of replacement | 10012245 |
| Delusional disorder, erotomanic type | 10012249 |
| Delusional disorder, grandiose type | 10012250 |
| Delusional disorder, jealous type | 10012251 |
| Delusional disorder, mixed type | 10012252 |
| Delusional disorder, persecutory type | 10053195 |
| Delusional disorder, somatic type | 10012254 |
| Delusional disorder, unspecified type | 10012255 |
| Delusional perception | 10012258 |

| Dementia of the Alzheimer's type, with delusions | 10012295 |
|--------------------------------------------------|----------|
| Depressive delusion | 10063033 |
| Derailment | 10012411 |
| Epileptic psychosis | 10059232 |
| Erotomanic delusion | 10015134 |
| Flight of ideas | 10016777 |
| Hallucination | 10019063 |
| Hallucination, auditory | 10019070 |
| Hallucination, gustatory | 10019071 |
| Hallucination, olfactory | 10019072 |
| Hallucination, synaesthetic | 10062824 |
| Hallucination, tactile | 10019074 |
| Hallucination, visual | 10019075 |
| Hallucinations, mixed | 10019079 |
| Hypnagogic hallucination | 10020927 |
| Hypnopompic hallucination | 10020928 |
| Hysterical psychosis | 10062645 |
| Ideas of reference | 10021212 |
| Illusion | 10021403 |
| Jealous delusion | 10023164 |
| Loose associations | 10024825 |
| Mixed delusion | 10076429 |
| Neologism | 10028916 |
| Neuroleptic-induced deficit syndrome | 10075295 |
| Paranoia | 10033864 |
| Paranoid personality disorder | 10033869 |
| Parkinson's disease psychosis | 10074835 |
| Paroxysmal perceptual alteration | 10063117 |
| Persecutory delusion | 10034702 |

| Post-injection delirium sedation syndrome 10070669 Post-injection delirium sedation syndrome 10072851 Posturing 10036437 Psychosis postoperative 10065617 Psychotic behaviour 10037249 Psychotic disorder 10061920 Psychotic disorder due to a general medical condition 10061921 Reactive psychosis 10053632 Rebound psychosis 10074833 Schizoaffective disorder 10039621 Schizoaffective disorder bipolar type 10068890 Schizophrenia 10039626 Schizophreniform disorder 10039647 Schizotypal personality disorder 10039651 Senile psychotic disorder 10040535 |
|---|
| Posturing 10036437 Psychosis postoperative 10065617 Psychotic behaviour 10037249 Psychotic disorder 10061920 Psychotic disorder due to a general medical condition 10061921 Reactive psychosis 10053632 Rebound psychosis 10074833 Schizoaffective disorder 10039621 Schizoaffective disorder bipolar type 10068889 Schizoaffective disorder depressive type 10068890 Schizophrenia 10039626 Schizophreniform disorder 10039651 Senile psychosis 10039987 Shared psychotic disorder 10040535 |
| Psychosis postoperative 10065617 Psychotic behaviour 10037249 Psychotic disorder 10061920 Psychotic disorder due to a general medical condition 10061921 Reactive psychosis 10053632 Rebound psychosis 10074833 Schizoaffective disorder 10039621 Schizoaffective disorder 10068889 Schizoaffective disorder depressive type 10068890 Schizophrenia 10039626 Schizophreniform disorder 10039647 Schizotypal personality disorder 10039987 Shared psychotic disorder 10040535 |
| Psychotic behaviour 10037249 Psychotic disorder 10061920 Psychotic disorder due to a general medical condition 10061921 Reactive psychosis 10053632 Rebound psychosis 10074833 Schizoaffective disorder 10039621 Schizoaffective disorder bipolar type 10068899 Schizoaffective disorder depressive type 10068890 Schizophrenia 10039626 Schizophrenia 10039647 Schizotypal personality disorder 10039987 Shared psychotic disorder 10040535 |
| Psychotic disorder 10061920 Psychotic disorder due to a general medical condition 10061921 Reactive psychosis 10053632 Rebound psychosis 10074833 Schizoaffective disorder 10039621 Schizoaffective disorder bipolar type 10068889 Schizoaffective disorder depressive type 10068890 Schizophrenia 10039626 Schizophreniform disorder 10039647 Schizotypal personality disorder 10039987 Shared psychotic disorder 10040535 |
| Psychotic disorder due to a general medical condition Reactive psychosis Rebound psychosis 10074833 Schizoaffective disorder 10039621 Schizoaffective disorder bipolar type 10068889 Schizoaffective disorder depressive type 10068890 Schizophrenia 10039626 Schizophreniform disorder 10039647 Schizotypal personality disorder 10039987 Shared psychotic disorder 10040535 |
| Reactive psychosis 10053632 Rebound psychosis 10074833 Schizoaffective disorder 10039621 Schizoaffective disorder bipolar type 10068889 Schizoaffective disorder depressive type 10068890 Schizophrenia 10039626 Schizophreniform disorder 10039647 Schizotypal personality disorder 10039651 Senile psychosis 10039987 Shared psychotic disorder 10040535 |
| Rebound psychosis 10074833 Schizoaffective disorder 10039621 Schizoaffective disorder bipolar type 10068889 Schizoaffective disorder depressive type 10068890 Schizophrenia 10039626 Schizophreniform disorder 10039647 Schizotypal personality disorder 10039651 Senile psychosis 10039987 Shared psychotic disorder 10040535 |
| Schizoaffective disorder10039621Schizoaffective disorder bipolar type10068889Schizoaffective disorder depressive type10068890Schizophrenia10039626Schizophreniform disorder10039647Schizotypal personality disorder10039651Senile psychosis10039987Shared psychotic disorder10040535 |
| Schizoaffective disorder bipolar type Schizoaffective disorder depressive type 10068890 Schizophrenia 10039626 Schizophreniform disorder 10039647 Schizotypal personality disorder 10039651 Senile psychosis 10039987 Shared psychotic disorder 10040535 |
| Schizoaffective disorder depressive type Schizophrenia 10039626 Schizophreniform disorder 10039647 Schizotypal personality disorder Senile psychosis 10039987 Shared psychotic disorder 10040535 |
| Schizophrenia 10039626 Schizophreniform disorder 10039647 Schizotypal personality disorder 10039651 Senile psychosis 10039987 Shared psychotic disorder 10040535 |
| Schizophreniform disorder 10039647 Schizotypal personality disorder 10039651 Senile psychosis 10039987 Shared psychotic disorder 10040535 |
| Schizotypal personality disorder 10039651 Senile psychosis 10039987 Shared psychotic disorder 10040535 |
| Senile psychosis 10039987 Shared psychotic disorder 10040535 |
| Shared psychotic disorder 10040535 |
| 0 5 11 5 |
| Somatic delusion 10041317 |
| Somatic hallucination 10062684 |
| Substance-induced psychotic disorder 10072388 |
| Tangentiality 10043114 |
| Thought blocking 10043495 |
| Thought broadcasting 10052214 |
| Thought insertion 10043496 |
| Thought withdrawal 10043497 |
| Transient psychosis 10056326 |
| Waxy flexibility 10047853 |

# 9. Mood Disorders

Medical concept of mood disorders. All preferred terms from HLGT 'Mood disorders and disturbances NEC', under SOC 'Psychiatric disorders'.

| Preferred Term | PT Code |
|----------------------------------|----------|
| Affect lability | 10054196 |
| Affective ambivalence | 10077173 |
| Affective disorder | 10001443 |
| Alexithymia | 10077719 |
| Anger | 10002368 |
| Apathy | 10002942 |
| Blunted affect | 10005885 |
| Boredom | 10048909 |
| Constricted affect | 10010778 |
| Crying | 10011469 |
| Diencephalic syndrome of infancy | 10012774 |
| Dysphoria | 10013954 |
| Emotional disorder | 10014551 |
| Emotional distress | 10049119 |
| Emotional poverty | 10014557 |
| Euphoric mood | 10015535 |
| Flat affect | 10016759 |
| Frustration tolerance decreased | 10077753 |
| Inappropriate affect | 10021588 |
| Irritability | 10022998 |
| Laziness | 10051602 |
| Lethargy | 10024264 |
| Listless | 10024642 |
| Moaning | 10027783 |
| Mood altered | 10027940 |

| Mood disorder due to a general medical condition | 10027944 |
|--------------------------------------------------|----------|
| Mood swings | 10027951 |
| Morose | 10027977 |
| Neuroleptic-induced deficit syndrome | 10075295 |
| Premenstrual dysphoric disorder | 10051537 |
| Premenstrual syndrome | 10036618 |
| Screaming | 10039740 |
| Seasonal affective disorder | 10039775 |
| Steroid withdrawal syndrome | 10042028 |
| Substance-induced mood disorder | 10072387 |

# 10. Anxiety

Notes: Medical concept of anxiety disorders. All preferred terms from HLGT "Anxiety disorders and symptoms", under SOC "Psychiatric disorders".

| Preferred Terms | PT Code |
|-------------------------|----------|
| Acrophobia | 10000605 |
| Activation syndrome | 10066817 |
| Acute stress disorder | 10001084 |
| Aerophobia | 10080300 |
| Agitation | 10001497 |
| Agitation postoperative | 10049989 |
| Agoraphobia | 10001502 |
| Akathisia | 10001540 |
| Algophobia | 10078056 |
| Animal phobia | 10002518 |
| Anniversary reaction | 10074066 |
| Anticipatory anxiety | 10002758 |
| Anxiety | 10002855 |
| Anxiety disorder | 10057666 |

| Anxiety disorder due to a general medical condition | 10002859 |
|-----------------------------------------------------|----------|
| Arachnophobia | 10051408 |
| Astraphobia | 10078372 |
| Autophobia | 10071070 |
| Body dysmorphic disorder | 10052793 |
| Burnout syndrome | 10065369 |
| Catastrophic reaction | 10082329 |
| Cibophobia | 10082413 |
| Claustrophobia | 10009244 |
| Compulsions | 10010219 |
| Compulsive cheek biting | 10076510 |
| Compulsive handwashing | 10071263 |
| Compulsive hoarding | 10068007 |
| Compulsive lip biting | 10066241 |
| Compulsive shopping | 10067948 |
| Dermatillomania | 10065701 |
| Dysmorphophobia | 10049096 |
| Emetophobia | 10070637 |
| Fear | 10016275 |
| Fear of animals | 10016276 |
| Fear of closed spaces | 10016277 |
| Fear of crowded places | 10050365 |
| Fear of death | 10066392 |
| Fear of disease | 10016278 |
| Fear of eating | 10050366 |
| Fear of falling | 10048744 |
| Fear of injection | 10073753 |
| Fear of open spaces | 10016279 |
| Fear of pregnancy | 10067035 |

| Fear of weight gain | 10016280 |
|---|---|
| Fear-related avoidance of activities | 10080136 |
| Generalised anxiety disorder | 10018075 |
| Glossophobia | 10080077 |
| Haemophobia | 10073458 |
| Haphephobia | 10067580 |
| Herpetophobia | 10081809 |
| Hydrophobia | 10053317 |
| Hyperarousal | 10080831 |
| Immunisation anxiety related reaction | 10075205 |
| Kinesiophobia | 10078430 |
| Limited symptom panic attack | 10024511 |
| Mysophobia | 10078769 |
| Nail picking | 10066779 |
| Nervousness | 10029216 |
| Neurosis | 10029333 |
| Noctiphobia | 10057946 |
| Nocturnal fear | 10057948 |
| Nosophobia | 10063546 |
| Obsessive need for symmetry | 10077179 |
| Obsessive rumination | 10056264 |
| Obsessive thoughts | 10029897 |
| Obsessive-compulsive disorder | 10029898 |
| Obsessive-compulsive symptom | 10077894 |
| Ochlophobia | 10050095 |
| Osmophobia | 10060765 |
| Paediatric autoimmune neuropsychiatric disorders associated with streptococcal infection | 10072147 |
| Panic attack | 10033664 |

| Panic disorder | 10033666 |
|--------------------------------|----------|
| Panic reaction | 10033670 |
| Paruresis | 10069024 |
| Performance fear | 10034432 |
| Phagophobia | 10050096 |
| Pharmacophobia | 10069423 |
| Phobia | 10034912 |
| Phobia of driving | 10056676 |
| Phobia of exams | 10034913 |
| Phobic avoidance | 10034918 |
| Phonophobia | 10054956 |
| Photaugiaphobia | 10064420 |
| Postpartum anxiety | 10082233 |
| Postpartum neurosis | 10036419 |
| Postpartum stress disorder | 10056394 |
| Post-traumatic stress disorder | 10036316 |
| Procedural anxiety | 10075204 |
| Pseudoangina | 10056610 |
| Selective mutism | 10039917 |
| Separation anxiety disorder | 10040045 |
| Sitophobia | 10080170 |
| Social anxiety disorder | 10041242 |
| Social fear | 10041247 |
| Stress | 10042209 |
| Tension | 10043268 |
| Terminal agitation | 10077416 |
| Thanatophobia | 10064723 |
| Thermophobia | 10075147 |
| Trichotemnomania | 10072752 |

| Trichotillomania | 10044629 |
|------------------|----------|
|------------------|----------|

## 11. Sleep Disorders

Medical concept of sleep disorders. All preferred terms from (1) HLGT 'Sleep Disorders and Disturbances', 'Psychiatric disorders' SOC plus (2) HLGT 'Sleep disturbances (including subtypes)', 'Nervous system' SOC. Numerous duplicated preferred terms e.g. middle insomnia.

| HLGT Sleep Disorders and Disturbances, HLGT Code 10040991 | |
|-----------------------------------------------------------|----------|
| Preferred Term | PT Code |
| Abnormal dreams | 10000125 |
| Abnormal sleep-related event | 10061613 |
| Advanced sleep phase | 10001423 |
| Behavioural induced insufficient sleep syndrome | 10081938 |
| Behavioural insomnia of childhood | 10072072 |
| Breathing-related sleep disorder | 10006344 |
| Cataplexy | 10007737 |
| Circadian rhythm sleep disorder | 10009191 |
| Confusional arousal | 10067494 |
| Delayed sleep phase | 10012209 |
| Dyssomnia | 10061827 |
| Exploding head syndrome | 10080684 |
| Hypersomnia | 10020765 |
| Hypersomnia related to another mental condition | 10020767 |
| Hypersomnia-bulimia syndrome | 10053712 |
| Hypnagogic hallucination | 10020927 |
| Hypnopompic hallucination | 10020928 |
| Hyposomnia | 10067530 |
| Initial insomnia | 10022035 |
| Insomnia | 10022437 |
| Insomnia related to another mental condition | 10022443 |

| Irregular sleep phase | 10022995 |
|-------------------------------------------------------------------|----------|
| Irregular sleep wake rhythm disorder | 10080301 |
| Loss of dreaming | 10065085 |
| Middle insomnia | 10027590 |
| Narcolepsy | 10028713 |
| Nightmare | 10029412 |
| Non-24-hour sleep-wake disorder | 10078086 |
| Parasomnia | 10061910 |
| Periodic limb movement disorder | 10064600 |
| Pickwickian syndrome | 10035004 |
| Poor quality sleep | 10062519 |
| Rapid eye movement sleep behaviour disorder | 10077299 |
| Rapid eye movements sleep abnormal | 10037841 |
| Shift work disorder | 10078088 |
| Sleep apnoea syndrome | 10040979 |
| Sleep attacks | 10040981 |
| Sleep disorder | 10040984 |
| Sleep disorder due to a general medical condition | 10063910 |
| Sleep disorder due to general medical condition, hypersomnia type | 10040985 |
| Sleep disorder due to general medical condition, insomnia type | 10040986 |
| Sleep disorder due to general medical condition, mixed type | 10040987 |
| Sleep disorder due to general medical condition, parasomnia type | 10040988 |
| Sleep inertia | 10067493 |
| Sleep paralysis | 10041002 |
| Sleep sex | 10067492 |
| Sleep talking | 10041009 |
| Sleep terror | 10041010 |
| Sleep-related eating disorder | 10067315 |
| Somnambulism | 10041347 |
| | • |

| Somnolence | 10041349 |
|-------------------------------------------------------------|----------|
| Somnolence neonatal | 10041350 |
| Sopor | 10058709 |
| Stupor | 10042264 |
| Terminal insomnia | 10068932 |
| Upper airway resistance syndrome | 10063968 |
| HLGT Sleep disturbances (incl subtypes), HLGT code 10040998 | |
| Abnormal dreams | 10000125 |
| Abnormal sleep-related event | 10061613 |
| Advanced sleep phase | 10001423 |
| Behavioural induced insufficient sleep syndrome | 10081938 |
| Behavioural insomnia of childhood | 10072072 |
| Breathing-related sleep disorder | 10006344 |
| Cataplexy | 10007737 |
| Central-alveolar hypoventilation | 10007982 |
| Circadian rhythm sleep disorder | 10009191 |
| Confusional arousal | 10067494 |
| Delayed sleep phase | 10012209 |
| Dyssomnia | 10061827 |
| Fatal familial insomnia | 10072077 |
| Hypersomnia | 10020765 |
| Hyposomnia | 10067530 |
| Initial insomnia | 10022035 |
| Insomnia | 10022437 |
| Irregular sleep phase | 10022995 |
| Irregular sleep wake rhythm disorder | 10080301 |
| Loss of dreaming | 10065085 |
| Microsleep | 10076954 |
| Middle insomnia | 10027590 |

| | • |
|---------------------------------------------|----------|
| Narcolepsy | 10028713 |
| Non-24-hour sleep-wake disorder | 10078086 |
| Periodic limb movement disorder | 10064600 |
| Pickwickian syndrome | 10035004 |
| Poor quality sleep | 10062519 |
| Rapid eye movement sleep behaviour disorder | 10077299 |
| Rapid eye movements sleep abnormal | 10037841 |
| Shift work disorder | 10078088 |
| Sleep apnoea syndrome | 10040979 |
| Sleep deficit | 10080881 |
| Sleep inertia | 10067493 |
| Sleep paralysis | 10041002 |
| Sleep sex | 10067492 |
| Sleep talking | 10041009 |
| Sleep terror | 10041010 |
| Sleep-related eating disorder | 10067315 |
| Somnambulism | 10041347 |
| Sudden onset of sleep | 10050014 |
| Terminal insomnia | 10068932 |
| Upper airway resistance syndrome | 10063968 |

## 12. Injection Site Reactions (ISR) from Study Drug Injections

Study drug ISR data available in the database, i.e. data collected from non-serious ISR AE eCRF form and collected serious adverse events with 'STUDY DRUG INJECTION SITE' included in the AE term.

#### 13. Seizures

Medical concept of seizures. Only narrow terms from SMQ 'Convulsions' selected plus selected PTs of possible seizure events from HLT 'Disturbances in consciousness NEC' under SOC 'Nervous systems disorders' and HLT 'Confusion and disorientation' under SOC 'Psychiatric disorders'.

| SMQ: 'Convulsions' SMQ Code: 20000079 Category: A Scope: Narrow | |
|-----------------------------------------------------------------|----------|
| Preferred Term | PT Code |
| 1p36 deletion syndrome | 10082398 |
| 2-Hydroxyglutaric aciduria | 10078971 |
| Acquired epileptic aphasia | 10052075 |
| Acute encephalitis with refractory, repetitive partial seizures | 10076948 |
| Alcoholic seizure | 10056347 |
| Aspartate-glutamate-transporter deficiency | 10079140 |
| Atonic seizures | 10003628 |
| Atypical benign partial epilepsy | 10056699 |
| Automatism epileptic | 10003831 |
| Autonomic seizure | 10049612 |
| Baltic myoclonic epilepsy | 10054895 |
| Benign familial neonatal convulsions | 10067866 |
| Benign rolandic epilepsy | 10070530 |
| Biotinidase deficiency | 10071434 |
| Change in seizure presentation | 10075606 |
| Clonic convulsion | 10053398 |
| Convulsion in childhood | 10052391 |
| Convulsions local | 10010920 |
| Convulsive threshold lowered | 10010927 |
| CSWS syndrome | 10078827 |
| Deja vu | 10012177 |
| Double cortex syndrome | 10073490 |
| Dreamy state | 10013634 |
| Drug withdrawal convulsions | 10013752 |
| Early infantile epileptic encephalopathy with burst-suppression | 10071545 |

| Eclampsia | 10014129 |
|------------------------------------------------|----------|
| Epilepsy | 10015037 |
| Epilepsy surgery | 10079824 |
| Epilepsy with myoclonic-atonic seizures | 10081179 |
| Epileptic aura | 10015049 |
| Epileptic psychosis | 10059232 |
| Febrile convulsion | 10016284 |
| Febrile infection-related epilepsy syndrome | 10079438 |
| Focal dyscognitive seizures | 10079424 |
| Frontal lobe epilepsy | 10049424 |
| Generalised non-convulsive epilepsy | 10018090 |
| Generalised tonic-clonic seizure | 10018100 |
| Glucose transporter type 1 deficiency syndrome | 10078727 |
| Grey matter heterotopia | 10082084 |
| Hemimegalencephaly | 10078100 |
| Hyperglycaemic seizure | 10071394 |
| Hypocalcaemic seizure | 10072456 |
| Hypoglycaemic seizure | 10048803 |
| Hyponatraemic seizure | 10073183 |
| Idiopathic generalised epilepsy | 10071081 |
| Infantile spasms | 10021750 |
| Juvenile myoclonic epilepsy | 10071082 |
| Lafora's myoclonic epilepsy | 10054030 |
| Lennox-Gastaut syndrome | 10048816 |
| Migraine-triggered seizure | 10076676 |
| Molybdenum cofactor deficiency | 10069687 |
| Multiple subpial transection | 10079825 |
| Myoclonic epilepsy | 10054859 |
| Myoclonic epilepsy and ragged-red fibres | 10069825 |

| Partial seizures 10061334 Partial seizures with secondary generalisation 10056209 Petit mal epilepsy 10034759 Polymicrogyria 10073489 Post stroke epilepsy 10076982 Post stroke seizure 10076981 Postictal headache 10052470 Postictal paralysis 10052469 Postictal psychosis 10070669 Postictal state 10048727 Post-traumatic epilepsy 10036312 Schizencephaly 10073487 Seizure 10039906 Seizure anoxic 10039907 Seizure cluster 10071048 Severe myoclonic epilepsy of infancy 10071048 Severe myoclonic epilepsy of infancy 10040703 Status epilepticus 10040703 Status epilepticus 10040703 Status epilepticus 10043209 Tonic clonic movements 10051171 Tonic convulsion 10043209 Tonic convulsion 10075125 Topectomy 10073488 Transient epileptic amnesia | Neonatal epileptic seizure | 10082068 |
|---|---|---|
| Partial seizures with secondary generalisation 10056209 Petit mal epilepsy 10034759 Polymicrogyria 10073489 Post stroke epilepsy 10076982 Post stroke seizure 10076981 Postictal headache 10052470 Postictal paralysis 10052469 Postictal psychosis 10070669 Post-traumatic epilepsy 10036312 Schizencephaly 10073487 Seizure 10039906 Seizure anoxic 10039907 Seizure cluster 10071350 Seizure like phenomena 10071048 Severe myoclonic epilepsy of infancy 10073677 Simple partial seizures 10040703 Status epilepticus 10040703 Status epilepticus 10043209 Tonic clonic movements 10051171 Tonic convulsion 10043994 Tonic posturing 10073488 Transient epileptic amnesia 10081728 | Neonatal seizure | 10082067 |
| Petit mal epilepsy 10034759 Polymicrogyria 10073489 Post stroke epilepsy 10076982 Post stroke seizure 10076981 Postictal headache 10052470 Postictal paralysis 10052469 Postictal psychosis 10070669 Postictal state 10048727 Post-traumatic epilepsy 10036312 Schizencephaly 10073487 Seizure 10039906 Seizure anoxic 10039907 Seizure cluster 10071350 Seizure like phenomena 10071048 Severe myoclonic epilepsy of infancy 10073677 Simple partial seizures 10040703 Status epilepticus 10040703 Status epilepticus 10043209 Temporal lobe epilepsy 10063894 Temporal lobe epilepsy 10043209 Tonic clonic movements 10051171 Tonic posturing 10075125 Topectomy 10073488 Transient epileptic amnesia 10081728 | Partial seizures | 10061334 |
| Polymicrogyria 10073489 Post stroke epilepsy 10076982 Post stroke seizure 10076981 Postictal headache 10052470 Postictal paralysis 10052469 Postictal psychosis 10070669 Post-traumatic epilepsy 10036312 Schizencephaly 10073487 Seizure 10039906 Seizure anoxic 10039907 Seizure cluster 10071350 Seizure like phenomena 10071048 Severe myoclonic epilepsy of infancy 10073677 Simple partial seizures 10040703 Status epilepticus 10040703 Status epilepticus 10040703 Temporal lobe epilepsy 10063894 Temporal lobe epilepsy 10043209 Tonic clonic movements 10051171 Tonic posturing 10075125 Topectomy 10073488 Transient epileptic amnesia 10081728 | Partial seizures with secondary generalisation | 10056209 |
| Post stroke epilepsy 10076982 Post stroke seizure 10076981 Post ictal headache 10052470 Postictal paralysis 10052469 Postictal psychosis 10070669 Postictal state 10048727 Post-traumatic epilepsy 10036312 Schizencephaly 10073487 Seizure 10039906 Seizure anoxic 10039907 Seizure cluster 10071350 Seizure like phenomena 10071048 Severe myoclonic epilepsy of infancy 10073677 Simple partial seizures 10040703 Status epilepticus 10040703 Status epilepticus 10043209 Tonic clonic movements 10051171 Tonic clonic movements 10051171 Tonic convulsion 10043994 Tonic posturing 10073488 Transient epileptic amnesia 10081728 | Petit mal epilepsy | 10034759 |
| Post stroke seizure 10076981 Postictal headache 10052470 Postictal paralysis 10052469 Postictal psychosis 10070669 Postictal state 10048727 Post-traumatic epilepsy 10036312 Schizencephaly 10073487 Seizure 10039906 Seizure anoxic 10039907 Seizure cluster 10071048 Severe myoclonic epilepsy of infancy 10073677 Simple partial seizures 10040703 Status epilepticus 10040703 Status epilepticus 10043994 Temporal lobe epilepsy 10043209 Tonic clonic movements 10051171 Tonic convulsion 10043994 Tonic posturing 10073488 Transient epileptic amnesia 10081728 | Polymicrogyria | 10073489 |
| Postictal headache 10052470 Postictal paralysis 10052469 Postictal psychosis 10070669 Postictal state 10048727 Post-traumatic epilepsy 10036312 Schizencephaly 10073487 Seizure 10039906 Seizure anoxic 10039907 Seizure cluster 10071350 Seizure like phenomena 10071048 Severe myoclonic epilepsy of infancy 10073677 Simple partial seizures 10040703 Status epilepticus 10040703 Status epilepticus 10043994 Temporal lobe epilepsy 10043994 Tonic clonic movements 10043994 Tonic posturing 10075125 Topectomy 10073488 Transient epileptic amnesia 10081728 | Post stroke epilepsy | 10076982 |
| Postictal paralysis 10052469 Postictal psychosis 10070669 Postictal state 10048727 Post-traumatic epilepsy 10036312 Schizencephaly 10073487 Seizure 10039906 Seizure anoxic 10039907 Seizure cluster 10071350 Seizure like phenomena 10071048 Severe myoclonic epilepsy of infancy 10073677 Simple partial seizures 10040703 Status epilepticus 10041962 Sudden unexplained death in epilepsy 10063894 Temporal lobe epilepsy 10043209 Tonic clonic movements 10051171 Tonic convulsion 10043994 Tonic posturing 10075125 Topectomy 10073488 Transient epileptic amnesia 10081728 | Post stroke seizure | 10076981 |
| Postictal psychosis 10070669 Postictal state 10048727 Post-traumatic epilepsy 10036312 Schizencephaly 10073487 Seizure 10039906 Seizure anoxic 10039907 Seizure cluster 10071350 Seizure like phenomena 10071048 Severe myoclonic epilepsy of infancy 10073677 Simple partial seizures 10040703 Status epilepticus 10041962 Sudden unexplained death in epilepsy 10063894 Temporal lobe epilepsy 10051171 Tonic clonic movements 10051171 Tonic convulsion 10043994 Tonic posturing 10075125 Topectomy 10073488 Transient epileptic amnesia 10081728 | Postictal headache | 10052470 |
| Postictal state 10048727 Post-traumatic epilepsy 10036312 Schizencephaly 10073487 Seizure 10039906 Seizure anoxic 10039907 Seizure cluster 10071350 Seizure like phenomena 10071048 Severe myoclonic epilepsy of infancy 10073677 Simple partial seizures 10040703 Status epilepticus 10041962 Sudden unexplained death in epilepsy 10063894 Temporal lobe epilepsy 10051171 Tonic clonic movements 10051171 Tonic convulsion 10043994 Tonic posturing 10075125 Topectomy 10073488 Transient epileptic amnesia 10081728 | Postictal paralysis | 10052469 |
| Post-traumatic epilepsy 10036312 Schizencephaly 10073487 Seizure 10039906 Seizure anoxic 10039907 Seizure cluster 10071350 Seizure like phenomena 10071048 Severe myoclonic epilepsy of infancy 10073677 Simple partial seizures 10040703 Status epilepticus 10041962 Sudden unexplained death in epilepsy 10063894 Temporal lobe epilepsy 10043209 Tonic clonic movements 10051171 Tonic convulsion 10043994 Tonic posturing 10075125 Topectomy 10073488 Transient epileptic amnesia 10081728 | Postictal psychosis | 10070669 |
| Schizencephaly 10073487 Seizure 10039906 Seizure anoxic 10039907 Seizure cluster 10071350 Seizure like phenomena 10071048 Severe myoclonic epilepsy of infancy 10073677 Simple partial seizures 10040703 Status epilepticus 10041962 Sudden unexplained death in epilepsy 10063894 Temporal lobe epilepsy 10043209 Tonic clonic movements 10051171 Tonic convulsion 10043994 Tonic posturing 10075125 Topectomy 10073488 Transient epileptic amnesia 10081728 | Postictal state | 10048727 |
| Seizure 10039906 Seizure anoxic 10039907 Seizure cluster 10071350 Seizure like phenomena 10071048 Severe myoclonic epilepsy of infancy 10073677 Simple partial seizures 10040703 Status epilepticus 10041962 Sudden unexplained death in epilepsy 10063894 Temporal lobe epilepsy 10043209 Tonic clonic movements 10051171 Tonic convulsion 10043994 Tonic posturing 10075125 Topectomy 10073488 Transient epileptic amnesia 10081728 | Post-traumatic epilepsy | 10036312 |
| Seizure anoxic 10039907 Seizure cluster 10071350 Seizure like phenomena 10071048 Severe myoclonic epilepsy of infancy 10073677 Simple partial seizures 10040703 Status epilepticus 10041962 Sudden unexplained death in epilepsy 10063894 Temporal lobe epilepsy 10043209 Tonic clonic movements 10051171 Tonic convulsion 10043994 Tonic posturing 10075125 Topectomy 10073488 Transient epileptic amnesia 10081728 | Schizencephaly | 10073487 |
| Seizure cluster 10071350 Seizure like phenomena 10071048 Severe myoclonic epilepsy of infancy 10073677 Simple partial seizures 10040703 Status epilepticus 10041962 Sudden unexplained death in epilepsy 10063894 Temporal lobe epilepsy 10043209 Tonic clonic movements 10051171 Tonic convulsion 10043994 Tonic posturing 10075125 Topectomy 10073488 Transient epileptic amnesia 10081728 | Seizure | 10039906 |
| Seizure like phenomena 10071048 Severe myoclonic epilepsy of infancy 10073677 Simple partial seizures 10040703 Status epilepticus 10041962 Sudden unexplained death in epilepsy 10063894 Temporal lobe epilepsy 10043209 Tonic clonic movements 10051171 Tonic convulsion 10043994 Tonic posturing 10075125 Topectomy 10081728 | Seizure anoxic | 10039907 |
| Severe myoclonic epilepsy of infancy Simple partial seizures 10040703 Status epilepticus 10041962 Sudden unexplained death in epilepsy Temporal lobe epilepsy Tonic clonic movements 10051171 Tonic convulsion 10043294 Tonic posturing 10075125 Topectomy Transient epileptic amnesia | Seizure cluster | 10071350 |
| Simple partial seizures 10040703 Status epilepticus 10041962 Sudden unexplained death in epilepsy 10063894 Temporal lobe epilepsy 10043209 Tonic clonic movements 10051171 Tonic convulsion 10043994 Tonic posturing 10075125 Topectomy 10073488 Transient epileptic amnesia 10081728 | Seizure like phenomena | 10071048 |
| Status epilepticus 10041962 Sudden unexplained death in epilepsy 10063894 Temporal lobe epilepsy 10043209 Tonic clonic movements 10051171 Tonic convulsion 10043994 Tonic posturing 10075125 Topectomy 10073488 Transient epileptic amnesia 10081728 | Severe myoclonic epilepsy of infancy | 10073677 |
| Sudden unexplained death in epilepsy Temporal lobe epilepsy Tonic clonic movements Tonic convulsion Tonic posturing Topectomy Topectomy Transient epileptic amnesia 10063894 10043209 10051171 10043294 10075125 10073488 | Simple partial seizures | 10040703 |
| Temporal lobe epilepsy Tonic clonic movements 10051171 Tonic convulsion 10043209 Tonic convulsion 10043994 Tonic posturing 10075125 Topectomy 10073488 Transient epileptic amnesia 10081728 | Status epilepticus | 10041962 |
| Tonic clonic movements 10051171 Tonic convulsion 10043994 Tonic posturing 10075125 Topectomy 10073488 Transient epileptic amnesia 10081728 | Sudden unexplained death in epilepsy | 10063894 |
| Tonic convulsion 10043994 Tonic posturing 10075125 Topectomy 10073488 Transient epileptic amnesia 10081728 | Temporal lobe epilepsy | 10043209 |
| Tonic posturing 10075125 Topectomy 10073488 Transient epileptic amnesia 10081728 | Tonic clonic movements | 10051171 |
| Topectomy 10073488 Transient epileptic amnesia 10081728 | Tonic convulsion | 10043994 |
| Transient epileptic amnesia 10081728 | Tonic posturing | 10075125 |
| · · · | Topectomy | 10073488 |
| Tuberous sclerosis complex 10080584 | Transient epileptic amnesia | 10081728 |
| | Tuberous sclerosis complex | 10080584 |

| Uncinate fits | 10045476 |
|---|---|
| Additional selected preferred terms from HLT 'Disturbances in consciousness NEC' under SOC 'Nervous systems disorders' and HLT 'Confusion and disorientation' under SOC 'Psychiatric disorders'. | |
| Preferred Term | PT Code |
| Confusional state | 10010305 |
| Loss of consciousness | 10024855 |
| Syncope | 10042772 |
| Sopor | 10058709 |
| Stupor | 10042264 |
| Altered state of consciousness | 10001854 |
| Depressed level of consciousness | 10012373 |
| Consciousness fluctuating | 10050093 |

## 14. Weight Gain

Medical concept of weight gain. Selected PTs from HLT 'General nutritional disorders NEC', under SOC 'Metabolism and nutrition disorders', and HLT 'Physical examination procedures and organ system status', under SOC 'Investigations' and HLT 'General signs and symptoms NEC', under SOC 'General disorders and administration site conditions'.

| Preferred Term | PT Code |
|-------------------------------|----------|
| Abdominal fat apron | 10077983 |
| Overweight | 10033307 |
| Abnormal weight gain | 10000188 |
| Central obesity | 10065941 |
| Obesity | 10029883 |
| Weight abnormal | 10056814 |
| Weight increased | 10047899 |
| Waist circumference increased | 10064863 |
| Body mass index abnormal | 10074506 |
| Body mass index increased | 10005897 |
| Fat tissue increased | 10016251 |

## 15. Rhabdomyolysis

Medical concept of rhabdomyolysis. Only narrow terms only for SMQ 'Rhabdomyolysis/myopathy' plus 2 additional preferred terms selected from HGLT 'muscle disorders' under SOC 'Musculoskeletal and connective tissue disorders'.

| SMQ: 'Rhabdomyolysis/myopathy' SMQ Code: 20000002 Category: A Scope: Narrow | |
|---|---|
| Preferred Term | PT Code |
| Muscle necrosis | 10028320 |
| Myoglobin blood increased | 10028625 |
| Myoglobin blood present | 10059888 |
| Myoglobin urine present | 10028631 |
| Myoglobinaemia | 10058735 |
| Myoglobinuria | 10028629 |
| Myopathy | 10028641 |
| Myopathy toxic | 10028648 |
| Necrotising myositis | 10074769 |
| Rhabdomyolysis | 10039020 |
| Thyrotoxic myopathy | 10081524 |
| Additional selected preferred terms from HLGT 'muscle disorders' under SOC 'Musculoskeletal and connective tissue disorders' | |
| Preferred Term | PT Code |
| Myalgia | 10028411 |
| Myositis | 10028653 |

#### 16. Pancreatitis

Medical concept of acute pancreatitis. Only narrow terms of SMQ 'Acute pancreatitis' selected. Algorithmic approach for this SMQ not used due to complexity in applying and poor specificity of remaining categories. Category A selected as PTs because more specific for concept (only narrow terms).

| SMQ: 'Acute pancreatitis' SMQ Code: 20000022 Category: A Scope: Narrow | |
|---|---|
| Preferred Term | PT Code |
| Cullen's sign | 10059029 |
| Grey Turner's sign | 10075426 |
| Haemorrhagic necrotic pancreatitis | 10076058 |
| Hereditary pancreatitis | 10056976 |
| Ischaemic pancreatitis | 10066127 |
| Oedematous pancreatitis | 10052400 |
| Pancreatic abscess | 10048984 |
| Pancreatic cyst drainage | 10082531 |
| Pancreatic haemorrhage | 10033625 |
| Pancreatic necrosis | 10058096 |
| Pancreatic phlegmon | 10056975 |
| Pancreatic pseudoaneurysm | 10081762 |
| Pancreatic pseudocyst | 10033635 |
| Pancreatic pseudocyst drainage | 10033636 |
| Pancreatitis | 10033645 |
| Pancreatitis acute | 10033647 |
| Pancreatitis haemorrhagic | 10033650 |
| Pancreatitis necrotising | 10033654 |
| Pancreatitis relapsing | 10033657 |
| Pancreatorenal syndrome | 10056277 |

## 17. Impact on Creatinine

Medical concept of worsening renal function/renal failure in the context of impact on creatinine. Only narrow terms from SMQ 'Acute renal failure' plus all PTs from HLT 'Renal failure and impairment', under SOC 'Renal and urinary disorders'. Numerous duplicated preferred terms e.g. renal failure.
| SMQ: 'Acute renal failure' SMQ Code: 20000003 Category: A Scope: Narrow | |
|---|---|
| Preferred Term | PT Code |
| Acute kidney injury | 10069339 |
| Acute phosphate nephropathy | 10069688 |
| Anuria | 10002847 |
| Azotaemia | 10003885 |
| Continuous haemodiafiltration | 10066338 |
| Dialysis | 10061105 |
| Foetal renal impairment | 10078987 |
| Haemodialysis | 10018875 |
| Haemofiltration | 10053090 |
| Neonatal anuria | 10049778 |
| Nephropathy toxic | 10029155 |
| Oliguria | 10030302 |
| Peritoneal dialysis | 10034660 |
| Prerenal failure | 10072370 |
| Renal failure | 10038435 |
| Renal failure neonatal | 10038447 |
| Renal impairment | 10062237 |
| Renal impairment neonatal | 10049776 |
| Subactute kidney injury | 10081980 |
| Plus, all PTs from HLT 'Renal failure and impairment' under SOC 'Renal and urinary disorders' | |
| Preferred Term | PT Code |
| Acute Kidney injury | 10069339 |
| Anuria | 10002847 |
| Atypical haemolytic uraemic syndrome | 10079840 |

| Cardiorenal syndrome | 10068230 |
|----------------------------------|----------|
| Chronic kidney disease | 10064848 |
| Crush syndrome | 10050702 |
| Diabetic end stage renal disease | 10012660 |
| End stage renal disease | 10077512 |
| Foetal renal impairment | 10078987 |
| Haemolytic uraemic syndrome | 10018932 |
| Hepatorenal failure | 10019845 |
| Hepatorenal syndrome | 10019846 |
| Nail-patella syndrome | 10063431 |
| Neonatal anuria | 10049778 |
| Oliguria | 10030302 |
| Pancreatorenal syndrome | 10056277 |
| Postoperative renal failure | 10056675 |
| Postrenal failure | 10059345 |
| Prerenal failure | 10072370 |
| Propofol infusion syndrome | 10063181 |
| Renal failure | 10038435 |
| Renal failure neonatal | 10038447 |
| Renal impairment | 10062237 |
| Renal impairment neonatal | 10049776 |
| Renal injury | 10061481 |
| Scleroderma renal crisis | 10062553 |
| Traumatic anuria | 10044501 |
| | · |

#### 18. Safety in Pregnancy

Use AE terms co-reported in pregnancy exposures to CAB and/or RPV.

# 12.11. Appendix 11: Abbreviations & Trade Marks

#### 12.11.1. Abbreviations

| Abbreviation | Description |
|---|---|
| ADaM | • |
| | Analysis Data Model Adverse Event |
| AEGI | |
| AESI | Adverse Events of Special Interest |
| ART | Antiretroviral Therapy |
| A&R | Analysis and Reporting |
| BMI | Body Mass index |
| CAB | Cabotegravir |
| CDISC | Clinical Data Interchange Standards Consortium |
| CI | Confidence Interval |
| CPMS | Clinical Pharmacology Modelling & Simulation |
| CS | Clinical Statistics |
| CSR | Clinical Study Report |
| CTR | Clinical Trial Register |
| DBF | Database Freeze |
| DBR | Database Release |
| DOB | Date of Birth |
| DP | Decimal Places |
| DTG | Dolutegravir |
| eCRF | Electronic Case Record Form |
| EMA | European Medicines Agency |
| FDA | Food and Drug Administration |
| FDAAA | Food and Drug Administration Clinical Results Disclosure Requirements |
| GSK | GlaxoSmithKline |
| HIVDQoL | HIV Dependent Quality of Life |
| HIV | Human Immunodeficiency Virus |
| HIVTSQc | Change Version of HIV Treatment Satisfaction Questionnaire |
| HIVTSQs | Status Version of HIV Treatment Satisfaction Questionnaire |
| HLGT | High Level Group Term |
| HLT | High Level Term |
| HSR | Hypersensitivity Reaction |
| IA | Interim Analysis |
| ICH | International Conference on Harmonization |
| IDSL | Integrated Data Standards Library |
| INI | Integrase Inhibitors |
| IP | Investigational Product |
| ITT | Intent-To-Treat |
| ITT-E | Intent-To-Treat Exposed |
| NA | Not Applicable |
| NCEP | National Cholesterol Education Program |
| NNRTI | Non-Nucleoside Reverse Transcriptase Inhibitors |
| NRTI | Nucleoside Reverse Transcriptase Inhibitors |
| PCI | Potential Clinical Importance |
| PDMP | Protocol Deviation Management Plan |
| PI | Protease Inhibitors |
| PK | Pharmacokinetic |
| LIV | r natmacokineuc |

| Abbreviation | Description |
|--------------|--------------------------------------------------|
| PP | Per Protocol |
| PT | Preferred Term |
| QC | Quality Control |
| QTcF | Frederica's QT Interval Corrected for Heart Rate |
| QTcB | Bazett's QT Interval Corrected for Heart Rate |
| RAP | Reporting & Analysis Plan |
| RPV | Rilpivirine |
| SAE | Serious Adverse Event |
| SAC | Statistical Analysis Complete |
| SD | Standard Deviation |
| SDTM | Study Data Tabulation Model |
| SMQ | Standardised MedDRA Query |
| SOC | System Organ Class |
| SOP | Standard Operation Procedure |
| TA | Therapeutic Area |
| TFL | Tables, Figures & Listings |

#### 12.11.2. Trademarks

| Trademarks of the GlaxoSmithKline<br>Group of Companies |
|---------------------------------------------------------|
| Dolutegravir |
| Triumeq |

| Trademarks not owned by the GlaxoSmithKline Group of Companies |
|----------------------------------------------------------------|
| Rilpivirine |
| SAS |

#### 12.12. Appendix 12: List of Data Displays

#### 12.12.1. Data Display Numbering

The following numbering will be applied for RAP generated displays:

| Section | Tables | Figures |
|------------------|-------------|-------------|
| Study Population | 1.01 to 1.n | 1.01 to 1.n |
| Efficacy | 2.01 to 2.n | 2.01 to 2.n |
| Safety | 3.01 to 3.n | 3.01 to 3.n |
| Health Outcomes | 6.01 to 6.n | 6.01 to 6.n |
| Virology | 7.01 to 7.n | 7.01 to 7.n |
| Section | Listings | |
| ICH Listings | 1 to x | |
| Other Listings | y to z | |

#### 12.12.2. Mock Example Shell Referencing

Non IDSL specifications will be referenced as indicated and if required example mock-up displays provided in Appendix 13: Example Mock Shells for Data Displays.

The example mock-up displays from other reporting efforts will be named in the format: Study Number/HARP Reporting Effort/Output Type (T/F/L)/Display Number, where T stands for Table, F stands for Figure and L stands for Listing. For example, the Table 1.1 from primary\_02 reporting effort for Study 201585 will be named by 201585/primary 02/T1.1.

Other example mock-up displays will be named using the following format.

| Section | Figure | Table | Listing |
|------------------|---------|---------|---------|
| Study Population | POP_Fn | POP_Tn | POP_Ln |
| Efficacy | EFF_Fn | EFF_Tn | EFF_Ln |
| Safety | SAFE_Fn | SAFE_Tn | SAFE_Ln |
| Health Outcomes | HO_Fn | HO_Tn | HO_Ln |
| Virology | VIR_Fn | VIR_Tn | VIR_Ln |

NOTES:

Non-Standard displays are indicated in the 'IDSL / Example Shell' or 'Programming Notes' column.'

#### 12.12.3. Deliverables

| Delivery [1] | Description |
|--------------|---------------------------------------------------------|
| HL | Headline |
| M12 | All participants complete Month 12 |
| M26 | All participants on CAB LA + RPV LA complete Month 26 * |
| EOS | End of Study |

#### NOTES:

<sup>\*</sup>M26 and EOS analyses might not be produced

<sup>1.</sup> Indicates priority (i.e. order) in which displays will be generated for the reporting effort

## 12.12.4. Study Population Tables

| Study | IDSL/ | | | | |
|---|---|---|---|---|---|
| No. | Population | Example<br>Shell | Title | Programming Notes | Deliverable |
| Subje | t Disposition | | | | |
| 1.01. | ITT-E | ES5 | Summary of Reasons for Withdrawal at Each Study Phase | Replace 'Epoch' with 'Phase' in column header. Screening Phase will not be included. Add a footnote "Note: Entry into Long-Term Follow-up is based on presence of a long-term follow-up visit in the eCRF (i.e. LTFU Month 1, LTFU Month 3, etc.)" | M12, M26,<br>EOS |
| 1.02. | ITT-E | ES4 | Summary of Subject Disposition at Each Study Phase | | M12, M26,<br>EOS |
| 1.03. | Screened | ES6 | Summary of Screening Status and Reasons for Screening Failures | | M12, M26,<br>EOS |
| 1.04. | Enrolled | NS1 | Summary of Number of Subjects Enrolled by Country and Site ID | | M12, M26,<br>EOS |
| 1.05. | ITT-E | DV1 | Summary of Important Protocol Deviations | | M12, M26,<br>EOS |
| 1.06. | Screened | 207966/pri<br>mary_02/T<br>1.12 | Summary of Study Populations | | M12, M26,<br>EOS |

| Study | Study Population Tables | | | | |
|---|---|---|---|---|---|
| No. | Population | IDSL /<br>Example<br>Shell | Title | Programming Notes | Deliverable |
| 1.07. | ITT-E | 207966/pri<br>mary_02/T<br>1.13 | Summary of Protocol Deviations Leading to Exclusion from the Per-Protocol Population | | M12, M26,<br>EOS |
| 1.08. | ITT-E | ES1 | Summary of Subject Accountability: Study Conclusion Record | | HL, M12, M26,<br>EOS |
| 1.09. | ITT-E | 207966/pri<br>mary_02/T<br>1.8 | Summary of Subject Accountability: Withdrawals by Visit | | M12, M26,<br>EOS |
| 1.10. | ITT-E | 207966/pri<br>mary_02/T<br>1.9 | Summary of Study Drug Discontinuation | | M12, M26,<br>EOS |
| 1.11. | ITT-E | 207966/pri<br>mary_02/T<br>1.11 | Summary of Inclusion/Exclusion Criteria Deviations | | M12, M26,<br>EOS |
| Demog | raphic and B | aseline Chara | cteristics | | |
| 1.12. | ITT-E | 207966/pri<br>mary_02/T<br>1.14 | Summary of Demographic Characteristics | | HL, M12, M26,<br>EOS |
| 1.13. | Enrolled | 207966/pri<br>mary_02/T<br>1.15 | Summary of Age Ranges | | M12, M26,<br>EOS |
| 1.14. | ITT-E | DM5 | Summary of Race and Racial Combinations | | M12, M26,<br>EOS |

| Study | Study Population Tables | | | | |
|---|---|---|---|---|---|
| No. | Population | IDSL /<br>Example<br>Shell | Title | Programming Notes | Deliverable |
| 1.15. | ITT-E | DM6 | Summary of Race and Racial Combinations Details | | M12, M26,<br>EOS |
| 1.16. | ITT-E | 207966/pri<br>mary_02/T<br>1.18 | Summary of Hepatitis Status at Entry | | M12, M26,<br>EOS |
| 1.17. | ITT-E | 207966/pri<br>mary_02/T<br>1.19 | Summary of Derived Baseline CDC Stages of HIV Infection | | M12, M26,<br>EOS |
| 1.18. | ITT-E | 207966/pri<br>mary_02/T<br>1.21 | Distribution of CD4+ Cell Count Results at Baseline | Do not include 'Screening' | M12, M26,<br>EOS |
| 1.19. | ITT-E | 207966/pri<br>mary_02/T<br>1.23 | Summary of HIV Risk Factors | | M12, M26,<br>EOS |
| Medica | l Conditions | and Medication | ons | | |
| 1.20. | ITT-E | MH1 | Summary of Current Medical Conditions | | M12, M26,<br>EOS |
| 1.21. | ITT-E | MH1 | Summary of Past Medical Conditions | | M12, M26,<br>EOS |
| 1.22. | ITT-E | MH4 | Summary of Current Cardiac, Gastrointestinal, Metabolism and Nutrition, Psychiatric, Renal and Urinary, Nervous System Conditions, and Hepatobiliary Disorders | | M12, M26,<br>EOS |

| Study | Study Population Tables | | | | |
|---|---|---|---|---|---|
| No. | Population | IDSL /<br>Example<br>Shell | Title | Programming Notes | Deliverable |
| 1.23. | ITT-E | MH4 | Summary of Past Cardiac, Gastrointestinal, Metabolism and Nutrition, Psychiatric, Renal and Urinary, Nervous System Conditions, and Hepatobiliary Disorders | | M12, M26,<br>EOS |
| 1.24. | ITT_E | CM8 | Summary of Concomitant Non-ART Medication Ingredient Combinations | | M12, M26,<br>EOS |
| 1.25. | ITT-E | 207966/pri<br>mary_02/T<br>1.30 | Summary of Lipid Modifying Agent Use at Baseline | | M12, M26,<br>EOS |
| 1.26. | ITT-E | 207966/pri<br>mary_02/T<br>1.31 | Summary of Lipid Modifying Agent Use Started during the Maintenance Phase | | M12, M26,<br>EOS |
| 1.27. | ITT-E | 207966/pri<br>mary_02/T<br>1.32 | Summary of Substance Use at Entry | | M12, M26,<br>EOS |
| Expos | ure and Treatr | nent Complia | ince | • | |
| 1.28. | Safety | 207966/pri<br>mary_02/T<br>3.1 | Summary of Extent of Exposure to Investigational Product | | M12, M26,<br>EOS |
| 1.29. | Safety | 207966/pri<br>mary_02/T<br>3.4 | Summary of Adherence to CAB/RPV Injection Dosing Schedule | Only display for Q2M | M12, M26,<br>EOS |

# 12.12.5. Efficacy Tables

| Efficac | Efficacy: Tables | | | | |
|---|---|---|---|---|---|
| No. | Population | IDSL /<br>Example<br>Shell | Title | Programming Notes | Deliverable |
| Primar | y Efficacy An | alyses | | | • |
| 2.01. | ITT-E | 207966/primar<br>y_02/T2.3 | Summary of Study Outcomes (50 c/mL Threshold) at Month 12 – Snapshot Analysis – ITT-E | For M26, replace the 'Month 12' in the title with 'Month 26' | HL, M12, M26,<br>EOS |
| 2.02. | PP | 207966/primar<br>y_02/T2.3 | Summary of Study Outcomes (50 c/mL Threshold) at Month 12 – Snapshot Analysis – Per-Protocol | For M26, replace the 'Month 12' in the title with 'Month 26' | M12, M26,<br>EOS |
| Secon | dary and Expl | oratory Efficacy | Analyses | | |
| 2.03. | ITT-E | 207966/primar<br>y_02/T2.13 | Proportion of Subjects with Plasma HIV-1 RNA >=50 c/mL by Visit – Snapshot Analysis | | M12, M26,<br>EOS |
| 2.04. | ITT-E | 207966/primar<br>y_02/T2.14 | Proportion of Subjects with Plasma HIV-1 RNA >=50 c/mL by Subgroup and Visit – Snapshot Analysis | | M12, M26,<br>EOS |
| 2.05. | ITT-E | 207966/primar<br>y_02/T2.15 | Proportion of Subjects with Plasma HIV-1 RNA <50 c/mL by Visit – Snapshot Analysis | | M12, M26,<br>EOS |
| 2.06. | ITT-E | 207966/primar<br>y_02/T2.16 | Proportion of Subjects with Plasma HIV-1 RNA <50 c/mL by Subgroup and Visit – Snapshot Analysis | | M12, M26,<br>EOS |
| 2.07. | ITT-E | 207966/primar<br>y_02/T2.22 | Summary of Plasma HIV-1 RNA (log10 c/mL) by Visit | | M12, M26,<br>EOS |
| 2.08. | ITT-E | 207966/primar<br>y_02/T2.23 | Cumulative Proportion of Subjects Meeting Confirmed Virologic Failure Criteria by Visit during the Maintenance Phase (Up to Month 12) | For M26, replace the 'Month 12' in the title with 'Month 26' | M12, M26,<br>EOS |
| 2.09. | ITT-E | 207966/primar<br>y_02/T2.24 | Cumulative Proportion of Subjects Meeting Confirmed Virologic Failure Criteria | | M12, M26,<br>EOS |

| Efficac | Efficacy: Tables | | | | |
|---|---|---|---|---|---|
| No. | Population | IDSL /<br>Example<br>Shell | Title | Programming Notes | Deliverable |
| 2.10. | CVF | 207966/primar<br>y_02/T2.25 | Distribution of Quantitative Plasma HIV-1 RNA Results at Suspected and Confirmation of Confirmed Virologic Failure | | M12, M26,<br>EOS |
| 2.11. | ITT-E | 207966/primar<br>y_02/T2.28 | Summary of Subjects per Viral Load Category by Visit | | M12, M26,<br>EOS |
| 2.12. | ITT-E | 207966/primar<br>y_02/T2.29 | Summary of Change from Baseline in CD4+ Cell Count (cells/mm^3) by Visit | | M12, M26,<br>EOS |
| 2.13. | ITT-E | 207966/primar<br>y_02/T2.31 | Summary of CD4+ Cell Count (cells/mm^3) by Visit | | M12, M26,<br>EOS |
| 2.14. | ITT-E | 207966/primar<br>y_02/T2.35 | Summary of HIV-1 Associated Conditions Including Recurrences | | M12, M26,<br>EOS |
| 2.15. | ITT-E | 207966/primar<br>y_02/T2.36 | Summary of HIV-1 Associated Conditions Excluding Recurrences | | M12, M26,<br>EOS |
| 2.16. | ITT-E | 207966/primar<br>y_02/T2.37 | Summary of HIV-1 Disease Progression and/or Deaths | | M12, M26,<br>EOS |
| 2.17. | ITT-E | 207966/primar<br>y_02/T2.22 | Summary of Change from Baseline in Plasma HIV-1 RNA (log10 c/mL) by Visit | Add footnote: "Note: Baseline values are actual plasma HIV-1 RNA (log10 c/mL) values." Display actual values at Baseline and change from baseline for post-baseline visits | M12, M26,<br>EOS |

# 12.12.6. Efficacy Figures

| Efficac | Efficacy: Figures | | | | |
|---|---|---|---|---|---|
| No. | Population | IDSL /<br>Example<br>Shell | Title | Programming Notes | Deliverable |
| Primar | y Efficacy Ana | alyses | | | |
| 2.01. | ITT-E | 207966/primar<br>y_02/F2.1 | Proportion (95% CI) of Subjects with HIV-1 RNA >=50 c/mL by Visit - Snapshot Analysis | | M12, M26,<br>EOS |
| Second | dary and Expl | oratory Efficacy | Analyses | | |
| 2.02. | ITT-E | 207966/primar<br>y_02/F2.3 | Proportion (95% CI) of Subjects with HIV-1 RNA <50 c/mL by Visit - Snapshot Analysis | | M12, M26,<br>EOS |
| 2.03. | ITT-E | 207966/primar<br>y_02/F2.7 | Individual Plasma HIV-1 RNA (log10 c/mL) Profiles by Visit – for CVF Subjects | | M12, M26,<br>EOS |
| 2.04. | ITT-E | 207966/primar<br>y_02/F2.8 | Individual Plasma HIV-1 RNA (log10 c/mL) Profiles by Visit for Subjects Who are in the Category of 'HIV-1 RNA >=50 c/mL' at Month 12 per Snapshot Algorithm | For M26, replace the 'Month 12' in the title with 'Month 26' | M12, M26,<br>EOS |

# 12.12.7. Safety Tables

| Safety | Safety: Tables | | | | |
|---|---|---|---|---|---|
| No. | Population | IDSL /<br>Example<br>Shell | Title | Programming Notes | Deliverable |
| Advers | e Events (AE | s) | | | |
| 3.01. | Safety | AE1 | Summary of All Adverse Events by System Organ Class and Preferred Term | | M12, M26,<br>EOS |
| 3.02. | Safety | AE3 | Summary of Common (>=5%) Adverse Events by Overall Frequency | | M12, M26,<br>EOS |
| 3.03. | Safety | AE3 | Summary of Common (>=1%) Grade 2-4 Adverse Events by Overall Frequency | | M12, M26,<br>EOS |
| 3.04. | Safety | AE1 | Summary All Drug-Related Adverse Events by System Organ Class | | M12, M26,<br>EOS |
| 3.05. | Safety | 207966/primar<br>y_02/T3.25 | Summary of Subjects and Number of Occurrences of Common (>=5%) Non-Serious Adverse Events by System Organ Class | Add footnote: 'Note: Common adverse events are those with >=5% incidence in either treatment group. | M12, M26,<br>EOS |
| 3.06. | Safety | AE3 | Summary of Common (>=1%) Drug-Related Grade 2-4<br>Adverse Events by Overall Frequency | Add footnote: 'Note: Common adverse events are those with >=1% incidence in either treatment group. | M12, M26,<br>EOS |
| 3.07. | Safety | 207966/prima<br>yr_02/T3.26 | Summary of Subjects and Number of Occurrences of SAEs, Fatal SAEs, and Drug-related SAEs | | HL, M12, M26,<br>EOS |

| Safety | : Tables | | | | |
|---|---|---|---|---|---|
| No. | Population | IDSL /<br>Example<br>Shell | Title | Programming Notes | Deliverable |
| Other | Significant Ad | verse Events | | | |
| 3.08. | Safety | AE1 | Summary of Adverse Events Leading to Withdrawal/Permanent Discontinuation of Investigational Product by System Organ Class | | HL, M12, M26,<br>EOS |
| Labora | atory: Chemis | try and Hematol | ogy | | • |
| 3.09. | Safety | 207966/primar<br>y_02/T3.39 | Summary of Chemistry Changes from Baseline by Visit | | M12, M26,<br>EOS |
| 3.10. | Safety | 207966/primar<br>y_02/T3.41 | Summary of Hematology Changes from Baseline by Visit | | M12, M26,<br>EOS |
| Labora | tory: Urinalys | sis | | | • |
| 3.11. | Safety | 207966/primar<br>y_02/T3.48 | Summary of Urine Concentration Changes from Baseline by Visit | | M12, M26,<br>EOS |
| Labora | atory: Hepatok | oiliary (Liver) | | | |
| 3.12. | Safety | LIVER1 | Summary of Liver Monitoring/Stopping Event Reporting | | M12, M26,<br>EOS |
| 3.13. | Safety | 207966/primar<br>y_02/T3.57 | Summary of Subjects Meeting Hepatobiliary Abnormality Criteria | | M12, M26,<br>EOS |

| Safety | Safety: Tables | | | | |
|---|---|---|---|---|---|
| No. | Population | IDSL /<br>Example<br>Shell | Title | Programming Notes | Deliverable |
| ECG | | | | | |
| 3.14. | Safety | EG1 | Summary of ECG Findings | | M12, M26,<br>EOS |
| 3.15. | Safety | 207966/primar<br>y_02/T3.61 | Summary of QTc Values by Category | | M12, M26,<br>EOS |
| 3.16. | Safety | 207966/primar<br>y_02/T3.62 | Summary of Change from Baseline QTc Values by Category | | M12, M26,<br>EOS |
| Vital S | igns | | | | |
| 3.17. | Safety | VS1 | Summary of Change from Baseline in Vital Signs by Visit | | M12, M26,<br>EOS |
| Study | Drug Injection | Site Reaction A | dverse Events (display for Q2M arm only) | | |
| 3.18. | Safety | 207966/primar<br>y_02/T3.28 | Summary of Study Drug Injection Site Reaction Adverse Events (Event-level Summary) | | HL, M12, M26,<br>EOS |
| 3.19. | Safety | 207966/primar<br>y_02/T3.29 | Summary of Subject-level Characteristics of Study Drug<br>Injection Site Reaction Adverse Events – Overall and<br>Common | | M12, M26,<br>EOS |
| 3.20. | Safety | 207966/primar<br>y_02/T3.30 | Summary of Study Drug Injection Site Reaction Adverse<br>Events by Visit and Maximum Severity – Overall and<br>Common | Replace definition of common in the footnote with 'Note: Common ISR includes pain, induration, nodules and any other ISR with >=5% subjects in Q2M treatment arm' | M12, M26,<br>EOS |

| Safety | Safety: Tables | | | | |
|---|---|---|---|---|---|
| No. | Population | IDSL /<br>Example<br>Shell | Title | Programming Notes | Deliverable |
| 3.21. | Safety | 207966/primar<br>y_02/T3.31 | Summary of Drug-related Study Drug Injection Site<br>Reaction Adverse Events (Event-level Summary) – CAB | | M12, M26,<br>EOS |
| 3.22. | Safety | 207966/primar<br>y_02/T3.32 | Summary of Drug-related Subject-level Characteristics of Study Drug Injection Site Reaction Adverse Events – Overall and Common (CAB) | | M12, M26,<br>EOS |
| 3.23. | Safety | 207966/primar<br>y_02/T3.33 | Summary of Overall and Common Drug-related Study Drug<br>Injection Site Reaction Adverse Events by Visit and<br>Maximum Severity – CAB | | M12, M26,<br>EOS |
| 3.24. | Safety | 207966/primar<br>y_02/T3.34 | Summary of Maximum Drug-related Study Drug Injection<br>Site Reaction Adverse Event Grade by Needle Length –<br>Common (CAB) | Replace definition of common in the footnote with 'Note: Common ISR includes pain, induration, nodules and any other ISR with >=5% subjects in Q2M treatment arm' | M12, M26,<br>EOS |
| 3.25. | Safety | 207966/primar<br>y_02/T3.35 | Summary of Drug-related Study Drug Injection Site Reaction Adverse Events (Event-level Summary) – RPV | | M12, M26,<br>EOS |
| 3.26. | Safety | 207966/primar<br>y_02/T3.36 | Summary of Drug-related Subject-level Characteristics of Study Drug Injection Site Reaction Adverse Events – Overall and Common (RPV) | | M12, M26,<br>EOS |
| 3.27. | Safety | 207966/primar<br>y_02/T3.37 | Summary of Overall and Common Drug-related Study Drug<br>Injection Site Reaction Adverse Events by Visit and<br>Maximum Severity – RPV | | M12, M26,<br>EOS |

| Safety: | Safety: Tables | | | | |
|---|---|---|---|---|---|
| No. | Population | IDSL /<br>Example<br>Shell | Title | Programming Notes | Deliverable |
| 3.28. | Safety | 207966/primar<br>y_02/T3.38 | Summary of Maximum Drug-related Study Drug Injection<br>Site Reaction Adverse Event Grade by Needle Length –<br>Common (RPV) | Replace definition of common in the footnote with 'Note: Common ISR includes pain, induration, nodules and any other ISR with >=5% subjects in Q2M treatment arm' | M12, M26,<br>EOS |
| Advers | e Events of S | pecial Interest | | | |
| 3.29. | Safety | 207966/primar<br>y_02/T3.72 | Summary of Depression Adverse Events of Special<br>Interest by System Organ Class and Preferred Term<br>(Number of Subjects and Occurrences) | | M12, M26,<br>EOS |
| 3.30. | Safety | 207966/primar<br>y_02/T3.76 | Summary of Anxiety Adverse Events of Special Interest by System Organ Class and Preferred Term (Number of Subjects and Occurrences) | | M12, M26,<br>EOS |
| 3.31. | Safety | 207966/primar<br>y_02/T3.71 | Summary of Suicidal Ideation/Behaviour Adverse Events of<br>Special Interest by System Organ Class and Preferred<br>Term (Number of Subjects and Occurrences) | | M12, M26,<br>EOS |
| 3.32. | Safety | 207966/primar<br>y_02/T3.66 | Summary of Depression, Anxiety and Suicidal Ideation/Behaviour Adverse Events by System Organ Class, Maximum DAIDS Toxicity Grade, and History of Depression, Anxiety and Suicidal Ideation/Behaviour at Baseline | For M26 and EOS, include additional stratification by 'any history' vs. 'no history' | M12, M26,<br>EOS |
| 3.33. | Safety | 207966/primar<br>y_02/T3.78 | Summary of Seizure Adverse Events of Special Interest by<br>System Organ Class and Preferred Term (Number of<br>Subjects and Occurrences) | | M12, M26,<br>EOS |

| Safety | Safety: Tables | | | | |
|---|---|---|---|---|---|
| No. | Population | IDSL /<br>Example<br>Shell | Title | Programming Notes | Deliverable |
| 3.34. | Safety | 207966/primar<br>y_02/T3.67 | Summary of Hepatic Safety Profile: Assessment of Risk of Hepatoxicity Adverse Events of Special Interest by System Organ Class and Preferred Term (Number of Subjects and Occurrences) | | M12, M26,<br>EOS |
| 3.35. | Safety | 207966/primar<br>y_02/T3.68 | Summary of Hypersensitivity Reaction (HSR) Adverse<br>Events of Special Interest by System Organ Class and<br>Preferred Term (Number of Subjects and Occurrences) | | M12, M26,<br>EOS |
| 3.36. | Safety | 207966/primar<br>y_02/T3.69 | Summary of Rash Adverse Events of Special Interest by<br>System Organ Class and Preferred Term (Number of<br>Subjects and Occurrences) | | M12, M26,<br>EOS |
| 3.37. | Safety | 207966/primar<br>y_02/T3.70 | Summary of Prolongation of the Corrected QT Interval of<br>the ECG in Supra Therapeutic Doses Adverse Events of<br>Special Interest by System Organ Class and Preferred<br>Term (Number of Subjects and Occurrences) | | M12, M26,<br>EOS |
| 3.38. | Safety | 207966/primar<br>y_02/T3.73 | Summary of Bipolar Disorder Adverse Events of Special Interest by System Organ Class and Preferred Term (Number of Subjects and Occurrences) | | M12, M26,<br>EOS |
| 3.39. | Safety | 207966/primar<br>y_02/T3.74 | Summary of Psychosis Adverse Events of Special Interest by System Organ Class and Preferred Term (Number of Subjects and Occurrences) | | M12, M26,<br>EOS |
| 3.40. | Safety | 207966/primar<br>y_02/T3.75 | Summary of Mood Disorder Adverse Events of Special<br>Interest by System Organ Class and Preferred Term<br>(Number of Subjects and Occurrences) | | M12, M26,<br>EOS |

| Safety | Safety: Tables | | | | |
|---|---|---|---|---|---|
| No. | Population | IDSL /<br>Example<br>Shell | Title | Programming Notes | Deliverable |
| 3.41. | Safety | 207966/primar<br>y_02/T3.77 | Summary of Sleep Disorder Adverse Events of Special Interest by System Organ Class and Preferred Term (Number of Subjects and Occurrences) | | M12, M26,<br>EOS |
| 3.42. | Safety | 207966/primar<br>y_02/T3.79 | Summary of Weight Gain Adverse Events of Special Interest by System Organ Class and Preferred Term (Number of Subjects and Occurrences) | | M12, M26,<br>EOS |
| 3.43. | Safety | 207966/primar<br>y_02/T3.80 | Summary of Rhabdomyolysis Adverse Events of Special Interest by System Organ Class and Preferred Term (Number of Subjects and Occurrences) | | M12, M26,<br>EOS |
| 3.44. | Safety | 207966/primar<br>y_02/T3.81 | Summary of Pancreatitis Adverse Events of Special Interest by System Organ Class and Preferred Term (Number of Subjects and Occurrences) | | M12, M26,<br>EOS |
| 3.45. | Safety | 207966/primar<br>y_02/T3.82 | Summary of Impact on Creatinine Adverse Events of Special Interest by System Organ Class and Preferred Term (Number of Subjects and Occurrences) | | M12, M26,<br>EOS |
| 3.46. | Safety | 207966/primar<br>y_02/T3.83 | Summary of Safety in Pregnancy Adverse Events of Special Interest by System Organ Class and Preferred Term (Number of Subjects and Occurrences) | | M12, M26,<br>EOS |
| 3.47. | Safety | 207966/primar<br>y_02/T3.6 | Summary of All Adverse Events by System Organ Class and Maximum Toxicity | | HL, M12, M26,<br>EOS |
| 3.48. | Safety | 207966/primar<br>y_02/T3.13 | Summary of All Drug-related Adverse Events by System Organ Class and Maximum Toxicity | | HL, M12, M26,<br>EOS |

| Safety: | Safety: Tables | | | | |
|---|---|---|---|---|---|
| No. | Population | IDSL /<br>Example<br>Shell | Title | Programming Notes | Deliverable |
| 3.49. | Safety | 207966/primar<br>y_02/T3.43 | Summary of Maximum Post-Baseline Emergent Chemistry Toxicities | | M12, M26,<br>EOS |
| 3.50. | Safety | 207966/primar<br>y_02/T3.45 | Summary of Maximum Post-Baseline Emergent Hematology Toxicities | | M12, M26,<br>EOS |

## 12.12.8. Safety Figures

| Safety | : Figures | | | | |
|---|---|---|---|---|---|
| No. | Population | IDSL /<br>Example<br>Shell | Title | Programming Notes | Deliverable |
| Advers | se Events | | | | |
| 3.01. | Safety | 207966/primar<br>y_02/F3.1 | Plot of Common Adverse Events and Relative Risk – Q2M vs. DTG + RPV - Excluding Study Drug ISRs | | M12, M26,<br>EOS |
| Study | Drug Injection | Site Reaction A | dverse Events (display for Q2M arm only) | | |
| 3.02. | Safety | 207966/primar<br>y_02/F3.2 | Plot of Common Study Drug Injection Site Reaction<br>Adverse Events | Only display first panel | M12, M26,<br>EOS |
| 3.03. | Safety | 207966/primar<br>y_02/F3.3 | Plot of Onset, Duration, and Severity of Overall and Common Study Drug Injection Site Reaction AEs by Maximum Grade - CAB and/or RPV | | M12, M26,<br>EOS |
| 3.04. | Safety | 207966/primar<br>y_02/F3.4 | Plot of Onset, Duration, and Severity of Overall and<br>Common Drug-related Study Drug Injection Site Reaction<br>AEs by Maximum Grade - CAB | | M12, M26,<br>EOS |
| 3.05. | Safety | 207966/primar<br>y_02/F3.5 | Plot of Onset, Duration, and Severity of Overall and<br>Common Drug-related Study Drug Injection Site Reaction<br>AEs by Maximum Grade - RPV | | M12, M26,<br>EOS |
| 3.06. | Safety | 207966/primar<br>y_02/F3.6 | Plot of Incidence of Maintenance Phase Study Drug<br>Injection Site Reaction Adverse Events by Visit (Overall<br>and Common) - CAB and/or RPV | | M12, M26,<br>EOS |
| 3.07. | Safety | 207966/primar<br>y_02/F3.7 | Plot of Incidence of Maintenance Phase Drug-Related<br>Study Drug Injection Site Reaction Adverse Events by Visit<br>(Overall and Common) - CAB | | M12, M26,<br>EOS |

| Safety | : Figures | | | | |
|---|---|---|---|---|---|
| No. | Population | IDSL /<br>Example<br>Shell | Title | Programming Notes | Deliverable |
| 3.08. | Safety | 207966/primar<br>y_02/F3.8 | Plot of Incidence of Maintenance Phase Drug-Related<br>Study Drug Injection Site Reaction Adverse Events by Visit<br>(Overall and Common) - RPV | | M12, M26,<br>EOS |
| 3.09. | Safety | 207966/primar<br>y_02/F3.9 | Plot of Incidence of Grade 3-5 Maintenance Phase Study<br>Drug Injection Site Reaction Adverse Events by Visit<br>(Overall and Common) - CAB and/or RPV | | M12, M26,<br>EOS |
| 3.10. | Safety | 207966/primar<br>y_02/F3.10 | Plot of Incidence of Grade 3-5 Maintenance Phase Drug-<br>related Study Drug Injection Site Reaction Adverse Events<br>by Visit (Overall and Common) - CAB | | M12, M26,<br>EOS |
| 3.11. | Safety | 207966/primar<br>y_02/F3.11 | Plot of Incidence of Grade 3-5 Maintenance Phase Drug-<br>related Study Drug Injection Site Reaction Adverse Events<br>by Visit (Overall and Common) - RPV | | M12, M26,<br>EOS |
| Labora | itory | | | | |
| 3.12. | Safety | 207966/primar<br>y_02/F3.12 | Scatter Plot of Maximum vs. Baseline for ALT | | M12, M26,<br>EOS |
| 3.13. | Safety | 207966/primar<br>y_02/F3.13 | Scatter Plot of Maximum Total Bilirubin vs. Maximum ALT | | M12, M26,<br>EOS |
| 3.14. | Safety | 207966/primar<br>y_02/F3.14 | Matrix Plot of Maximum Liver Chemistries | | M12, M26,<br>EOS |
| 3.15. | Safety | 207966/primar<br>y_02/F3.15 | Bar Chart of Lipid NCEP Categories at Month 12 vs. Baseline - Triglycerides, Total Cholesterol, LDL Cholesterol | For M26, replace the 'Month 12' in the title with 'Month 26' | M12, M26,<br>EOS |
| 3.16. | Safety | 207966/primar<br>y_02/F3.16 | Bar Chart of Lipid NCEP Categories at Month 12 vs. Baseline - HDL Cholesterol | For M26, replace the 'Month 12' in the title with 'Month 26' | M12, M26,<br>EOS |

| Safety: Figures | | | | | |
|---|---|---|---|---|---|
| No. | Population | IDSL /<br>Example<br>Shell | Title | Programming Notes | Deliverable |
| Exposi | Exposure (display for Q2M arm only) | | | | |
| 3.17. | Safety | 207966/primar<br>y_02/F3.17 | Histogram of Timeliness of Injections | | M12, M26,<br>EOS |

#### 12.12.9. Health Outcomes Tables

| Health | Health Outcomes: Tables | | | | |
|---|---|---|---|---|---|
| No. | Population | IDSL /<br>Example<br>Shell | Title | Programming Notes | Deliverable |
| HIV De | pendent Qual | ity of Life (HIVD | QoL) | | |
| 6.01. | 6.01. ITT-E HO_T1 Proportion of Subjects with Each Individual Questionnaire Item Score in HIVDQoL by Visit | | | | |
| 6.02. | ITT-E | HO_T2 | Summary of HIVDQoL in Overview Items, Domain<br>Weighted Impact Scores and Average Weighted Impact<br>Score by Visit | | M12 |
| 6.03. | ITT-E | HO_T3 | Summary of HIVDQoL Change from Baseline in Overview Items, Domain Weighted Impact Scores and Average Weighted Impact Score by Visit | | M12 |
| HIV Tr | eatment Satis | faction Question | nnaire Status Version (HIVTSQs) | | |
| 6.04. | ITT-E | 207966/primar<br>y_02/T6.14 | Proportion of Subjects with HIVTSQs - Individual Item Scores by Visit | Note: no LOCF | M12 |
| 6.05. | ITT-E | 207966/primar<br>y_02/T6.16 | Summary of HIVTSQs - Total Treatment Satisfaction Score by Visit | | M12 |
| 6.06. | ITT-E | 207966/primar<br>y_02/T6.18 | Summary of HIVTSQs - Change from Baseline in Total Treatment Satisfaction Score by Visit | Note: Do not include column for prior exposure | M12 |
| 6.07. | ITT-E | 207966/primar<br>y_02/T6.20 | Summary of HIVTSQs - Change from Baseline in Individual Item Score by Visit | Note: no LOCF; do not include column for prior exposure | M12 |

| Health | Health Outcomes: Tables | | | | |
|---|---|---|---|---|---|
| No. | Population | IDSL /<br>Example<br>Shell | Title | Programming Notes | Deliverable |
| HIV Tre | eatment Satist | faction Question | naire Change Version (HIVTSQc) | | |
| 6.08. | ITT-E | 207966/primar<br>y_02/T6.23 | Proportion of Subjects with HIVTSQc - Individual Item Change Score at Month 12 | | M12 |
| 6.09. | ITT-E | 207966/primar<br>y_02/T6.25 | Summary of HIVTSQc - Total Treatment Satisfaction<br>Change Score at Month 12 | | M12 |
| 6.10. | ITT-E | 207966/primar<br>y_02/T6.27 | Summary of HIVTSQc - Individual Item Change Score at Month 12 | | M12 |
| Prefere | ence (display | for Q2M arm only | y) | | |
| 6.11. | ITT-E | 207966/primar<br>y_02/T6.38 | Proportion of Subjects with Response to Each Individual Question in Preference Questionnaire at Month 12 for Subjects in Q2M | Display questions and responses per the data. Do not include footnotes [1] and [2] | M12 |
| Reason | Reasons for Switch (display for Q2M arm only) | | | | |
| 6.12. | ITT-E | 207966/primar<br>y_02/T6.41 | Reasons for Switch at Baseline for Subjects from Oral CAB + RPV to Q2M | Display responses per the data. | M12 |

## 12.12.10. Virology Tables

| Virolog | Virology: Tables | | | | |
|---|---|---|---|---|---|
| No. | Population | IDSL /<br>Example<br>Shell | Title | Programming Notes | Deliverable |
| Genoty | ype | | | | • |
| 7.01. | CVF | 207966/primar<br>y_02/T7.1 | Summary of the Prevalence of Known INI Resistance<br>Mutations at Time of CVF - Plasma Sample | | M12, M26,<br>EOS |
| 7.02. | CVF | 207966/primar<br>y_02/T7.2 | Summary of the Prevalence of Major Resistance Mutations of NRTI, NNRTI and PI Class at Time of CVF - Plasma Sample | | M12, M26,<br>EOS |
| 7.03. | CVF | 207966/primar<br>y_02/T7.3 | Summary of Genotypic Susceptibility at Time of CVF - Plasma Sample | | M12, M26,<br>EOS |
| Pheno | type | | | | |
| 7.04. | CVF | 207966/primar<br>y_02/T7.4 | Summary of Phenotype Susceptibility at Time of CVF - Plasma Sample | | M12, M26,<br>EOS |
| 7.05. | CVF | 207966/primar<br>y_02/T7.5 | Summary of Phenotype: Number of Drugs to Which Subject is Phenotypic Resistant or Partial Sensitive or Sensitive at Time of CVF - Plasma Sample | | M12, M26,<br>EOS |
| 7.06. | CVF | 207966/primar<br>y_02/T7.6 | Summary of Fold Change to CAB and RPV at Time of CVF - Plasma Sample | Display for Q2M arm only | M12, M26,<br>EOS |
| 7.07. | CVF | 207966/primar<br>y_02/T7.7 | Summary of Net Assessment at Time of CVF - Plasma Sample | | M12, M26,<br>EOS |

| Virolog | Virology: Tables | | | | |
|---|---|---|---|---|---|
| No. | Population | IDSL /<br>Example<br>Shell | Title | Programming Notes | Deliverable |
| Miscell | aneous | | | | |
| 7.08. | CVF | 207966/primar<br>y_02/T7.8 | Summary of Viral load, Genotypic and Phenotypic data for Subjects Who Met Confirmed Virologic Failure Criteria during the Maintenance Phase | | M12, M26,<br>EOS |

## 12.12.11. ICH Listings

Strata and Latest Subject Id will not be included in any listings taken from 207966/primary\_02.

| ICH: L | ICH: Listings | | | | |
|---|---|---|---|---|---|
| No. | Population | IDSL /<br>Example<br>Shell | Title | Programming Notes | Deliverable |
| Study | Population | | | | |
| 1. | Screened | 207966/primar<br>y_02/L3 | Listing of Reasons for Screen Failure | | M12, M26,<br>EOS |
| 2. | ITT-E | 207966/primar<br>y_03/L4 | Listing of Reasons for Study Withdrawal | | M12, M26,<br>EOS |
| 3. | Enrolled | 207966/primar<br>y_02/L2 | Listing of Treatment Assignment | Do not include footnotes and columns for randomization number, randomization and actual strata and deviation. Do not display randomized treatment | M12, M26,<br>EOS |
| 4. | ITT-E | 207966/primar<br>y_02/L6 | Listing of Important Protocol Deviations | | M12, M26,<br>EOS |
| 5. | ITT-E | 207966/primar<br>y_02/L8 | Listing of Subjects with Inclusion/Exclusion Criteria Deviations | | M12, M26,<br>EOS |
| 6. | ITT-E | 207966/primar<br>y_02/L7 | Listing of Protocol Deviations Leading to Exclusion from the Per-Protocol Population | | M12, M26,<br>EOS |
| 7. | ITT-E | 207966/primar<br>y_02/L9 | Listing of Demographic Characteristics | | M12, M26,<br>EOS |

| ICH: L | ICH: Listings | | | | |
|---|---|---|---|---|---|
| No. | Population | IDSL /<br>Example<br>Shell | Title | Programming Notes | Deliverable |
| 8. | ITT-E | 207966/primar<br>y_02/L10 | Listing of Race | | M12, M26,<br>EOS |
| 9. | ITT-E | 207966/primar<br>y_02/L36 | Listing of Concomitant ART Medications Received | Do not include final column for phase during which concomitant | M12, M26,<br>EOS |
| 10. | ITT-E | 207966/primar<br>y_02/L5 | Listing of Reasons for Study Drug Discontinuation | | M12, M26,<br>EOS |
| Efficad | у | | | | |
| 11. | ITT-E | 207966/primar<br>y_02/L11 | Listing of Study Outcome (50 c/mL Threshold) at Month 12 - Snapshot Analysis | For M26, replace the 'Month 12' in the title with 'Month 26' | M12, M26,<br>EOS |
| Safety | : Exposure | | | | |
| 12. | Safety | 207966/primar<br>y_02/L12 | Listing of Investigational Product Exposure Data | | M12, M26,<br>EOS |
| Advers | se Events | | | | |
| 13. | Safety | 207966/primar<br>y_02/L19 | Listing of All Adverse Events | | M12, M26,<br>EOS |
| 14. | Safety | 207966/primar<br>y_02/L13 | Listing of Subject Numbers for Individual Adverse Events | | M12, M26,<br>EOS |
| 15. | Safety | 207966/primar<br>y_02/L15 | Listing of Fatal Adverse Events | | M12, M26,<br>EOS |
| 16. | Safety | 207966/primar<br>y_02/L16 | Listing of Non-Fatal Serious Adverse Events | | M12, M26,<br>EOS |

| ICH: Li | ICH: Listings | | | | |
|---|---|---|---|---|---|
| No. | Population | IDSL /<br>Example<br>Shell | Title | Programming Notes | Deliverable |
| 17. | Safety | 207966/primar<br>y_02/L14 | Listing of Reasons for Considering as a Serious Adverse<br>Event | | M12, M26,<br>EOS |
| 18. | Safety | 207966/primar<br>y_02/L17 | Listing of Adverse Events Leading to Withdrawal/Permanent Discontinuation of Investigational Product | | M12, M26,<br>EOS |
| Safety | Hepatobiliary | y (Liver) | | • | |
| 19. | Safety | 207966/primar<br>y_02/L21 | Listing of Medical Conditions for Subjects with Liver Stopping Events | | M12, M26,<br>EOS |
| 20. | Safety | 207966/primar<br>y_02/L22 | Listing of Substance Use for Subjects with Liver Stopping Events | | M12, M26,<br>EOS |
| Safety | ECG | | | • | |
| 21. | Safety | 207966/primar<br>y_02/L23 | Listing of ECG Values for Subjects with a Value of Potential Clinical Importance | | M12, M26,<br>EOS |
| 22. | Safety | 207966/primar<br>y_02/L24 | Listing of ECG Findings | | M12, M26,<br>EOS |

## 12.12.12. Non-ICH Listings

Strata and Latest Subject Id will not be included in any listings taken from 207966/primary\_02.

| Non-IC | Non-ICH: Listings | | | | |
|---|---|---|---|---|---|
| No. | Population | IDSL /<br>Example<br>Shell | Title | Programming Notes | Deliverable |
| Study | Population | | | | |
| 23. | ITT-E | 207966/primar<br>y_02/L34 | Listing of Subjects Who were Rescreened | Do not include annotation [1] | M12, M26,<br>EOS |
| 24. | ITT-E | 207966/primar<br>y_02/L37 | Listing of ART Medications Received during Long-term Follow-up Phase | | M12, M26,<br>EOS |
| 25. | ITT-E | 207966/primar<br>y_02/L39 | Listing of Medical History of Seizure | | M12, M26,<br>EOS |
| Advers | se Events | | | | • |
| 26. | LTFU | 207966/primar<br>y_02/L19 | Listing of All Adverse Events (Long-term Follow-up Phase) | | M12, M26,<br>EOS |
| Efficad | у | | | | • |
| 27. | CVF | 207966/primar<br>y_02/L40 | Listing of All Plasma HIV-1 RNA Data for Subjects with Confirmed Virologic Failure | | M12, M26,<br>EOS |
| 28. | ITT-E | 207966/primar<br>y_02/L41 | Listing of All Plasma HIV-1 RNA Data for Subjects with Viral Load >=50 c/mL during the Maintenance Phase | | M12, M26,<br>EOS |
| 29. | ITT-E | 207966/primar<br>y_02/L43 | Listing of HIV-1 Associated Conditions | | M12, M26,<br>EOS |
| 30. | CVF | 207966/primar<br>y_02/L62 | Listing of Replication Capacity in IN and PR/RT Region | | M12, M26,<br>EOS |

## 12.13. Appendix 13: Example Mock Shells for Data Displays

Available upon request.